

Title: Special Drug Use Surveillance of Adcetris IV Infusion (All-Case Surveillance)
"Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell
Lymphoma"

NCT Number: NCT02139592

Statistical analysis plan Approve Date: 27-Jan-2017

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

# Statistical Analysis Plan

# ADCETRIS IV Infusion – Special Drug Use Surveillance (All-case Surveillance) "Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell Lymphoma"



3rd version: Prepared on January 27, 2017

## Table of Contents

| 1.0 | Definition of Analysis sets and Terms and Handling of Test/Measurement Data | |
|---|---|---|
| 1.1 | Analysis sets | |
| 1.1 | .1 Safety analysis set | 1 |
| 1.1 | .2 Efficacy analysis set | 1 |
| 1.2 | Definition | 1 |
| 1.3 | Display digits | 9 |
| 1.4 | Level of significance and confidence coefficient | 9 |
| 1.5 | Handling of test data | 9 |
| 1.6 | Handling of missing data | 12 |
| 1.7 | Others | 12 |
| 2.0 | Patient Disposition (Patient Disposition Diagram) | 13 |
| 3.0 | Patient Demographics and Baseline Characteristics | 14 |
| 3.1 | Patient Demographics and Baseline Characteristics | 14 |
| 3.2 | Prior drug therapy (details) | 16 |
| 4.0 | Treatment Given | 18 |
| 4.1 | Treatment given | 18 |
| 4.2 | Premedication to prevent infusion reaction | 20 |
| 4.3 | Patient demographics and baseline characteristics by initial dose of Adcetris | 20 |
| 5.0 | Safety Analysis | 22 |
| 5.1 | Occurrences of adverse events and adverse drug reactions/infections | 22 |
| 5.1 | .1 Occurrence of adverse events | 22 |
| 5.1 | .2 Occurrence of adverse drug reactions/infections | 24 |
| 5.2 | Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occ | currences of |
| | adverse events and adverse drug reactions/infections by outcome | 25 |
| 5.2 | 2.1 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and | occurrence |
| of | adverse events by outcome | 25 |
| 5.2 | Occurrence of adverse events by CTCAE Grade (the worst one) | 26 |
| 5.2 | 2.3 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and | loccurrence |
| of | adverse drug reactions/infections by outcome | |
| 5.2 | Occurrence of adverse drug reactions/infections by CTCAE Grade (the worst one) | 30 |
| 5.3 | Percentage of patients with adverse drug reactions/infections by patient demographics a | nd baseline |
| | characteristics and treatment given | |
| 5.4 | Occurrence of adverse drug reactions/infections by age group | 33 |
| 5.5 | Occurrence of adverse drug reactions/infections by presence or absence and grade of concur | rent hepatic |
| | disorder | |
| 5.6 | Occurrence of adverse drug reactions/infections by presence or absence and grade of conc | |
| | disorder | |
| 5.7 | Occurrence of serious adverse events | 35 |

| 5.8 | Cha | ange in test data over time | 36 |
|---|---|---|---|
| 5. | 8.1 | Change in laboratory test results over time | 36 |
| 5.9 | An | alysis of items of particular interest | 36 |
| 5. | 9.1 | Occurrence of the adverse drug reaction of peripheral nerve disorder and infections | 36 |
| 5. | 9.2 | Occurrence of peripheral nerve disorders considered related to Adcetris by patient demograph | ics |
| ar | nd base | eline characteristics and treatment given | 37 |
| 5. | 9.3 | Treatment with Adcetris at the onset of peripheral nerve disorders considered related to Adcetris | 39 |
| 5. | 9.4 | Outcome of peripheral nerve disorders (≥CTCAE Grade 3) considered related to Adcetris by act | ion |
| ta | ken wi | ith Adcetris | 39 |
| 5. | 9.5 | Occurrence of infections considered related to Adcetris by presence or absence of drugs used | for |
| th | e prev | ention of infection | 40 |
| 5. | 9.6 | Occurrence of infections considered related to Adcetris by presence or absence of pr | ior |
| he | ematop | ooietic stem cell transplantation | 41 |
| 5. | 9.7 | Occurrence of neutropenia considered related to Adcetris by patient demographics and basel | ine |
| cł | naracte | ristics | 41 |
| 5. | 9.8 | Treatment with Adcetris at the onset of neutropenia considered related to Adcetris | 42 |
| 5. | 9.9 | Outcome of neutropenia considered related to Adcetris by action taken with Adcetris | 43 |
| 5. | 9.10 | Occurrence of infusion reaction considered related to Adcetris | 43 |
| 5. | 9.11 | Occurrence of the new onset of infusion reaction observed within 2 days after treatment w | rith |
| A | dcetris | and considered related to Adcetris (time of the new onset) | 44 |
| 5. | 9.12 | Occurrence of infusion reaction observed within 2 days after treatment with Adcetris a | ınd |
| co | onsider | red related to Adcetris by use or non-use of premedication to prevent infusion reaction | 44 |
| 5. | 9.13 | Occurrence of adverse drug reactions of pulmonary disorder and infections | 46 |
| 5.10 | Lis | t of actions taken with Adcetris in patients experiencing peripheral nerve disorders considered rela | ted |
| | to A | Adcetris | 46 |
| 5.11 | Lis | t of actions taken with Adcetris in patients experiencing neutropenia considered related to Adcetris | 47 |
| 6.0 | Eff | icacy Analysis | 48 |
| 6.1 | Bes | st response | 48 |
| 6.2 | Day | ys to the best response | 48 |
| 6.3 | Ov | erall survival | 48 |
| Appen | dix: D | efinition of Pulmonary Disorders (MedDRA Preferred Terms) | 49 |

#### 1.0 Definition of Analysis Sets and Terms and Handling of Test/Measurement Data

#### 1.1 Analysis sets

#### 1.1.1 Safety analysis set

In this survey, the safety analysis set is defined as patients treated with Adcetris IV Infusion with no major protocol violation and evaluable for safety.

#### 1.1.2 Efficacy analysis set

In this survey, the efficacy analysis set is defined as patients treated with Adcetris IV Infusion with no major protocol violation and evaluable for efficacy.

#### Definition

| Term | Definition |
|---|---|
| This/the product | Refers to Adcetris for intravenous drip infusion in this Statistical Analysis |
| | Plan. |
| SOC | MedDRA/J System Organ Class |
| HLGT | MedDRA/J High Level Group Term |
| PT | MedDRA/J Preferred Term |
| LLT | MedDRA/J Lowest Level Term |
| Patients registered | Patients whose registration has been approved |
| Patients whose case report | Patients whose case report forms have been collected |
| forms are available | |
| Patients whose case report | Patients registered but whose case report form have not been collected |
| forms are not available | |
| Fixed patients | Patients whose case report forms are available, with the date of case report |
| | form completion entered in the PMS system |
| Non-fixed patients | Patients whose case report forms are available, with the date of case report |
| | form completion not entered in the PMS system |
| Safety analysis set | Fixed patients included in the safety analysis set |
| Safety analysis set (Hodgkin's | Patients included in the safety analysis set whose diagnosis is Hodgkin's |
| lymphoma) | lymphoma |
| Safety analysis set (anaplastic | Patients included in the safety analysis set whose diagnosis is anaplastic |
| large-cell lymphoma) | large-cell lymphoma |
| Patients excluded from the | Fixed patients excluded from the safety analysis set |
| safety analysis set | |
| Efficacy analysis set | Patients included in the safety analysis set who are also included in the |
| | efficacy analysis set |
| Patients excluded from the | Patients included in the safety analysis set who are excluded from the |
| efficacy analysis set | efficacy analysis set |
| Patients completing treatment | Patients completing 16 cycles of treatment with Adcetris |
| Patients discontinuing treatment | Patients not completing 16 cycles of treatment with Adcetris |

| Term | Definition |
|---|---|
| Adverse drug reactions, etc. | Refers to "adverse drug reactions and infections." |
| | Adverse events not considered "not related" to Adcetris by the |
| | investigator. |
| | In this Statistical Analysis Plan, the term "adverse drug reactions and |
| | infections" is used in titles and the term "adverse drug reactions, etc." is |
| | used in text and tables. |
| Serious adverse events | Adverse events considered "serious" by the investigator. |
| | Events listed in the MedDRA Coding List in the Takeda Medically |
| | Significant AE List should be regarded as serious even if they are |
| | considered "non-serious" by the investigator. |
| Number of patients with | Number of patients experiencing adverse events or adverse drug reactions, |
| adverse events/adverse drug | etc. |
| reactions | |
| Number of adverse | Number of adverse events or adverse drug reactions, etc., observed |
| events/adverse drug reactions | |
| Percentage of patients with | [For safety analysis using patients included in the safety analysis set] |
| adverse events/adverse drug | Is calculated using the following formula: (number of patients with |
| reactions | adverse events/adverse drug reactions) / (number of patients included in |
| | the safety analysis set) $\times$ 100. |
| | [For safety analysis using patients excluded from the safety analysis set] |
| | Is calculated using the following formula: (number of patients with |
| | adverse events/adverse drug reactions) / (number of patients excluded |
| | from the safety analysis set) × 100. |
| Percentage of adverse | [For safety analysis using patients included in the safety analysis set] |
| events/adverse drug reactions | Is calculated using the following formula: (number of adverse |
| observed | events/adverse drug reactions observed) / (number of patients included in |
| | the safety analysis set) $\times$ 100. |
| | [For safety analysis using patients excluded from the safety analysis set] |
| | Is calculated using the following formula:( number of adverse |
| | events/adverse drug reactions observed) / (number of patients excluded |
| | from the safety analysis set) × 100. |
| Time of onset | |
| | (or adverse drug reactions, etc.) – date of the initial dose of Adcetris + 1. |
| If the day, month, and year of onset of adverse events (or a | |
| | reactions, etc.) are unknown, the time of onset should be handled as |
| | missing, and the category for the time of onset should be "unknown." |
| Time to the worst grade | Is calculated using the following formula: date of the worst CTCAE grade |
| | - date of the initial dose of Adcetris + 1. |

| Term | Definition | | |
|---|---|---|---|
| | If the day, month, and year of the worst CTCAE grade are unknown, the | | |
| | date of the worst CTCAE grade should be handled as missing, and the | | |
| | category for the date of the worst CTCAE grade should be "unknown." | | |
| Patients with concurrent hepatic | Patients having a | concurrent illness that falls u | under the category of |
| disorder | Standardized Med | DRA Query (SMQ) Code 20 | 0000005 (SMQ Hepatic |
| | disorders [Scope: | Narrow]) | |
| Grade of hepatic disorder | The ALT or AST | level at baseline with the h | nighest grade will be used to |
| | determine the grad | le of hepatic disorder. The g | rades of ALT and AST levels |
| | will be determined | d according to the following | tables, and the grade should |
| | be "unknown" if e | either the ALT or AST level | s missing: |
| | ALT | | |
| | | Male | Female |
| | None | ≤42 IU/L | ≤23 IU/L |
| | Grade 1 | >42 to ≤126 IU/L | >23 to ≤69 IU/L |
| | Grade 2 | >126 to ≤210 IU/L | >69 to ≤115 IU/L |
| | ≥Grade 3 | >210 IU/L | >115 IU/L |
| | AST | , | |
| | None ≤30 IU/L | | |
| | Grade 1 >30 to ≤90 IU/L | | |
| | Grade 2 >90 to ≤150 IU/L | | |
| | ≥Grade 3 | >150 IU/L | |
| Patients with concurrent renal | Patients having a concurrent illness that falls under the category of Takeda | | |
| disorder | MedDRA Query ( | TMQ) (Renal disease) | |
| Grade of renal disorder | The serum creatin | ine level at baseline will be | classified as shown in the |
| | table below. If the | serum creatinine level at ba | seline is missing, the grade |
| | of renal disorder s | hould be "unknown:" | |
| | Serum creatinine | | |
| | | Male | Female |
| | None | ≤1.07 mg/dL | ≤0.79 mg/dL |
| | Grade 1 | >1.07 to ≤1.605 mg/dL | >0.79 to ≤1.185 mg/dL |
| | Grade 2 | >1.605 to ≤3.21 mg/dL | >1.185 to ≤2.37 mg/dL |
| | ≥Grade 3 >3.21 mg/dL >2.37 mg/d | | >2.37 mg/dL |
| Patients with a past history of | Patients with a past history that falls under the category of Appendix | | |
| pulmonary disorder | "Definition of Pulmonary Disorders" | | |
| | (If "No concurrent illness existed at the initiation of treatment with | | |
| | Adcetris" is selected in the field of "Past history/concurrent illness of | | |
| | pulmonary disorders" in the case report form, the pulmonary disorder | | |

| Term | Definition |
|---|---|
| | should be regarded as a past history.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of Appendix |
| pulmonary disorder | "Definition of Pulmonary Disorders" |
| | (If "A concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | pulmonary disorders" in the case report form, the pulmonary disorder |
| | should be regarded as a concurrent illness.) |
| Patients with a past history of | Patients with a past history that falls under the category of MedDRA SMQ |
| malignant tumour | Code 20000194 (SMQ Malignant tumours [Scope: Narrow]) |
| | (If "No concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | malignant tumours" in the case report form, the pulmonary disorder should |
| | be regarded as a past history.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| malignant tumour | SMQ Code 20000194 (SMQ Malignant tumours [Scope: Narrow]) |
| | (If "A concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | malignant tumours" in the case report form, the pulmonary disorder should |
| | be as a concurrent illness.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| diabetes mellitus | SMQ Code 20000041 (SMQ Hyperglycaemia/new onset diabetes mellitus |
| | [Scope: Narrow]) |
| Patients with hypertension | Patients with a concurrent illness that falls under the category of MedDRA |
| | SMQ Code 20000147 (SMQ Hypertension [Scope: Narrow]) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| dyslipidaemia | SMQ Code 20000026 (SMQ Dyslipidaemia [Scope: Narrow]) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| hyperuricaemia | PT Code 10020903 (Hyperuricaemia) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| infection | SOC Code 10021881 (Infections and infestations) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of SMQ |
| peripheral neuropathy | Code 20000034 (SMQ Peripheral neuropathy [Scope: Narrow]) |
| Patients with other concurrent | Patients with any concurrent illness other than those listed above |
| illnesses | |
| Antibiotics/synthetic | Drugs with the first three digits of YJ Code being either one of 611 to 616, |
| antibacterial agents | 619, or 624 that are entered in the field of "Drugs used for the prevention |
| | C: C: 1: 22 (IC 11 |
| | of infection" (If more than one antibiotics/synthetic antibacterial agents |
| | are used in the same patient, it will be counted as one patient.) |

| digits being 6290002 or 6290004 that are entered in the field of "Drugs used for the prevention of infection" (If more than one antifungals are used in the same patient, it will be counted as one patient.) Antivirals Drugs with the first three digits of YJ Code being 625 that are entered in the field of "Drugs used for the prevention of infection" (If more than one antivirals are used in the same patient, it will be counted as one patient.) Trimethoprim-sulfamethoxazole combinations Drugs with YJ Code being 62901000 that are entered in the field of "Drugs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations are used in the same patient, it will be counted as one patient). Other prophylactics against infections are used in the same patient, it will be counted as one patient). Any drug entered in the field of "Drugs used for the prevention of infection" other than prophylactics against infections firsted above (If more than one other prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Adverse events with "Sensory neuropathy" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders in the field of "Adverse events: [1] Peripheral nerve disorders in the field of "Adverse events: [1] Peripheral nerve disorders in the field of "Adverse events: | Term | Definition |
|---|---|---|
| Antivirals Drugs with the first three digits of YJ Code being 625 that are entered in the field of "Drugs used for the prevention of infection" (If more than one antivirals are used in the same patient, it will be counted as one patient.) Trimethoprim-sulfamethoxazole combinations Purgs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations "Drugs with YJ Code being 62901000 that are entered in the field of "Drugs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations are used in the same patient, it will be counted as one patient.) Other prophylactics against infections are used in the same patient, it will be counted as one patient.) Any drug entered in the field of "Drugs used for the prevention of infection" other than prophylactics against infections isted above (If more than one other prophylactics against infections isted above (If more than one other prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events. [1] Peripheral nerve disorders" in the field of "Adverse events. [1] Peripheral nerve disorders" in the field of "Adverse events. [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders] in the case report form. MedDRA PT Code 10034581 (and the case report form. MedDRA PT Code 10039331 should be assigned, regardless of data entered in "Symptoms" in the field. Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events [1] Peripheral nerve disorders" in the field of "Adverse events [1] Peripheral nerve disorders" in the field of "Adverse events [1] Peripheral nerve disorders | | digits being 6290002 or 6290004 that are entered in the field of "Drugs |
| Antivirals Drugs with the first three digits of YJ Code being 625 that are entered in the field of "Drugs used for the prevention of infection" (If more than one antivirals are used in the same patient, it will be counted as one patient.) Trimethoprim-sulfamethoxazole combinations Drugs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations in the field of "Drugs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations are used in the same patient, it will be counted as one patient.) Other prophylactics against infections listed above (If more than one other prophylactics against infections listed above (If more than one other prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Motor neuropathy" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse event) Pulmonary disorders (as adverse events) Pulmonary Disorders (as adv | | used for the prevention of infection" (If more than one antifungals are |
| the field of "Drugs used for the prevention of infection" (If more than one antivirals are used in the same patient, it will be counted as one patient.) Trimethoprim-sulfamethoxazole combinations "Drugs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations are used in the same patient, it will be counted as one patient.) Other prophylactics against infections are used in the same patient, it will be counted as one patient.) Any drug entered in the field of "Drugs used for the prevention of infections of infections of infections of infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral merve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders in the field of "Adverse events: [1] Peripheral nerve disorders in the field of "Adverse events: [1] Peripheral nerve disorders in the field of "Adverse events: [1] Peripheral nerve disorders in the case report form. MedDRA PT Code 1002931 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse events) Pulmonary disorders (as adverse events) Pulmonary Disorders Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms en | | used in the same patient, it will be counted as one patient.) |
| antivirals are used in the same patient, it will be counted as one patient.) Trimethoprim-sulfamethoxazole combinations "Drugs with YJ Code being 62901000 that are entered in the field of "Drugs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations are used in the same patient, it will be counted as one patient.) Other prophylactics against infections infections infections infections other than prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy adverse events with "Sensory neuropathy" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in | Antivirals | Drugs with the first three digits of YJ Code being 625 that are entered in |
| Trimethoprim-sulfamethoxazole combinations Drugs with YJ Code being 62901000 that are entered in the field of "Drugs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations are used in the same patient, it will be counted as one patient.) Other prophylactics against infections infection of infection of other than prophylactics against infections listed above (If more than one other prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders of data entered in "Symptoms" in the field. Pulmonary disorders (as an adverse event) Adverse events that fall under the category of Appendix "Definition of Pulmonary Disorders" Adverse events that fall under the category of Appendix "Definition of Pulmonary Disorders" (as an adverse event) Patients with the onset of Patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA FILGT Code 10004018 (Bacterial infection) or 10039135 (Rickettsia infection)) Patients with the onset of f | | the field of "Drugs used for the prevention of infection" (If more than one |
| combinations "Drugs used for the prevention of infection" (If more than one trimethoprim-sulfamethoxazole combinations are used in the same patient, it will be counted as one patient.) Other prophylactics against infections Any drug entered in the field of "Drugs used for the prevention of infections infection" other than prophylactics against infections listed above (If more than one other prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral metror disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders in the field of "Adverse events: [1] Peripheral nerve disorders in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse events) Pulmonary disorders (Adverse events that fall under the category of Appendix "Definition of Pulmonary Disorders" MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA PLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia i | | antivirals are used in the same patient, it will be counted as one patient.) |
| trimethoprim-sulfamethoxazole combinations are used in the same patient, it will be counted as one patient.) Other prophylactics against infections Any drug entered in the field of "Drugs used for the prevention of infections infection" other than prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral motor neuropathy (as an adverse event) Peripheral motor neuropathy (as an adverse event) Adverse events with "Sensory neuropathy" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders in the field of "Adverse events" in the field. Peripheral motor neuropathy (as an adverse event) Adverse events with "Motor neuropathy" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of Pulmonary Disorders" Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA PT Code 100041881 (Infections and infestations) Patients with the onset of MedDRA PT. Code 100041881 (Infections and infestation) Patients with adverse drug reactions that fall under the category of MedDRA PT. Gode 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection | Trimethoprim-sulfamethoxazole | Drugs with YJ Code being 62901000 that are entered in the field of |
| it will be counted as one patient.) Other prophylactics against infections Any drug entered in the field of "Drugs used for the prevention of infections infections infection" other than prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders of data entered in "Symptoms" in the field. Pulmonary disorders (as an adverse event) Pulmonary Disorders (as adverse events) Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 1004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | combinations | "Drugs used for the prevention of infection" (If more than one |
| Other prophylactics against infections Any drug entered in the field of "Drugs used for the prevention of infections infections infection" other than prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders of data entered in "Symptoms" in the field. Pulmonary disorders (as an adverse event) Adverse events that fall under the category of Appendix "Definition of (as an adverse events) Pulmonary Disorders" (as an adverse event) Pulmonary Disorders" (as an adverse event) Pulmonary Disorders" (as an adverse event) Pulmonary Disorders (as an adverse event) Pulmonary Disor | | trimethoprim-sulfamethoxazole combinations are used in the same patient, |
| infections infection other than prophylactics against infections listed above (If more than one other prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Adverse events with "Sensory neuropathy" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Adverse events with "Motor neuropathy" entered in the "Category of peripheral nerve disorders" in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of (as adverse events) Pulmonary Disorders" Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of Patients with adverse drug reactions that fall under the category of infection MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) | | it will be counted as one patient.) |
| than one other prophylactics against infections are used in the same patient, it will be counted as one patient.) Peripheral sensory neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of Pulmonary Disorders" Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal | Other prophylactics against | Any drug entered in the field of "Drugs used for the prevention of |
| Peripheral sensory neuropathy (as an adverse event) Peripheral sensory neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of (as adverse events) Pulmonary Disorders" Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of Patients with adverse drug reactions that fall under the category of medDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | infections | infection" other than prophylactics against infections listed above (If more |
| Peripheral sensory neuropathy (as an adverse event) Adverse events with "Sensory neuropathy" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of (as adverse events) Pulmonary Disorders" Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA SOC Code 10021881 (Infections and infestations) Patients with adverse drug reactions that fall under the category of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | | than one other prophylactics against infections are used in the same |
| (as an adverse event) peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of (as adverse events) Pulmonary Disorders" Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | | patient, it will be counted as one patient.) |
| nerve disorders] in the case report form. MedDRA PT Code 10034620 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse events) Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of infection Patients with adverse drug reactions that fall under the category of MedDRA PI Code 10021881 (Infections and infestations) Patients with the onset of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection)) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of MedDRA HLGT Code 10004018 (Bacterial infection) or 10039135 (Rickettsia infection)) Patients with the onset of fungal | Peripheral sensory neuropathy | Adverse events with "Sensory neuropathy" entered in the "Category of |
| should be assigned regardless of data entered in "Symptoms" in the field. Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders" in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of Pulmonary Disorders" Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of Patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | (as an adverse event) | peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral |
| Peripheral motor neuropathy (as an adverse event) Peripheral nerve disorders' in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders' in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse events) Adverse events that fall under the category of Appendix "Definition of Pulmonary Disorders" MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | | nerve disorders] in the case report form. MedDRA PT Code 10034620 |
| (as an adverse event) peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse events) Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | | should be assigned regardless of data entered in "Symptoms" in the field. |
| nerve disorders] in the case report form. MedDRA PT Code 10034580 should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse events) Adverse events that fall under the category of Appendix "Definition of (as adverse events) Pulmonary Disorders" Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of infection MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | Peripheral motor neuropathy | Adverse events with "Motor neuropathy" entered in the "Category of |
| should be assigned regardless of data entered in "Symptoms" in the field. Peripheral neuropathy (as an adverse event) disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of (as adverse events) Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of infection MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | (as an adverse event) | peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral |
| Peripheral neuropathy (as an adverse event) Adverse events with "Other" entered in the "Category of peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of (as adverse events) Infusion reaction MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of Infection Patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | | nerve disorders] in the case report form. MedDRA PT Code 10034580 |
| disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders Adverse events that fall under the category of Appendix "Definition of Pulmonary Disorders" Infusion reaction (as an adverse event) MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | | should be assigned regardless of data entered in "Symptoms" in the field. |
| in the case report form. MedDRA PT Code 10029331 should be assigned, regardless of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse events) Infusion reaction (as an adverse event) MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of infection Patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | Peripheral neuropathy | Adverse events with "Other" entered in the "Category of peripheral nerve |
| regardless of data entered in "Symptoms" in the field. Pulmonary disorders (as adverse events) Infusion reaction (as an adverse event) MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of infection Patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | (as an adverse event) | disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] |
| Pulmonary disorders (as adverse events) Infusion reaction (as an adverse event) Patients with the onset of infection Patients with the onset of bacterial infection Patients with adverse drug reactions that fall under the category of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | | in the case report form. MedDRA PT Code 10029331 should be assigned, |
| (as adverse events) Infusion reaction (as an adverse event) Patients with the onset of infection Patients with the onset of bacterial infection Patients with the onset of bacterial infection Patients with the onset of Patients with adverse drug reactions that fall under the category of bacterial infection Patients with adverse drug reactions that fall under the category of bacterial infection Patients with adverse drug reactions that fall under the category of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with adverse drug reactions that fall under the category of | | regardless of data entered in "Symptoms" in the field. |
| Infusion reaction (as an adverse event) Patients with the onset of infection Patients with the onset of bacterial infection MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of Patients with adverse drug reactions that fall under the category of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | Pulmonary disorders | Adverse events that fall under the category of Appendix "Definition of |
| (as an adverse event) regardless of symptoms entered in the field of "Adverse events: [4] Infusion reaction." Patients with the onset of Patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of Patients with adverse drug reactions that fall under the category of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | (as adverse events) | Pulmonary Disorders" |
| Patients with the onset of Patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of Patients with adverse drug reactions that fall under the category of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | Infusion reaction | MedDRA PT Code 10051792 (Infusion related reaction) will be assigned, |
| Patients with the onset of infection Patients with adverse drug reactions that fall under the category of MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of Patients with adverse drug reactions that fall under the category of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | (as an adverse event) | regardless of symptoms entered in the field of "Adverse events: [4] |
| infection MedDRA SOC Code 10021881 (Infections and infestations) Patients with the onset of Patients with adverse drug reactions that fall under the category of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | | Infusion reaction." |
| Patients with the onset of bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | Patients with the onset of | Patients with adverse drug reactions that fall under the category of |
| bacterial infection MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | infection | MedDRA SOC Code 10021881 (Infections and infestations) |
| (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | Patients with the onset of | Patients with adverse drug reactions that fall under the category of |
| (Rickettsia infection) Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | bacterial infection | MedDRA HLGT Code 10004018 (Bacterial infection), 10008555 |
| Patients with the onset of fungal Patients with adverse drug reactions that fall under the category of | | (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 |
| | | (Rickettsia infection) |
| infection MedDRA HLGT Code 10017528 (Fungal infection) | Patients with the onset of fungal | Patients with adverse drug reactions that fall under the category of |
| | infection | MedDRA HLGT Code 10017528 (Fungal infection) |

| Term | | Definition |
|---|---|---|
| Patients with the onset of viral | Patients with adverse drug reactions that fall under the category of | |
| infection | MedDRA HLGT Code 10047438 (Viral infection) | |
| Age | If the month and day of the initial dose of Adcetris is < the month and day | |
| | of birth, the patient's age will be calculated using the following formula: | |
| | Year of the initial dose of Adcetris – year of birth – 1. | |
| | If the month and d | ay of the initial dose of Adcetris is ≥ the month and day |
| | of birth, the patien | t's age will be calculated using the following formula: |
| | Year of the initial | dose of Adcetris – year of birth. |
| | If the month and d | ay of birth are unknown, they should be "January 1," |
| | and if the day of b | irth is unknown, it should the first day of the month. |
| | If the day, month, | and year of birth are unknown but the patient's age is |
| | known, the patient | s's age should be used as it is. |
| BMI | BMI should be cal | culated using the following formula: Weight |
| | (kg)/(0.0001 × hei | ght (cm) × height (cm). The obtained value should be |
| | rounded off to one | decimal place. |
| Disease duration | The disease duration | on should be calculated using the following formula: |
| | ["Date of the initial | al dose of Adcetris" - "date of diagnosis of Hodgkin's or |
| | anaplastic large-ce | ell lymphoma" +1]/365.25. |
| | The day of diagno | sis should be the first day of the month provided. If the |
| | month of diagnosis is unknown, the date of diagnosis should be "January | |
| | 1st" of the year provided. | |
| Mean dose of Adcetris | Is calculated as the total value of each dose of Adcetris given at each | |
| | treatment cycle divided by the number of cycles. | |
| Dose of Adcetris per 3 weeks | Is calculated using the following formula: Total "dose of Adcetris"/(["date | |
| | of the last dose of | Adcetris" - "date of the initial dose of Adcetris" + |
| | 21)/21]. | |
| | If only 1 cycle of t | reatment is given, the "date of the last dose of Adcetris" |
| | and the "date of th | e initial dose of Adcetris" should be regarded as the |
| | same. | |
| Degree of decreased neutrophil | The neutrophil count at baseline will be classified as shown in the table | |
| count at baseline | below. If the neutr | ophil count at baseline is missing, the degree of the |
| | neutrophil count a | t baseline should be handled as missing: |
| | No decrease | ≥2,000 /mm <sup>3</sup> |
| | Grade 1 | ≥1,500 to <2,000 /mm <sup>3</sup> |
| | Grade 2 $\geq 1,000 \text{ to } < 1,500 \text{ /mm}^3$ | |
| | Grade 3 | ≥500 to <1,000 /mm <sup>3</sup> |
| | Grade 4 | <500 /mm <sup>3</sup> |
| Days from the month of the | Is calculated using the following formula: date of the initial dose of | |
| completion of the final regimen | Adcetris – date of | of the completion of the final regimen of prior drug |

| Term | Definition |
|---|---|
| of prior drug therapy to the date | therapy + 1. |
| of 1 cycle of treatment with | If the month of "the completion of the final regimen of prior drug therapy" |
| Adcetris | is missing, the date of the completion of the final regimen of prior drug |
| | therapy should be handled as missing. |
| Days from the month of the | Is calculated using the following formula: date of the initial dose of |
| completion of the most recent | Adcetris – date of the completion of the most recent prior radiotherapy + |
| prior radiotherapy to the date of | 1. |
| 1 cycle of treatment with | If the month of "the completion of the most recent prior radiotherapy" is |
| Adcetris | missing, the date of the completion of the most recent prior radiotherapy |
| | should be handled as missing. |
| Days from the date of the last | For patients with post-baseline hematopoietic stem cell transplantation |
| dose of Adcetris to | (autologous), this data item will be calculated using the following formula: |
| hematopoietic stem cell | date of post-baseline hematopoietic stem cell transplantation (autologous) |
| transplantation (autologous) | - date of the last dose of Adcetris + 1. If the date of post-baseline |
| (Post-baseline hematopoietic | hematopoietic stem cell transplantation (autologous) is missing, this data |
| stem cell transplantation: | item should be handled as missing. |
| autologous) | For patients with no post-baseline hematopoietic stem cell transplantation |
| | (autologous), this data item should be handled as missing. |
| Duration of treatment with | For patients with post-baseline hematopoietic stem cell transplantation |
| Adcetris prior to hematopoietic | (autologous), this data item will be calculated using the following formula: |
| stem cell transplantation | date of the last dose of Adcetris – date of the initial dose of Adcetris + 1. If |
| (autologous) | the date of post-baseline hematopoietic stem cell transplantation |
| (Post-baseline hematopoietic | (autologous) is missing, this data item should be handled as missing. |
| stem cell transplantation: | For patients with no post-baseline hematopoietic stem cell transplantation |
| autologous) | (autologous), this data item should be handled as missing. |
| Days from the date of the last | For patients with post-baseline hematopoietic stem cell transplantation |
| dose of Adcetris to | (homologous), this data item will be calculated using the following |
| hematopoietic stem cell | formula: date of hematopoietic stem cell transplantation (homologous) – |
| transplantation (homologous) | date of the last dose of Adcetris + 1. If the date of post-baseline |
| (Post-baseline hematopoietic | hematopoietic stem cell transplantation (homologous) is missing, this data |
| stem cell transplantation: | item should be handled as missing. |
| homologous) | For patients with no post-baseline hematopoietic stem cell transplantation |
| | (homologous), this data item should be handled as missing. |
| Duration of treatment with | For patients with post-baseline hematopoietic stem cell transplantation |
| Adcetris prior to hematopoietic | (homologous), this data item will be calculated using the following |
| stem cell transplantation | formula: date of the last dose of Adcetris – date of the initial dose of |
| (homologous) | Adcetris + 1. If the date of post-baseline hematopoietic stem cell |
| (Post-baseline hematopoietic | transplantation (homologous) is missing, this data item should be handled |
| stem cell transplantation: | as missing. |

| Term | Definition |
|---|---|
| homologous) | For patients with no post-baseline hematopoietic stem cell transplantation |
| | (homologous), this data item should be handled as missing. |
| Date of the final observation | "Date of the final observation" in the case report form |
| | If not provided, the most recent date entered in the case report form should |
| | be used. |
| Summary statistics | Number of patients, mean, standard deviation, minimum, 25th percentile, |
| | median, 75th percentile, and maximum. |
| Overall survival | Time to the date of death from any cause after the date of the initial dose |
| | of Adcetris. Surviving patients will be censored on the date of survival |
| | confirmation. |
| | The date of outcome of an adverse event with "Died/fetal" recorded in the |
| | Outcome field will be used as the date of death, and the final observation |
| | date will be used as the date of survival confirmation. |
| | The overall survival (date of death or survival confirmation) = date of |
| | death or survival confirmation – date of the initial dose of Adcetris+1 |
| 1 year | One year is defined as 365.25 days. |
| 1 month | One month is defined as 30.4375 days. |

#### 1.2 Display digits

| Term | Definition |
|---|---|
| Percentage (%) | Percentage of patients with or percentage of adverse events or adverse drug |
| | reactions, etc.: |
| | The obtained value should be rounded off to two decimal places. |
| | Other: |
| | The obtained value should be rounded off to one decimal place. |
| Summary statistics | Mean, median, 25th percentile and 75th percentile: |
| | The raw data should be rounded off to one decimal place. |
| | Standard deviation: |
| | The raw data should be rounded off to two decimal places. |
| | Minimum and maximum: |
| | The same display digit as the one used for the corresponding data will be used. |
| P value | The obtained value should be rounded down to three decimal places. |
| | If the value is less than 0.001 after rounding down to three decimal places, it |
| | should be displayed as "p<0.001." |

#### 1.3 Level of significance and confidence coefficient

Level of significance: Two-sided 5% Confidence coefficient: Two-sided 95%

#### 1.4 Handling of test data

Test data will be handled according to the criteria shown below. If there are multiple data for the same criterion, the one with the test date being closest to the date of protocol-specified assessment should be used. If there is no difference in the number of days from the date of protocol-specified assessment, the later value should be used.

The number of days after the date of the initial dose of Adcetris is defined as 1 for the date of the initial dose of Adcetris and 0 for the day before the date of the initial dose of Adcetris.

| Time point for testing | Date of protocol-specified assessment | Acceptable time window |
|---|---|---|
| At the initial dose of | Date of the initial dose of Adcetris | -15 days to the d ate of the initial dose of |
| Adcetris | | Adcetris |
| After 1 cycle | • If Cycle 2 is initiated: Date of Cycle | • If Cycle 2 is initiated: Date of Cycle 2 |
| | 2 | • If Cycle 2 is not initiated: 21 days after |
| | • If Cycle 2 is not initiated: 21 days | the date of the initial dose of Adcetris |
| | after the date of the initial dose of | |
| | Adcetris s | |

| Time point for testing | Date of protocol-specified assessment | Acceptable time window |
|---|---|---|
| After 2 cycles | • If Cycle 3 is initiated: Date of Cycle | If Cycle 3 is initiated: From the day |
| | 3 | after the date of Cycle 2 to the day of |
| | • If Cycle 3 is not initiated: 21 days | Cycle 3 |
| | after the date of Cycle 2 | • If Cycle 3 is not initiated: From the day |
| | | after the date of Cycle 2 to 21 days |
| | | after the date of Cycle 2 |
| After 3 cycles | • If Cycle 4 is initiated: Date of Cycle | If Cycle 4 is initiated: From the day |
| | 4 | after the date of Cycle 3 to the day of |
| | • If Cycle 4 is not initiated: 21 days | Cycle 4 |
| | after the date of Cycle 3 | • If Cycle 4 is not initiated: From the day |
| | | after the date of Cycle 3 to 21 days |
| | | after the date of Cycle 3 |
| After 4 cycles | • If Cycle 5 is initiated: Date of Cycle | If Cycle 5 is initiated: From the day |
| | 5 | after the date of Cycle 4 to the day of |
| | If Cycle 5 is not initiated: 21 days | Cycle 5 |
| | after the date of Cycle 4 | • If Cycle 5 is not initiated: From the day |
| | | after the date of Cycle 4 to 21 days |
| | | after the date of Cycle 4 |
| After 5 cycles | If Cycle 6 is initiated: Date of Cycle | If Cycle 6 is initiated: From the day |
| | 6 | after the date of Cycle 5 to the day of |
| | • If Cycle 6 is not initiated: 21 days | Cycle 6 |
| | after the date of Cycle 5 | • If Cycle 6 is not initiated: From the day |
| | | after the date of Cycle 5 to 21 days |
| | | after the date of Cycle 5 |
| After 6 cycles | • If Cycle 7 is initiated: Date of Cycle | If Cycle 7 is initiated: From the day |
| | 7 | after the date of Cycle 6 to the day of |
| | If Cycle 7 is not initiated: 21 days | Cycle 7 |
| | after the date of Cycle 6 | • If Cycle 7 is not initiated: From the day |
| | | after the date of Cycle 6 to 21 days |
| | | after the date of Cycle 6 |
| After 7 cycles | If Cycle 8 is initiated: Date of Cycle | • If Cycle 8 is initiated: From the day |
| | 8 | after the date of Cycle 7 to the day of |
| | If Cycle 8 is not initiated: 21 days | Cycle 8 |
| | after the date of Cycle 7 | If Cycle 8 is not initiated: From the day |
| | | after the date of Cycle 7 to 21 days |
| | | after the date of Cycle 7 |

| Time point for testing | Date of protocol-specified assessment | Acceptable time window |
|---|---|---|
| After 8 cycles | • If Cycle 9 is initiated: Date of Cycle | If Cycle 9 is initiated: From the day |
| | 9 | after the date of Cycle 8 to the day of |
| | • If Cycle 9 is not initiated: 21 days | Cycle 9 |
| | after the date of Cycle 8 | • If Cycle 9 is not initiated: From the day |
| | | after the date of Cycle 8 to 21 days |
| | | after the date of Cycle 8 |
| After 9 cycles | If Cycle 10 is initiated: Date of | • If Cycle 10 is initiated: From the day |
| | Cycle 10 | after the date of Cycle 9 to the day of |
| | If Cycle 10 is not initiated: 21 days | Cycle 10 |
| | after the date of Cycle 9 | • If Cycle 10 is not initiated: From the |
| | | day after the date of Cycle 9 to 21 days |
| | | after the date of Cycle 9 |
| After 10 cycles | If Cycle 11 is initiated: Date of | If Cycle 11 is initiated: From the day |
| | Cycle 11 | after the date of Cycle 10 to the day of |
| | If Cycle 11 is not initiated: 21 days | Cycle 11 |
| | after the date of Cycle 10 | • If Cycle 11 is not initiated: From the |
| | | day after the date of Cycle 10 to 21 |
| | | days after the date of Cycle 10 |
| After 11 cycles | If Cycle 12 is initiated: Date of | • If Cycle 12 is initiated: From the day |
| | Cycle 12 | after the date of Cycle 11 to the day of |
| | If Cycle 12 is not initiated: 21 days | Cycle 12 |
| | after the date of Cycle 11 | • If Cycle 12 is not initiated: From the |
| | | day after the date of Cycle 11 to 21 |
| | | days after the date of Cycle 11 |
| After 12 cycles | If Cycle 13 is initiated: Date of | • If Cycle 13 is initiated: From the day |
| | Cycle 13 | after the date of Cycle 12 to the day of |
| | • If Cycle 13 is not initiated: 21 days | Cycle 13 |
| | after the date of Cycle 12 | • If Cycle 13 is not initiated: From the |
| | | day after the date of Cycle 12 to 21 |
| | | days after the date of Cycle 12 |
| After 13 cycles | If Cycle 14 is initiated: Date of | • If Cycle 14 is initiated: From the day |
| | Cycle 14 | after the date of Cycle 13 to the day of |
| | If Cycle 14 is not initiated: 21 days | Cycle 14 |
| | after the date of Cycle 13 | • If Cycle 14 is not initiated: From the |
| | | day after the date of Cycle 13 to 21 |
| | | days after the date of Cycle 13 |

| Time point for testing | Date of protocol-specified assessment | Acceptable time window |
|---|---|---|
| After 14 cycles | If Cycle 15 is initiated: Date of | If Cycle 15 is initiated: From the day |
| | Cycle 15 | after the date of Cycle 14 to the day of |
| | If Cycle 15 is not initiated: 21 days | Cycle 15 |
| | after the date of Cycle 14 | • If Cycle 15 is not initiated: From the |
| | | day after the date of Cycle 14 to 21 |
| | | days after the date of Cycle 14 |
| After 15 cycles | If Cycle 16 is initiated: Date of | If Cycle 16 is initiated: From the day |
| | Cycle 16 | after the date of Cycle 15 to the day of |
| | If Cycle 16 is not initiated: 21 days | Cycle 16 |
| | after the date of Cycle 15 | If Cycle 16 is not initiated: From the |
| | | day after the date of Cycle 15 to 21 |
| | | days after the date of Cycle 15 |

#### 1.5 Handling of missing data

- As a general rule, missing data will not be imputed.
- In the analysis of the frequency qualitative variables, missing data will be handles as "unknown." In the analysis of summary statistics of quantitative variables, missing data will be excluded.

#### 1.6 Others

- In the analysis for the preparation of documents for the Final Survey Report (final analysis), MedDRA version 19.1 will be used for adverse events, concurrent illness, and past history.
- If a patient has multiple data for a single laboratory test and date of testing, the mean value will be calculated for the analysis of laboratory test results.
- If the date of diagnostic imaging for the assessment of the best response is missing, it will be handled as missing.

#### 2.0 Patient Disposition (Patient Disposition Diagram)

(1) Analysis set to be used

Patients registered

#### (2) Data to be analyzed

Data to be analyzed includes the numbers of patients registered, institutions with patients registered, patients whose case report forms are available/not available, fixed/non-fixed patients, patients included in/excluded from the safety analysis set, and patients included in/excluded from the efficacy analysis set.

For the number of institutions with patients registered, the same institutions with different departments should not be counted more than once.

For patients whose case report forms are not available, the number of patients by reason for unavailability will be calculated. The reason for unavailability should be transfer or health problems of the investigator or other.

For patients included in safety evaluation, the number of patients by primary disease (Hodgkin's or anaplastic large-cell lymphoma or other) and the overall number of patients will be calculated. For patients included in efficacy evaluation, the number of patients by primary disease (Hodgkin's or anaplastic large-cell lymphoma) and the overall number of patients will be calculated.

For patients excluded from the safety/efficacy analysis set, the number of patients by reason for exclusion will be calculated, and a patient list will be generated.

The selection of patients to be included in safety evaluation and those who are to be included in efficacy evaluation will be made as shown below:

| Criterion | Safety | Efficacy |
|----------------------------------------------|------------|------------|
| Citterion | evaluation | evaluation |
| Adcetris has never been administered [found | × | × |
| afterwards] | | |
| No data for safety evaluation (data to | × | × |
| determine the presence or absence of adverse | | |
| events) are available | | |
| Non-primary disease | 0 | × |

o: Included, ×: Excluded

#### (3) Figure/table number

Figure 2.0 and Table 2.0

#### 3.0 Patient Demographics and Baseline Characteristics

#### 3.1 Patient Demographics and Baseline Characteristics

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the categories below, and the frequency will be calculated. In addition, summary statistics of continuous variable will be calculated:

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | <18 years, 18 to 39 years, 40 to 64 years, 65 to 74 years, or ≥75 years |
| | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| Diagnosis | Hodgkin's or anaplastic large-cell lymphoma or other |
| Status | Relapsed/refractory, or new-onset |
| CD30 | Positive, negative, or not measured |
| Site(s) of involvement | Lymph node, spleen, liver, lung, bone, central nerve, bone marrow, skin, and/or other |
| ALK (for patients | |
| with anaplastic | Positive, negative, or unknown |
| large-cell lymphoma) | |
| Clinical stage | I, II, III, IV, or unknown |
| B symptoms | Absent or present |
| ECOG Performance Status | 0, 1, 2, 3, or 4 |
| Therapeutic category | Outpatient, inpatient, or unkown |
| Hypersensitivity disposition | Absent, present, or unknown |
| Specific hypersensitivity disposition(s) | Medications, food allergy, and/or other |
| HCV antibody | Negative, positive, or unknown |
| HBs antigen | Negative, positive, or unknown |
| HBs antibody | Negative, positive, or unknown |
| HBV DNA | Negative, positive, or unknown |
| Past history of pulmonary disorders | Absent or present |
| Concurrent pulmonary disorders | Absent or present |

| Data item | Category |
|---|---|
| Past history of | Absort or present |
| malignant tumours | Absent or present |
| Concurrent malignant | Absent or present |
| tumours | About of present |
| Past history (other | |
| than pulmonary | Absent, present, or unknown |
| disorders and | Absent, present, of unknown |
| malignant tumours) | |
| Concurrent illness | |
| (other than pulmonary | Absent or present |
| disorders and | About of present |
| malignant tumours) | |
| Specific concurrent | |
| illness(es) (other than | Diabetes mellitus, hypertension, dyslipidaemia, hyperuricaemia, |
| pulmonary disorders | hepatic disease(s), renal disease(s), infections, peripheral nerve |
| and malignant | disorders, and/or other |
| tumours) | disorders, and/or other |
| Past history (other | |
| than pulmonary | Absort present or unknown |
| disorders and | Absent, present, or unknown |
| malignant tumours) | |
| Concurrent hepatic | Absent or present |
| disorders | Absent of present |
| Grade of hepatic | |
| disorder | None, Grade 1, Grade 2, ≥Grade 3, or unknown |
| (Grade based on AST | None, Grade 1, Grade 2, 2Grade 3, or unknown |
| and ALT levels) | |
| Concurrent renal | Absent or present |
| disorders | Prosent of present |
| Grade of renal | |
| disorder | None, Grade 1, Grade 2, ≥Grade 3, or unknown |
| (Grade based on | 11000, Grade 1, Grade 2, Corade 3, or diskilowii |
| serum creatinine) | |
| Concurrent peripheral | None, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |
| neuropathy | Trone, Grade 1, Grade 2, Grade 3, Grade 4, Or unknown |
| Weight | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, or ≥70 kg |
| BMI | $<18.5 \text{ kg/m}^2$ , $<18.5 \text{ to } 25 \text{ kg/m}^2$ , $<25 \text{ to } 30 \text{ kg/m}^2$ , or $\ge 30 \text{ kg/m}^2$ |
| Smoking history | Never, current, past, or unknown |

| Data item | Category |
|---|---|
| Prior drug therapy | Absent or present |
| Prior drug therapy | ABVD, CHOP, and/or other |
| regimen(s) | (If more than one drug therapies in the same regimen is used in the |
| | same patient, it will be counted as one patient.) |
| Number of prior drug | |
| therapy regimens | - |
| Days from the month | |
| of the completion of | |
| the final regimen of | |
| prior drug therapy to | |
| the date of 1 cycle of | - |
| treatment with | |
| Adcetris | |
| (Prior drug therapy: | |
| Yes) | |
| Prior radiotherapy | Absent or present |
| Days from the month | |
| of the completion of | |
| the most recent prior | |
| radiotherapy to the | |
| date of 1 cycle of | - |
| treatment with | |
| Adcetris | |
| (Prior radiotherapy: | |
| yes) | |
| Prior hematopoietic | Absent, present (autologous), present (homologous), present |
| stem cell | (autologous and homologous), or unknown |
| transplantation | (autologous and nomologous), or unknown |
| Other prior therapies | Absent, present, or unknown |
| Pregnancy during the | |
| observation period | Absent or present |
| (for females only) | |

Tables 3-1 to 3.1-3

#### 3.2 Prior drug therapy (details)

#### (1) Analysis sets to be used

Patients included in safety evaluation and patients included in safety evaluation (Hodgkin's

lymphoma) or patients included in safety evaluation (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For prior drug therapy, patients will be stratified into the categories below, and the frequency will be calculated. The percentage of prior drug therapy will be calculated using the number of patients with prior drug therapy as the denominator. In addition, specific prior drug therapies and their percentages will be presented in a pie chart:

| Data item | Category |
|---|---|
| | ABVD, CHOP, BEACOPP, C-MOPP, CHASE, CHOEP, DeVIC, |
| | EPOCH, ESHAP, GCD, GDP, GEM, ICE, THP-COP, or other |
| Specific prior drug | (If more than one drug therapies in the same regimen is used in the |
| therapy(ies) | same patient, it will be counted as one patient.) |
| | Prior drug therapies should be listed in descending order of the number |
| | of patients. However, "Other" should be listed lastly. |

#### (3) Figure/table number

Tables 3.2-1 to 3.2-3 and Figures 3.2-1 to 3.2-3

#### 4.0 Treatment Given

#### 4.1 Treatment given

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories below, and the frequency will be calculated. In addition, summary statistics of continuous variable will be calculated:

| Data item | Category |
|---|---|
| Initial dose of | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or >1.8 |
| Adcetris | mg/kg |
| Mean dose of Adcetris | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or >1.8 |
| Weari dose of Adcerrs | mg/kg |
| Dose of Adcetris per 3 | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or >1.8 |
| weeks | mg/kg |
| Duration of treatment | $1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, \text{ or } \ge 17 \text{ cycles}$ |
| with Adcetris | 1, 2, 3, 4, 3, 0, 7, 8, 9, 10, 11, 12, 13, 14, 13, 10, 01 ≥17 cycles |
| Reason(s) for | |
| discontinuation of | Treatment goal achieved, adverse event(s), lost to follow-up, transfer to |
| Adcetris | another hospital, pregnancy, inadequate response, and/or other |
| Post-baseline | |
| hematopoietic stem | Absent, present, or unknown |
| cell transplantation | |
| Type of post-baseline | |
| hematopoietic stem | Autologous or homologous |
| cell transplantation | |
| Days from the date of | |
| the last dose of | |
| Adcetris to | |
| hematopoietic stem | |
| cell transplantation | |
| (autologous) | |
| (Post-baseline | |
| hematopoietic stem | |
| cell transplantation: | |
| autologous) | |
| Duration of treatment | |
| with Adcetris prior to | |

| hematopoietic stem | |
|---|---|
| cell transplantation | |
| (autologous) | |
| (Post-baseline | |
| hematopoietic stem | |
| cell transplantation: | |
| autologous) | |
| Days from the date of | |
| the last dose of | |
| Adcetris to | |
| hematopoietic stem | |
| cell transplantation | |
| (homologous) | - |
| (Post-baseline | |
| hematopoietic stem | |
| cell transplantation: | |
| homologous) | |
| Duration of treatment | |
| with Adcetris prior to | |
| hematopoietic stem | |
| cell transplantation | |
| (homologous) | - |
| (Post-baseline | |
| hematopoietic stem | |
| cell transplantation: | |
| homologous) | |
| Drug(s) other than | |
| Adcetris used for the | Alasant an annual |
| treatment of the | Absent or present |
| primary disease | |
| Drug(s) used for the | |
| prevention of | Absent or present |
| infection | |
| Specific drug(s) used | Antibiotics/synthetic antibacterial agents, antifungals, antivirals, |
| for the prevention of | trimethoprim-sulfamethoxazole combinations, and/or other |
| infection | prophylactics against infections |
| 1 | ı |

Tables 4.1-1 to 4.1-3

#### 4.2 Premedication to prevent infusion reaction

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each cycle, patients will be stratified into the following categories, and the frequency will be calculated:

| Data item | Category |
|---|---|
| Premedication to | |
| prevent infusion | Absent, present, or unknown |
| reaction | |
| Specific | |
| premedication(s) used | A |
| to prevent infusion | Acetaminophen, antihistamines, and/or corticosteroids |
| reaction | |
| Specific | |
| premedication(s) used | Acetaminophen, antihistamines, corticosteroids, acetaminophen + |
| to prevent infusion | antihistamines, acetaminophen + corticosteroids, antihistamines + |
| reaction | corticosteroids, or acetaminophen + antihistamines + corticosteroids |
| (in each patient) | |

#### (3) Figure/table number

Tables 4.2-1 to 4.2-3

#### 4.3 Patient demographics and baseline characteristics by initial dose of Adcetris

#### (1) Analysis sets to be used

Patients included in safety evaluation and patients included in safety evaluation (Hodgkin's lymphoma) or patients included in safety evaluation (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the frequency will be calculated by initial dose of Adcetris (<1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg):

| Data item | Category |
|---|---|
| Age | <18 years, 18 to 39 years, 40 to 64 years, 65 to 74 years, or ≥75 years |
| ECOG Performance | 0, 1, 2, 3, or 4 |
| Status | |
| Concurrent hepatic | Absort on procent |
| disorders | Absent or present |
| Grade of hepatic | |
| disorder | None, Grade 1, Grade 2, ≥Grade 3, or unknown |
| (Grade based on AST | |

| Data item | Category |
|-----------------------|------------------------------------------------------|
| and ALT levels) | |
| Concurrent renal | A become an appropriate |
| disorders | Absent or present |
| Grade of renal | |
| disorder | None, Grade 1, Grade 2, ≥Grade 3, or unknown |
| (Grade based on | |
| serum creatinine) | |
| Concurrent infection | Absent or present |
| Concurrent peripheral | None, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |
| nerve disorder | |

Tables 4.3-1 to 4.3-3

#### 5.0 Safety Analysis

#### 5.1 Occurrences of adverse events and adverse drug reactions/infections

#### 5.1.1 Occurrence of adverse events

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

Data listed below will be analyzed.

For data entered in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form, MedDRA PT Code for peripheral sensory neuropathy, peripheral motor neuropathy, or peripheral neuropathy should be assigned, regardless of data entered in "Symptoms" field (see Section 1.2, the same applies hereinafter).

MedDRA PT Code for "Infusion related reaction" should be assigned to the field of "Adverse events: [4] Infusion reaction" in the case report form, regardless of data entered in "Symptoms" field (see Section 1.2, the same applies hereinafter).

Neutrophil count decreased (PT Code 10029366) will be replaced by Neutropenia (PT Code 10029354), Lymphocyte count decreased (PT Code 10025256) by Lymphopenia (PT Code 10025327), White blood cell count decreased (PT Code 10047942) by Leukopenia (PT Code 10024384), and Platelet count decreased (PT Code 10035528) by Thrombocytopenia (PT Code 10043554) (the same applies hereinafter).

| Data item | Data to be analyzed |
|---|---|
| Number of patients with adverse events | Number of patients experiencing adverse events |
| Number of adverse events | Number of adverse events observed. If the same patient has multiple occurrences of the same adverse event (PT), the total number of occurrences will be calculated. |
| Percentage of patients with adverse events | Is calculated using the following formula: number of patients with adverse events/number of patients included in the safety analysis set $\times$ 100. |
| Type of adverse events | The incidence of adverse events will be calculated by SOC and PT. For SOC, the number and percentage of patients with adverse events will be calculated. For PT, the number and percentage of adverse events will be calculated. SOCs will be presented in the internationally agreed order, and PTs will be presented in ascending order of HLGT and PT codes if their SOCs are "Investigations," and in ascending order of PT code otherwise. If the same patient has multiple occurrences of the same adverse event (PT), the event will be counted once per patient. |

Tables 5.1-1 to 5.1.1-3

#### 5.1.2 Occurrence of adverse drug reactions/infections

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

Data listed below will be analyzed.

| Data item | Data to be analyzed |
|---|---|
| Number of patients with adverse drug reactions, etc. | Number of patients experiencing adverse drug reactions, etc. |
| Number of adverse drug reactions, etc. | Number of adverse drug reactions, etc., observed. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the total number of occurrences will be calculated. |
| Percentage of patients with adverse drug reactions, etc. | Is calculated using the following formula: number of patients with adverse drug reactions, etc./number of patients included in the safety analysis set $\times$ 100. |
| Type of adverse drug reactions, etc. | The incidence of adverse drug reactions, etc., will be calculated by SOC and PT. For SOC, the number and percentage of patients with adverse drug reactions, etc., will be calculated. For PT, the number and percentage of adverse drug reactions, etc., will be calculated. SOCs will be presented in the internationally agreed order, and PTs will be presented in ascending order of HLGT and PT codes if their SOCs are "Investigations," and in ascending order of PT code otherwise. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the reaction will be counted once per patient. |

#### (3) Figure/table number

Tables 5.1-2 to 5.1.2-3

- 5.2 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrences of adverse events and adverse drug reactions/infections by outcome
  - 5.2.1 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrence of adverse events by outcome
    - (1) Analysis sets to be used

      Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic
    - (2) Data to be analyzed

large-cell lymphoma)

For each data item, patients will be stratified into the following categories, and the type of adverse events will be analyzed:

| Data item | Category |
|---|---|
| Seriousness | Serious or non-serious |
| CTCAE Grade (the worst one) | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| Time of onset | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, ≥337 days, or unknown |
| | 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly using a 21-day time window thereafter), 316 to 336 days, ≥337 days, or unknown |
| Time to the worst grade | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, ≥337 days, or unknown 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly using a 21-day time window thereafter), 316 to 336 days, ≥337 days, or unknown |
| Outcome | Recovered/resolved, recovering/resolving, not recovered/not resolved, recovered/resolved with sequelae, died/fatal, unknown, or not provided |

The type of adverse events will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse events by SOC/PT |
| | Number of adverse events observed by SOC/PT |
| Number of adverse events, | If the same patient has multiple occurrences of the same adverse |
| etc. | event (PT), all these occurrences will be counted (i.e., the overlap |
| | should be reflected). |
| | The number of adverse events will be calculated by SOC and PT. |
| | SOCs will be presented in the internationally agreed order, and |
| | PTs will be presented in ascending order of HLGT and PT codes |
| | if their SOCs are "Investigations," and in ascending order of PT |
| Seriousness, CTCAE Grade | code otherwise. |
| (the worst one), time of | If the same patient has multiple occurrences of the same adverse |
| onset, time to the worst grade, and outcome | event (PT), the total number of occurrences will be calculated per |
| | category (for example, if the same patient has one episode of |
| | serious diarrhea and one episode of non-serious diarrhea, these |
| | events will be counted once for each category). If the same patient |
| | has multiple occurrences of the same adverse event classified into |
| | the same category, all these occurrences will be counted (i.e., the |
| | overlap should be reflected). |

Tables 5.2.1-1 to 5.2.1-3

#### 5.2.2 Occurrence of adverse events by CTCAE Grade (the worst one)

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse events will be analyzed:

| Data item | Category |
|------------------------|--------------------------------|
| CTCAE Grade (the worst | ≤Grade 2, ≥Grade 3, or unknown |
| one) | |

The type of adverse events will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Type of adverse events | The incidence of adverse events for each CTCAE grade (the |
| | worst one) will be calculated by SOC and PT. For SOC, the |
| | number and percentage of patients with adverse events will be |
| | calculated. For PT, the number and percentage of adverse events |
| | will be calculated. SOCs will be presented in the internationally |

agreed order, and PTs will be presented in ascending order of HLGT and PT codes if their SOCs are "Investigations," and in ascending order of PT code otherwise. The CTCAE grade (the worst one) is higher in the order of ≥Grade 3, ≤Grade 2, and unknown. If the same patient has multiple occurrences of the same adverse event (PT), the event with the highest CTCAE grade will be counted once per patient.

(3) Figure/table number

Tables 5.2.2-1 to 5.2.2-3

# 5.2.3 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrence of adverse drug reactions/infections by outcome

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse drug reactions, etc., will be analyzed:

| Data item | Category |
|---|---|
| Seriousness | Serious or non-serious |
| CTCAE Grade (the worst one) | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 |
| | days, 169 to 252 days, 253 to 336 days, ≥337 days, or unknown |
| Time of onset | 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly |
| | using a 21-day time window thereafter), 316 to 336 days, ≥337 |
| | days, or unknown |
| | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 |
| Time to the worst grade | days, 169 to 252 days, 253 to 336 days, ≥337 days, or unknown |
| | 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly |
| | using a 21-day time window thereafter), 316 to 336 days, ≥337 |
| | days, or unknown |
| Outcome | Recovered/resolved, recovering/resolving, not recovered/not |
| | resolved, recovered/resolved with sequelae, died/fatal, unknown, |
| | or not provided |

The type of adverse drug reactions, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse drug reactions, etc., by SOC/PT |
| | If the same patient has multiple occurrences of the same adverse |
| | drug reactions, etc. (PT), all these occurrences will be counted |
| | (i.e., the overlap should be reflected). |
| Number of adverse drug | Number of adverse drug reactions, etc., observed by SOC/PT |
| reactions, etc. | Number of adverse drug feactions, etc., observed by SOC/F1 |
| | The number of adverse drug reactions, etc., will be calculated by |
| Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and outcome | SOC and PT. SOCs will be presented in the internationally agreed |
| | order, and PTs will be presented in ascending order of HLGT and |
| | PT codes if their SOCs are "Investigations," and in ascending |
| | order of PT code otherwise. |
| | If the same patient has multiple occurrences of the same adverse |
| | drug reaction, etc. (PT), the total number of occurrences will be |

calculated per category (for example, if the same patient has one episode of serious diarrhea and one episode of non-serious diarrhea, these adverse drug reactions will be counted once for each category). If the same patient has multiple occurrences of the same adverse drug reaction, etc., classified into the same category, all these occurrences will be counted (i.e., the overlap should be reflected).

(3) Figure/table number

Tables 5.2.3-1 to 5.2.3-3

#### 5.2.4 Occurrence of adverse drug reactions/infections by CTCAE Grade (the worst one)

(1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse drug reactions, etc., will be analyzed:

| Data item | Category |
|------------------------|--------------------------------|
| CTCAE Grade (the worst | ≤Grade 2, ≥Grade 3, or unknown |
| one) | |

The type of adverse drug reactions, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| | The incidence of adverse drug reactions, etc., for each CTCAE |
| | grade (the worst one) will be calculated by SOC and PT. For |
| | SOC, the number and percentage of patients with drug reactions, |
| | etc., will be calculated. For PT, the number and percentage of |
| | drug reactions, etc., will be calculated. SOCs will be presented in |
| True of odvorce drue | the internationally agreed order, and PTs will be presented in |
| Type of adverse drug | ascending order of HLGT and PT codes if their SOCs are |
| reactions, etc. | "Investigations," and in ascending order of PT code otherwise. |
| | The CTCAE grade (the worst one) is higher in the order of |
| | ≥Grade 3, ≤Grade 2, and unknown. If the same patient has |
| | multiple occurrences of the same adverse drug reaction, etc. |
| | (PT), the reaction with the highest CTCAE grade will be counted |
| | once per patient. |

#### (3) Figure/table number

Tables 5.2.4-1 to 5.2.4-3

# 5.3 Percentage of patients with adverse drug reactions/infections by patient demographics and baseline characteristics and treatment given

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the percentage of patients with adverse drug reactions, etc. (with point estimate and 95% confidence interval) will be determined.

For categories associated and not associated with ranking, Fisher's exact and Mann-Whitney U tests, respectively, will be used. If there is a category of "unknown," it will be excluded to perform

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| ALK (for patients with | |
| anaplastic large-cell | Positive, negative, or unknown |
| lymphoma) | |
| Clinical stage | I, II, III, IV, or unknown |
| B symptoms | Absent or present |
| ECOG Performance Status | 0, 1, 2, 3, or 4 |
| Past history of pulmonary | |
| disorders | Absent or present |
| Concurrent pulmonary | |
| disorders | Absent or present |
| Past history of malignant | |
| tumours | Absent or present |
| Concurrent malignant | |
| tumours | Absent or present |
| Concurrent hepatic | |
| disorders | Absent or present |
| Grade of hepatic disorder | |
| (Grade based on AST and | None, Grade 1, Grade 2, ≥Grade 3, or unknown |
| ALT levels) | |
| Concurrent renal disorders | Absent or present |
| Grade of renal disorder | |
| (Grade based on serum | None, Grade 1, Grade 2, ≥Grade 3, or unknown |
| creatinine) | |
| Weight | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, or ≥70 kg |
| BMI | $<18.5 \text{ kg/m}^2$ , $<18.5 \text{ to } 25 \text{ kg/m}^2$ , $<25 \text{ to } 30 \text{ kg/m}^2$ , or $\ge 30 \text{ kg/m}^2$ |
| Smoking history | Never, current, past, or unknown |
| Prior drug therapy | Absent or present |
| Prior radiotherapy | Absent or present |
| Prior hematopoietic stem | Absent, present (autologous), present (homologous), present |
| cell transplantation | (autologous and homologous), or unknown |
| Initial dose of Adaptris | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or |
| Initial dose of Adcetris | >1.8 mg/kg |

| Data item | Category |
|---|---|
| Mean dose of Adcetris | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or |
| | >1.8 mg/kg |
| Dose of Adcetris per 3 | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or |
| weeks | >1.8 mg/kg |
| Drug(s) other than Adcetris | |
| used for the treatment of | Absent or present |
| the primary disease | |

Tables 5.3-1 to 5.3-3
#### 5.4 Occurrence of adverse drug reactions/infections by age group

(1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

(2) Data to be analyzed

The similar calculation as the one described in Section 5.1.2, will be performed by age group (<18 years, 18 to 64 years, 65 to 74 years, or  $\ge 75$  years).

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Tables 5.4-1 to 5.4-3

- 5.5 Occurrence of adverse drug reactions/infections by presence or absence and grade of concurrent hepatic disorder
  - (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

(2) Data to be analyzed

The similar calculation as the one described in Section 5.1.2, will be performed by presence or absence and grade of concurrent hepatic disorder.

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Tables 5.5-1 to 5.5-3

- 5.6 Occurrence of adverse drug reactions/infections by presence or absence and grade of concurrent renal disorder
  - (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

(2) Data to be analyzed

The similar calculation as the one described in Section 5.1.2, will be performed by presence or absence and grade of concurrent renal disorder

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Tables 5.6-1 to 5.6-3

#### 5.7 Occurrence of serious adverse events

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

### (2) Data to be analyzed

Data listed below will be analyzed.

| Data item | Data to be analyzed |
|---|---|
| Number of patients with serious adverse events | Number of patients experiencing serious adverse events |
| | Number of serious adverse events observed |
| Number of serious | If the same patient has multiple occurrences of the same serious |
| adverse events | adverse event (PT), the total number of occurrences will be |
| | calculated. |
| Percentage of patients | Is calculated using the following formula: number of patients with |
| with serious adverse | serious adverse events/number of patients included in the safety |
| events | analysis set × 100. |
| | The incidence of serious adverse events will be calculated by SOC and PT. |
| | For SOC, the number and percentage of patients with serious |
| | adverse events will be calculated. For PT, the number and |
| | percentage of serious adverse events will be calculated SOCs will |
| Type of serious adverse | be presented in the internationally agreed order, and PTs will be |
| events | presented in ascending order of HLGT and PT codes if their SOCs |
| | are "Investigations," and in ascending order of PT code otherwise. |
| | If the same patient has multiple occurrences of the same serious |
| | adverse event (PT), the event will be counted once per patient. |
| | For serious adverse events considered not related to Adcetris, the |
| | number of these events will be presented in ( ). |

# (3) Figure/table number

Tables 5.7-1 to 5.7-3

#### 5.8 Change in test data over time

#### 5.8.1 Change in laboratory test results over time

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

Summary statistics of red blood cell count, hemoglobin level, white blood cell count, neutrophil count, lymphocyte count, platelet count, total bilirubin, AST, ALT, LDH, BUN, and serum creatinine will be calculated at each test time point [at baseline, after 1 cycle, ... and after 15 cycles]. In addition, box plots of hemoglobin level, neutrophil count, lymphocyte count, and platelet count will be generated at each test time point.

#### (3) Figure/table number

Tables 5.8.1-1 to 5.8.1-3 and Figures 5.8.1-1 to 5.8.1-3

#### 5.9 Analysis of items of particular interest

#### 5.9.1 Occurrence of the adverse drug reaction of peripheral nerve disorder and infections

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

The incidence of peripheral nerve disorders considered related to Adcetris will be calculated for each CTCAE grade (the worst one) by symptom of peripheral nerve disorder (peripheral sensory neuropathy, peripheral motor neuropathy, or peripheral neuropathy) and PT (see Section 1.2 for the definition of symptoms of peripheral nerve disorders). For symptoms of peripheral nerve disorders, the number and percentage of patients with peripheral nerve disorder will be calculated. For PT, the number and percentage of peripheral nerve disorder will be calculated. PTs will be presented in ascending order of PT code.

The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple occurrences of the same symptom of peripheral nerve disorder or the same PT, the symptom of peripheral nerve disorder or PT with the highest CTCAE grade (the worst one) will be counted for the respective category once per patient:

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | |
| one) for peripheral nerve | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| disorders | |

#### (3) Figure/table number

Tables 5.9.1-1 to 5.9.1-3

# 5.9.2 Occurrence of peripheral nerve disorders considered related to Adcetris by patient demographics and baseline characteristics and treatment given

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item of patient demographics and baseline characteristics and treatment given, patients will be stratified into the categories below, and the incidence of peripheral nerve disorders considered related to Adcetris will be calculated by CTCAE Grade (the worst one). The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple occurrences of the same peripheral nerve disorder (PT), the peripheral nerve disorder with the highest CTCAE grade will be counted once for the category:

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | |
| one) of peripheral nerve | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| disorder | |

Items and categories of patient demographics and baseline characteristics and treatment given

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| ECOG Performance Status | 0, 1, 2, 3, or 4 |
| Concurrent peripheral nerve disorders | None, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |
| Weight | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, or ≥70 kg |
| Prior ABVD or CHOP | Absent or present |
| Prior radiotherapy | Absent or present |
| Prior hematopoietic stem | Absent, present (autologous), present (homologous), present |
| cell transplantation | (autologous and homologous), or unknown |
| Initial dose of Adcetris | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg |
| Mean dose of Adcetris | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg |
| Dose of Adcetris per 3 | <1.2 mg/kg, 1.2 mg/kg, >1.2 mg/kg to <1.8 mg/kg, 1.8 mg/kg, or |
| weeks | >1.8 mg/kg |
| Concurrent diabetes mellitus | Absent or present |

(3) Figure/table number

Tables 5.9.2-1 to 5.9.2-3

#### 5.9.3 Treatment with Adcetris at the onset of peripheral nerve disorders considered related to Adcetris

#### (1) Analysis sets to be used

Patients included in the safety analysis set and safety analysis set (Hodgkin's lymphoma) or safety analysis set (anaplastic large-cell lymphoma) who experience peripheral nerve disorders considered related to Adcetris

#### (2) Data to be analyzed

For each CTCAE Grade (the worst one) of peripheral nerve disorders considered related to Adcetris, patients will be stratified into the categories below, and the incidence of peripheral nerve disorders will be calculated. If the same patient has multiple occurrences of the same peripheral nerve disorder (PT), the total number of occurrences will be calculated per category (for example, if the same patient has one episode of peripheral nerve disorder requiring dose reduction and one episode of peripheral nerve disorder leading to treatment discontinuation, these episodes of peripheral nerve disorder will be counted once for each category). The percentage of peripheral nerve disorders for each category will be calculated using the number of peripheral nerve disorders for each CTCAE grade (the worst one) as the denominator.

For each data item, missing data will be handled as "not provided."

| Data item | Category |
|---|---|
| Action taken to Adcetris | No action taken or action taken in response to the event or not |
| Action taken to Adcetris | provided |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), |
| Adcetris | treatment discontinuation, or not provided |

#### (3) Figure/table number

Tables 5.9.3-1 to 5.9.3-3

# 5.9.4 Outcome of peripheral nerve disorders (≥CTCAE Grade 3) considered related to Adcetris by action taken with Adcetris

#### (1) Analysis sets to be used

Patients included in safety evaluation and patients included in safety evaluation (Hodgkin's lymphoma) or patients included in safety evaluation (anaplastic large-cell lymphoma) who experience peripheral nerve disorder ( $\geq$ CTCAE Grade 3) considered related to Adcetris

#### (2) Data to be analyzed

For peripheral nerve disorders considered related to Adcetris, patients will be stratified into the categories below for each outcome and the incidence of these peripheral nerve disorders will be calculated. If the same patient has multiple occurrences of peripheral nerve disorder, the total number of occurrences will be calculated per category (for example, if the same patient has one episode of peripheral nerve disorder requiring dose reduction and one episode of peripheral nerve disorder leading to treatment discontinuation, these episodes of peripheral nerve disorder will be counted once for each category).

For each data item, missing data will be handled as "not provided." The percentage of peripheral nerve disorders for each category will be calculated using the total number of peripheral nerve

disorders for each category as the denominator:

| Data item | Category |
|---|---|
| Action taken to Adcetris | No action taken or action taken in response to the event or not provided |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), |
| Adcetris | treatment discontinuation, or not provided |

#### (3) Figure/table number

Tables 5.9.4-1 to 5.9.4-3

# 5.9.5 Occurrence of infections considered related to Adcetris by presence or absence of drugs used for the prevention of infection

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

Patients will be stratified into the categories below and the incidence of infections considered related to Adcetris for each CTCAE grade (the worst one) will be calculated by presence or absence of drugs used for the prevention of infection, using Mann-Whitney U test. The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple occurrences of the same infection, the occurrence with the highest CTCAE grade will be counted once for the category.

Similar analyses will be performed by use or non-use of antibiotics/synthetic antibacterial agents or trimethoprim-sulfamethoxazole combinations and by use or non-use of trimethoprim-sulfamethoxazole combinations for bacterial infection, by use or non-use of antifungals for fungal infection, and by use or non-use of antivirals for viral infection.

For patients included in safety evaluation who use antivirals for the prevention of viral infection but experience viral infection, a list of the following items will be generated: patient number, viral infection (name of the infection), age, sex, diagnosis, past history of hematopoietic stem cell transplantation (autologous or homologous), and drugs used for the prevention of infection (antivirals). If the same patient has multiple viral infections, all these viral infections will be counted.

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | None, Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infections | |

#### (3) Figure/table number

Tables 5.9.5-1 to 5.9.5-3 and 5.9.5-4

- 5.9.6 Occurrence of infections considered related to Adcetris by presence or absence of prior hematopoietic stem cell transplantation
  - (1) Analysis sets to be used

Patients included in safety evaluation and patients included in safety evaluation (Hodgkin's lymphoma) or patients included in safety evaluation (anaplastic large-cell lymphoma)

(2) Data to be analyzed

The incidence of infections considered related to Adcetris for each CTCAE grade (the worst one) will be calculated by presence or absence of prior hematopoietic stem cell transplantation (absent, present [autologous], present [autologous], present [autologous], or unknown) using Kruskal-Wallis test. The grade category of "unknown" will be excluded from the test.

The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple infections, the one with the highest CTCAE grade (the worst one) will be counted once for the category (the worst one).

Similary analyses will be performed for bacterial, fungal, and viral infections.

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | None, Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infection | |

#### (3) Figure/table number

Tables 5.9.6-1 to 5.9.6-3

- 5.9.7 Occurrence of neutropenia considered related to Adcetris by patient demographics and baseline characteristics
  - (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

(2) Data to be analyzed

For each data item of patient demographics and baseline characteristics, patients will be stratified into the categories below, and the incidence of neutropenia considered related to Adcetris will be calculated by CTCAE Grade (the worst one). The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple occurrences of neutropenia, the event with the highest CTCAE grade will be counted once.

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of neutropenia | |

Items and categories of patient demographics and baseline characteristics

| Data item | Category |
|---|---|
| Prior hematopoietic stem | Absent, present (autologous), present (homologous), present |
| cell transplantation | (autologous and homologous), or unknown |

| Degree of decreased | No decrease, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |
|---|---|
| neutrophil count at baseline | |
| Drugs used for the | Absort or present |
| prevention of infection | Absent or present |
| Specific drug(s) used for | Antibiotics/synthetic antibacterial agents, antifungals, antivirals, |
| the prevention of infection | trimethoprim-sulfamethoxazole combinations, or other |

#### (3) Figure/table number

Tables 5.9.7-1 to 5.9.7-3

#### 5.9.8 Treatment with Adcetris at the onset of neutropenia considered related to Adcetris

#### (1) Analysis sets to be used

Patients included in the safety analysis set and safety analysis set (Hodgkin's lymphoma) or safety analysis set (anaplastic large-cell lymphoma) who experience neutropenia considered related to Adcetris

#### (2) Data to be analyzed

For each CTCAE Grade (the worst one) of neutropenia considered related to Adcetris, patients will be stratified into the categories below, and the incidence of events of neutropenia will be calculated. If the same patient has multiple occurrences of neutropenia, the total number of occurrences will be calculated per category (for example, if the same patient has one episode of peripheral nerve disorder requiring dose reduction and one episode of peripheral nerve disorder leading to treatment discontinuation, these episodes of peripheral nerve disorder will be counted once for each category). The percentage of neutropenia for each category will be calculated using the number of neutropenia for each CTCAE grade (the worst one) as the denominator.

For each data item, missing data will be handled as "not provided."

| Data item | Category |
|---|---|
| Action taken to Adcetris | No action taken or action taken in response to the event or not provided |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), |
| Adcetris | treatment discontinuation or not provided |

#### (3) Figure/table number

Tables 5.9.8-1 to 5.9.8-3

#### 5.9.9 Outcome of neutropenia considered related to Adcetris by action taken with Adcetris

#### (1) Analysis sets to be used

Patients included in safety evaluation and patients included in safety evaluation (Hodgkin's lymphoma) or patients included in safety evaluation (anaplastic large-cell lymphoma) who experience neutropenia considered related to Adcetris

#### (2) Data to be analyzed

For neutropenia considered related to Adcetris, patients will be stratified into the categories below for each outcome and the incidence of neutropenia will be calculated. If the same patient has multiple occurrences of neutropenia, the total number of occurrences will be calculated per category (for example, if the same patient has one episode of neutropenia requiring dose reduction and one episode of neutropenia leading to treatment discontinuation, these episodes of neutropenia will be counted once for each category). The percentage of neutropenia for each category will be calculated using the total number of neutropenia for each category as the denominator.

For each data item, missing data will be handled as "not provided."

| Data item | Category |
|---|---|
| A ation taken to A deatric | No action taken or action taken in response to the event or not |
| Action taken to Adcetris | provided |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), |
| Adcetris | treatment discontinuation, or not provided |

#### (3) Figure/table number

Tables 5.9.9-1 to 5.9.9-3

#### 5.9.10 Occurrence of infusion reaction considered related to Adcetris

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

The incidence of infusion reaction considered related to Adcetris for each CTCAE grade (the worst one) will be calculated by infusion reaction and PT (see Section 1.2 for the definition of infusion reaction). For infusion reactions, the number and percentage of patients with infusion reaction will be calculated. For PT, the number and percentage of infusion reactions will be calculated. PTs will be presented in ascending order or PT Code.

The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple occurrences of infusion reaction or there are multiple occurrences of the same PT, the highest CTCAE grade (the worst one) for the patient or PT will be counted once for the category:

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infusion reaction | Grade 1, Grade 2, Grade 3, Grade 4, Grade 3, or diskilowii |

#### (3) Figure/table number

Tables 5.9.10-1 to 5.9.10-3

5.9.11 Occurrence of the new onset of infusion reaction observed within 2 days after treatment with Adcetris and considered related to Adcetris (time of the new onset)

#### (1) Analysis sets to be used

Patients included in safety evaluation and patients included in safety evaluation (Hodgkin's lymphoma) or patients included in safety evaluation (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

The incidence of the new onset of infusion reaction observed within 2 days after treatment with Adcetris and considered related to Adcetris will be calculated by time of onset. In addition, similar calculation will be performed by use or non-use of premedication to prevent infusion reaction. See the table below for the categories of time of onset:

| Data item | Category |
|---|---|
| | During infusion of Adcetris, after the completion of infusion of |
| Time of onset | Adcetris (≤1 hour, >1 hour to ≤12 hours, >12 hours to ≤24 hours, |
| | >24 hours), or unknown |

#### (3) Figure/table number

Tables 5.9.11-1 to 5.9.11-3

5.9.12 Occurrence of infusion reaction observed within 2 days after treatment with Adcetris and considered related to Adcetris by use or non-use of premedication to prevent infusion reaction

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

The total number of doses of Adcetris\*1 will be calculated by use or non-use of premedication to prevent infusion reaction (absent, present, or unknown). In addition, the incidence of infusion reaction observed within 2 days of the most recent treatment with Adcetris (i.e., observed on the day of treatment or on the day after treatment with Adcetris) and considered related to Adcetris will be calculated for each CTCAE grade (the worst one). The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple occurrences of infusion reaction during the same period, the one with the highest CTCAE grade (the worst one) will be counted once\*2.

The percentage of infusion reaction by use or non-use of premedication to prevent infusion reaction will be calculated using the total number of doses of Adcetris for each of these categories (i.e., use or non-use) as the denominator.

\*1: The total number of doses of Adcetris by use or non-use of premedication to prevent infusion reaction refers to the total doses per patient calculated by use or non-use of premedication. For example, if one patient receives 8 doses of Adcetris with premedication and 8 doses of Adcetris

without premedication, and another patient receives 10 doses of Adcetris with premedication and 6 doses of Adcetris without premedication, the total number of doses of Adcetris will be 18 (8 + 10) for the use of premedication and 14 (8 + 6) for the non-use of premedication.

\*2: For example, if the date the most recent treatment with Adcetris is January 1, 2016 and "Grade 2" infusion reaction is observed on January 1, 2016, and "Grade 3" infusion reaction on January 2, 2016, these two episodes of infusion reaction will be counted as one episode of "Grade 3" infusion reaction.

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infusion reaction | |

#### (3) Figure/table number

Tables 5.9.12-1 to 5.9.12-3

#### 5.9.13 Occurrence of adverse drug reactions of pulmonary disorder and infections

(1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

The incidence of pulmonary disorders considered related to Adcetris for each CTCAE grade (the worst one) will be calculated by pulmonary disorder and PT. PTs and PT Codes will be presented in ascending order.

In addition, the incidence of pulmonary disorders considered related to Adcetris for each CTCAE grade (the worst one) will be calculated by patient demographics and baseline characteristics.

The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple occurrences of pulmonary disorders or there are multiple occurrences of the same PT, the highest CTCAE grade (the worst one) for the patient or PT will be counted once for the category:

| Data item | | em | Category |
|---|---|---|---|
| CTCAE | Grade | (the worst | |
| one) | for | pulmonary | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| disorders | | | |

Items and categories of patient demographics and baseline characteristics

| Data item | Category |
|---|---|
| History of or concurrent pulmonary disorder | Absent or present |
| Smoking history | Non-smoker or smoker * Patients other than those who have never smoked will be classified into "smoker." |
| Prior radiotherapy | Absent or present |

#### (3) Figure/table number

Tables 5.9.13-1 to 5.9.13-4

- 5.10 analysis setanalysis setanalysis setList of actions taken with Adcetris in patients experiencing peripheral nerve disorders considered related to Adcetris
  - (1) Analysis sets to be used

Patients included in the safety analysis set analysis setanalysis setwho experience peripheral nerve disorders considered related to Adcetris

- (2) Data to be analyzed
- (3) For each patient, a list of the following data items: patient number, diagnosis, action taken or not taken with Adcetris, reason for action taken, date of dosing and dose for each cycle, date of onset of peripheral nerve disorder, CTCAE grade (the worst one), outcome, and the date of outcome. If the

same patient has multiple occurrences of peripheral nerve disorder, all these occurrences will be counted. Figure/table number

Table 5.10

#### 5.11 List of actions taken with Adcetris in patients experiencing neutropenia considered related to Adcetris

#### (1) Analysis sets to be used

Patients included in the safety analysis set analysis setanalysis setwho experience neutropenia considered related to Adcetris

#### (2) Data to be analyzed

For each patient, a list of the following data items: patient number, diagnosis, action taken or not taken with Adcetris, reason for action taken, date of dosing and dose for each cycle, date of onset of neutropenia, intervention provided for neutropenia, specific intervention (e.g., name of drugs/therapies) outcome, and the date of outcome. If the same patient has multiple occurrences of neutropenia, all these occurrences will be counted.

#### (3) Figure/table number

Table 5.11

#### 6.0 Efficacy Analysis

#### 6.1 Best response

(1) Analysis set to be used

Patients included in efficacy evaluation who complete best response assessmentanalysis set

#### (2) Data to be analyzed

The frequency of the best response after 16 cycles of treatment with Adcetris (or upon discontinuation of treatment with Adcetris) will be analyzed in patients Hodgkin's lymphoma and patients with anaplastic large-cell lymphoma. In addition, the point estimate of the response rate (CR + Cru + PR) with two-sided 95% confidence interval will be calculated, and a bar chart of the percentage of each category will be generated. Similar analyses will be performed by presence or absence of PET assessment, and a bar chart will be generated. For the handling of best response assessment data, see Section 1.7.

#### (3) Figure/table number

Table 6.1 and Figure 6.1

#### 6.2 Days to the best response

(1) Analysis set to be used

Patients included in efficacy evaluation who complete best response assessmentanalysis set

#### (2) Data to be analyzed

The frequency of days to the best response (1 to 21 days, 22 to 42 days, 43 to 63 days, [segmented similarly using a 21-day time window thereafter], 316 to 336 days, or ≥337 days) in patients with Hodgkin's lymphoma and patients with anaplastic large-cell lymphoma will be analyzed and summary statistics will be calculated. For the handling of best response assessment data, see Section 1.7. Figure/table number

Table 6.2 and Figure 6.2

#### 6.3 Overall survival

(3) Analysis sets to be used

Patients included in efficacy evaluation

(4) Data to be analyzed

The 1-year survivals with two-sided 95% confidence intervals in patients will be calculated using the Kaplan-Meier method, and a Kaplan-Meier plot will be generated for Hodgkin's lymphoma and patients and anaplastic large-cell lymphoma respectively.

(5) Figure/table number

Table 6.3 and Figure 6.3

# Appendix: Definition of Pulmonary Disorders (MedDRA Preferred Terms)

| <ul> <li>Acute interstitial</li> </ul> | <ul> <li>Idiopathic pneumonia</li> </ul> | <ul> <li>Pulmonary haemosiderosis</li> </ul> |
|---|---|---|
| pneumonitis (10066728) | syndrome (10063725) | (10037396) |
| <ul> <li>Acute lung injury</li> </ul> | <ul> <li>Idiopathic pulmonary</li> </ul> | <ul> <li>Pulmonary necrosis</li> </ul> |
| (10069351) | fibrosis (10021240) | (10058824) |
| <ul> <li>Acute respiratory distress</li> </ul> | <ul> <li>Interstitial lung disease</li> </ul> | <ul> <li>Pulmonary oedema</li> </ul> |
| syndrome (10001052) | (10022611) | (10037423) |
| <ul> <li>Acute respiratory failure</li> </ul> | • Lung disorder (10025082) | <ul> <li>Pulmonary radiation injury</li> </ul> |
| (10001053) | , | (10061473) |
| <ul> <li>Alveolar proteinosis</li> </ul> | <ul> <li>Lung infiltration</li> </ul> | <ul> <li>Pulmonary sarcoidosis</li> </ul> |
| (10001881) | (10025102) | (10037430) |
| • Alveolitis (10001889) | <ul> <li>Necrotising bronchiolitis</li> </ul> | <ul> <li>Pulmonary toxicity</li> </ul> |
| () | (10070831) | (10061924) |
| <ul> <li>Alveolitis allergic</li> </ul> | Obliterative bronchiolitis | Pulmonary vasculitis |
| (10001890) | (10029888) | (10037457) |
| Systemic sclerosis | <ul> <li>Organising pneumonia</li> </ul> | • Radiation alveolitis |
| pulmonary (10042954) | (10067472) | (10037754) |
| • Alveolitis necrotising | • Pneumonitis (10035742) | • Radiation fibrosis – lung |
| (10050343) | <sup>3</sup> Theumonitis (10033742) | (10037758) |
| | <ul> <li>Pneumonitis chemical</li> </ul> | <ul> <li>Radiation pneumonitis</li> </ul> |
| • Bronchiolitis (10006448) | | |
| D:00111 | (10035745) | (10037765) |
| • Diffuse alveolar damage | • Progressive massive | • Respiratory arrest |
| (10060902) | fibrosis (10036805) | (10038669) |
| • Eosinophilic pneumonia | Pulmonary alveolar | • Respiratory distress |
| (10014962) | haemorrhage (10037313) | (10038687) |
| Eosinophilic pneumonia | <ul> <li>Pulmonary eosinophilia</li> </ul> | <ul> <li>Respiratory failure</li> </ul> |
| acute (10052832) | (10037382) | (10038695) |
| <ul> <li>Eosinophilic pneumonia</li> </ul> | <ul> <li>Pulmonary fibrosis</li> </ul> | <ul> <li>Sarcoidosis (10039486)</li> </ul> |
| chronic (10052833) | (10037383) | |
| <ul> <li>Hypoxia (10021143)</li> </ul> | <ul> <li>Pulmonary granuloma</li> </ul> | |
| | (10037391) | |
| · | | |

The above definition is consistent with the one used in clinical studies of Adcetris.

# Statistical Analysis Plan

# ADCETRIS IV Infusion – Special Drug Use Surveillance (All-case Surveillance) "Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell Lymphoma"

| | Takeda Pharmaceutical Company Limited |
|------|---------------------------------------|
| PPD | |
| Stat | tistical Analysis Agent |
| | PPD |

# Table of Contents

| 1.0 | Definition of Terms and Handling of Test/Measurement Data | . 1 |
|---|---|---|
| 1.1 | Definition | . 1 |
| 1.2 | Display digits | 8 |
| 1.3 | Level of significance. | 8 |
| 1.4 | Handling of test data | 8 |
| 2.0 | Patient Disposition (Patient Disposition Diagram) | 10 |
| 3.0 | Patient Demographics and Baseline Characteristics | 11 |
| 4.0 | Treatment Given | 14 |
| 4.1 | Treatment given | 14 |
| 4.2 | Premedication to prevent infusion reaction | 15 |
| 5.0 | Safety Analysis | 16 |
| 5.1 | Occurrences of adverse events/infections and adverse drug reactions/infections | 16 |
| 5.1 | .1 Occurrence of adverse events/infections | 16 |
| 5.1 | .2 Occurrence of adverse drug reactions/infections | 17 |
| 5.2 | Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrences | of |
| | adverse events/infections and adverse drug reactions/infections by outcome | 18 |
| 5.2 | Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrent | ce |
| of a | adverse events/infections by outcome | 18 |
| 5.2 | Occurrence of adverse events/infections by CTCAE Grade (the worst one) | 19 |
| 5.2 | Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrent | ce |
| of a | adverse drug reactions/infections by outcome | 21 |
| 5.2 | Occurrence of adverse drug reactions/infections by CTCAE Grade (the worst one) | 23 |
| 5.3 | Percentage of patients with adverse drug reactions/infections by patient demographics and baseling | ne |
| | characteristics and treatment given | 23 |
| 5.4 | Occurrence of adverse drug reactions/infections by age group | 26 |
| 5.5 | Occurrence of adverse drug reactions/infections by presence or absence of concurrent hepatic disord | er |
| | | 26 |
| 5.6 | Occurrence of adverse drug reactions/infections by presence or absence of concurrent renal disorder2 | 26 |
| 5.7 | List of the occurrence of serious adverse events/infections | 27 |
| 5.8 | Change in test data over time | 28 |
| 5.8 | .1 Laboratory tests | 28 |
| 5.9 | Analysis of items of particular interest | 28 |
| 5.9 | .1 Occurrence of peripheral nerve disorder | 28 |
| 5.9 | .2 Occurrence of peripheral nerve disorders by patient demographics and baseline characteristics an | ıd |
| trea | atment given | 29 |
| 5.9 | .3 Treatment with Adcetris at the onset of peripheral nerve disorders | 30 |
| 5.9 | .4 Occurrence of infections by presence or absence of drugs used for the prevention of infection | 30 |
| 5.9 | Occurrence of neutropenia by patient demographics and baseline characteristics | 31 |

| 5.9 | 5.9.6 Treatment with Adcetris at the onset of neutropenia | |
|---|---|---|
| 5.9.7 Occurrence of infusion reaction | | 32 |
| 5.9 | Occurrence of infusion reaction by the use or non-use of premedication to prevent infusion | on reaction |
| | 32 | |
| 5.9 | Occurrence of pulmonary disorders | 33 |
| 5.10 | occurrence of infections by presence or absence of hematopoietic stem cell transplantation | 33 |
| 5.11 | ist of actions taken with Adcetris in patients experiencing peripheral nerve disorders | 33 |
| 5.12 | .12 List of actions taken with Adcetris in patients experiencing neutropenia | |
| 6.0 | fficacy Analysis | 35 |
| 6.1 | est response | 35 |
| 6.2 | verall survival | 35 |
| Append | | 36 |

# 1.0 Definition of Terms and Handling of Test/Measurement Data

# 1.1 Definition

| Term | Definition |
|---|---|
| This/the product | Refers to Adcetris for intravenous drip infusion in this Statistical Analysis |
| | Plan. |
| SOC | MedDRA/J System Organ Class |
| HLGT | MedDRA/J High Level Group Term |
| PT | MedDRA/J Preferred Term |
| LLT | MedDRA/J Lowest Level Term |
| Patients registered | Patients whose registration has been approved |
| Patients whose case report | Patients whose case report forms have been collected |
| forms are available | |
| Patients whose case report | Patients registered but whose case report form have not been collected |
| forms are not available | |
| Fixed patients | Patients whose case report forms are available, with the date of case report |
| | form completion entered in the PMS system |
| Non-fixed patients | Patients whose case report forms are available, with the date of case report |
| | form completion not entered in the PMS system |
| Safety analysis set | Fixed patients included in the safety analysis set |
| Safety analysis set (Hodgkin's | Patients included in the safety analysis set whose diagnosis is Hodgkin's |
| lymphoma) | lymphoma |
| Safety analysis set (anaplastic | Patients included in the safety analysis set whose diagnosis is anaplastic |
| large-cell lymphoma) | large-cell lymphoma |
| Patients excluded from the | Fixed patients excluded from the safety analysis set |
| safety analysis set | |
| Efficacy analysis set | Patients included in the safety analysis set who are also included in the |
| | efficacy analysis set |
| Patients excluded from the | Patients included in the safety analysis set who are excluded from the |
| efficacy analysis set | efficacy analysis set |
| Patients completing treatment | Patients completing 16 cycles of treatment with Adcetris |
| Patients discontinuing treatment | Patients not completing 16 cycles of treatment with Adcetris |
| Adverse events, etc. | Refers to "adverse events and infections." |
| | In this Statistical Analysis Plan, the term "adverse events and infections" |
| | is used in titles and the term "adverse events, etc." is used in text and |
| | tables. |
| Adverse drug reactions, etc. | Refers to "adverse drug reactions and infections." |
| | Adverse events, etc., not considered "not related" to Adcetris by the |
| | investigator. |

| Term | Definition |
|---|---|
| | In this Statistical Analysis Plan, the term "adverse drug reactions and |
| | infections" is used in titles and the term "adverse drug reactions, etc." is |
| | used in text and tables. |
| Serious adverse events, etc. | Refers to "serious adverse events and infections." |
| | Adverse events considered "serious" by the investigator. |
| | Events listed in the MedDRA Coding List in the Takeda Medically |
| | Significant AE List should be regarded as serious even if they are |
| | considered "non-serious" by the investigator. |
| | In this Statistical Analysis Plan, the term "serious adverse events and |
| | infections" is used in titles and the term "serious adverse events, etc." is |
| | used in text and tables. |
| Number of patients with | Number of patients experiencing adverse events, etc., or adverse drug |
| adverse events/adverse drug | reactions, etc. |
| reactions | |
| Number of adverse | Number of adverse events, etc., or adverse drug reactions, etc., observed |
| events/adverse drug reactions | |
| Percentage of patients with | [For safety analysis using patients included in the safety analysis set] |
| adverse events/adverse drug | Is calculated using the following formula: (number of patients with |
| reactions | adverse events/adverse drug reactions) / (number of patients included in |
| | the safety analysis set) × 100. |
| | [For safety analysis using patients excluded from the safety analysis set] |
| | Is calculated using the following formula: (number of patients with |
| | adverse events/adverse drug reactions) / (number of patients excluded |
| | from the safety analysis set) × 100. |
| Percentage of adverse | [For safety analysis using patients included in the safety analysis set] |
| events/adverse drug reactions | Is calculated using the following formula: (number of adverse |
| observed | events/adverse drug reactions observed) / (number of patients included in |
| | the safety analysis set) $\times$ 100. |
| | [For safety analysis using patients excluded from the safety analysis set] |
| | Is calculated using the following formula: (number of adverse |
| | events/adverse drug reactions observed) / (number of patients excluded |
| | from the safety analysis set) $\times$ 100. |
| Time of onset | Is calculated using the following formula: date of onset of adverse events, |
| | etc. (or adverse drug reactions, etc.) – date of the initial dose of Adcetris + |
| | 1. |
| | If the day and month of onset of adverse events, etc. (or adverse drug |
| | reactions, etc.) are unknown, the date of onset should be "January 1." |
| | However, if the year of the initial dose of Adcetris is the year of onset of |
| | adverse events, etc. (or adverse drug reactions, etc.), the date of onset |

| Term | Definition | | |
|---|---|---|---|
| | should be the day and month of the initial dose of Adcetris. | | |
| | If the day of onset of adverse events, etc. (or adverse drug reactions, etc.) | | |
| | is unknown, the date of onset should be the first day of the month. | | |
| | However, if the year and month of the initial dose of Adcetris is the year | | |
| | and month of onset of adverse events, etc. (or adverse drug reactions, etc.), | | |
| | the date of the initial dose of Adcetris should be the date of onset. | | |
| Patients with concurrent hepatic | Patients having a concurrent illness that falls under the category of | | |
| disorder | Standardized MedDRA Query (SMQ) Code 20000005 (SMQ Hepatic | | |
| | disorders [Scope: | Narrow]) | |
| Grade of hepatic disorder | The ALT or AST | level at baseline with the l | nighest CTCAE grade will be |
| | used to determine | the grade of hepatic disor | rder. The grades of ALT and |
| | AST levels will be | e determined according to the | ne following tables: |
| | ALT | Male | Female |
| | None | ≤42 IU/L | ≤23 IU/L |
| | Grade 1 | >42 to 126 IU/L | >23 to 69 IU/L |
| | Grade 2 | >126 to 210 IU/L | >69 to 115 IU/L |
| | ≥Grade 3 | >210 IU/L | >115 IU/L |
| | AST | | |
| | None | ≤30 IU/L | |
| | Grade 1 | >30 to 90 IU/L | |
| | Grade 2 | >90 to 150 IU/L | |
| | ≥Grade 3 | >150 IU/L | |
| Patients with concurrent renal | Patients having a concurrent illness that falls under the category of Takeda | | |
| disorder | MedDRA Query (TMQ) (Renal disease) | | |
| Grade of renal disorder: None | The serum creatin | ine level at baseline is: | |
| | $\leq$ 1.07 mg/dL for n | nales | |
| | ≤0.79 mg/dL for females | | |
| Grade of renal disorder: 1 | The serum creatinine level at baseline is: | | |
| | >1.07 to 1.605 mg | g/dL for males | |
| | >0.79 to 1.185 mg | y/dL for females | |
| Grade of renal disorder: 2 | The serum creatin | ine level at baseline is: | |
| | >1.605 to 3.21 mg | y/dL for males | |
| | >1.185 to 2.37 mg/dL for females | | |
| Grade of renal disorder: ≥3 | The serum creatin | ine level at baseline is: | |
| | >3.21 mg/dL for n | nales | |
| | >2.37 mg/dL for f | emales | |
| Patients with a past history of | Patients with a past history that falls under the category of Appendix | | |

| Term | Definition |
|---|---|
| pulmonary disorder | "Definition of Pulmonary Disorders" |
| | (If "No concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | pulmonary disorders" in the case report form, the pulmonary disorder |
| | should be regarded as a past history.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of Appendix |
| pulmonary disorder | "Definition of Pulmonary Disorders" |
| | (If "A concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | pulmonary disorders" in the case report form, the pulmonary disorder |
| | should be regarded as a concurrent illness.) |
| Patients with a past history of | Patients with a past history that falls under the category of MedDRA SMQ |
| malignant tumour | Code 20000194 (SMQ Malignant tumours [Scope: Narrow]) |
| | (If "No concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | malignant tumours" in the case report form, the pulmonary disorder should |
| | be regarded as a past history.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| malignant tumour | SMQ Code 20000194 (SMQ Malignant tumours [Scope: Narrow]) |
| | (If "A concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | malignant tumours" in the case report form, the pulmonary disorder should |
| | be as a concurrent illness.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| diabetes mellitus | SMQ Code 20000041 (SMQ Hyperglycaemia/new onset diabetes mellitus |
| | [Scope: Narrow]) |
| Patients with hypertension | Patients with a concurrent illness that falls under the category of MedDRA |
| | SMQ Code 20000147 (SMQ Hypertension [Scope: Narrow]) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| dyslipidaemia | SMQ Code 20000026 (SMQ Dyslipidaemia [Scope: Narrow]) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| hyperuricaemia | PT Code 10020903 (Hyperuricaemia) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| infection | SOC Code 10021881 (Infections and infestations) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of SMQ |
| peripheral neuropathy | Code 20000034 (SMQ Peripheral neuropathy [Scope: Narrow]) |
| Patients with other concurrent | Patients with any concurrent illness other than those listed above |
| illnesses | |
| Antibiotics/synthetic | Prophylactics against infections that fall under the category of those with |
| • | |

| Term | Definition |
|---|---|
| antibacterial agents | the first three digits of YJ Code being 611 to 616 or 619 (If more than one |
| | antibiotics/synthetic antibacterial agents are used in the same patient, it |
| | will be counted as one patient.) |
| Antifungals | Prophylactics against infections that fall under the category of those with |
| | the first three digits of YJ Code being 617 (If more than one antifungals |
| | are used in the same patient, it will be counted as one patient.) |
| Antivirals | Prophylactics against infections that fall under the category of those with |
| | the first three digits of YJ Code being 625 (If more than one antivirals are |
| | used in the same patient, it will be counted as one patient.) |
| Trimethoprim-sulfamethoxazole | Prophylactics against infections that fall under the category of those with |
| combinations | YJ Code being 629010007 to 9 |
| Other prophylactics against | Any drug entered in the field of "Drugs used for the prevention of |
| infections | infection" other than prophylactics against infections listed above (If more |
| | than one other prophylactics against infections are used in the same |
| | patient, it will be counted as one patient.) |
| Peripheral sensory neuropathy | Adverse events with "Sensory neuropathy" entered in the "Category of |
| (as an adverse event) | peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral |
| | nerve disorders] in the case report form. MedDRA PT Code 10034620 |
| | should be assigned regardless of data entered in "Symptoms" in the field. |
| Peripheral motor neuropathy | Adverse events with "Motor neuropathy" entered in the "Category of |
| (as an adverse event) | peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral |
| | nerve disorders] in the case report form. MedDRA PT Code 10034580 |
| | should be assigned regardless of data entered in "Symptoms" in the field. |
| Peripheral neuropathy | Adverse events with "Other" entered in the "Category of peripheral nerve |
| (as an adverse event) | disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] |
| | in the case report form. MedDRA PT Code 10029331 should be assigned, |
| | regardless of data entered in "Symptoms" in the field. |
| Pulmonary disorders | Adverse events that fall under the category of Appendix "Definition of |
| (as adverse events) | Pulmonary Disorders" |
| Infusion reaction | Adverse events entered in the field of "Adverse events: [4] Infusion |
| | reaction," regardless of data entered in "Symptoms" in the field. |
| Patients with the onset of | Patients with adverse drug reactions that fall under the category of |
| infection | MedDRA SOC Code 10021881 (Infections and infestations) |
| Patients with the onset of | Patients with adverse drug reactions that fall under the category of |
| bacterial infection | MedDRA HGLT Code 10004018 (Bacterial infection), 10008555 |
| | (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 |
| | (Rickettsia infection) |
| Patients with the onset of fungal | Patients with adverse drug reactions that fall under the category of |
| infection | MedDRA HGLT Code 10017528 (Fungal infection) |

| Term | Definition |
|---|---|
| Patients with the onset of viral | Patients with adverse drug reactions that fall under the category of |
| infection | MedDRA HGLT Code 10047438 (Viral infection) |
| Age | If the month and day of the initial dose of Adcetris is < the month and day |
| | of birth, the patient's age will be calculated using the following formula: |
| | Year of the initial dose of Adcetris – year of birth – 1. |
| | If the month and day of the initial dose of Adcetris is ≥ the month and day |
| | of birth, the patient's age will be calculated using the following formula: |
| | Year of the initial dose of Adcetris – year of birth. |
| | If the month and day of birth are unknown, they should be "January 1," |
| | and if the day of birth is unknown, it should the first day of the month. |
| BMI | BMI should be calculated using the following formula: Weight |
| | (kg)/(0.0001 × height (cm) × height (cm). The obtained value should be |
| | rounded off to one decimal place. |
| Disease duration | The disease duration should be calculated using the following formula: |
| | ["Date of the initial dose of Adcetris" – "date of diagnosis of Hodgkin's or |
| | anaplastic large-cell lymphoma" +1]/365.25. |
| | The day of diagnosis should be the first day of the month provided. If the |
| | month of diagnosis is unknown, the date of diagnosis should be "January |
| | 1st" of the year provided. |
| Mean dose of Adcetris | Is calculated as the total value of each dose of Adcetris given at each |
| | treatment cycle divided by the number of cycles. |
| Dose of Adcetris per 3 weeks | Is calculated using the following formula: Total "dose of Adcetris"/(["date |
| | of the last dose of Adcetris" - "date of the initial dose of Adcetris" + |
| | 21)/21]. |
| | If only 1 cycle of treatment is given, the "date of the last dose of Adcetris" |
| | and the "date of the initial dose of Adcetris" should be regarded as the |
| | same. |
| Degree of decreased neutrophil | Neutrophil count at baseline ≥2,000 /mm <sup>3</sup> |
| count at baseline: No decrease | |
| Degree of decreased neutrophil | Neutrophil count at baseline <2,000 to 1,500 /mm <sup>3</sup> |
| count at baseline: Grade 1 | |
| Degree of decreased neutrophil | Neutrophil count at baseline <1,500 to 1,000 /mm <sup>3</sup> |
| count at baseline: Grade 2 | |
| Degree of decreased neutrophil | Neutrophil count at baseline <1,000 to 500 /mm <sup>3</sup> |
| count at baseline: Grade 3 | |
| Degree of decreased neutrophil | Neutrophil count at baseline <500 /mm <sup>3</sup> |
| count at baseline: Grade 4 | |
| Date of the final observation | "Date of the final observation" in the case report form |
| | If not provided, the most recent date entered in the case report form should |

| Term | Definition |
|---|---|
| | be used. |
| Summary statistics | Includes mean, standard deviation, minimum, 25th percentile, median, |
| | 75th percentile, and maximum. |

#### 1.2 Display digits

| Term | Definition |
|---|---|
| Percentage (%) | Percentage of patients with or percentage of adverse events, etc., or adverse drug |
| | reactions, etc.: |
| | The obtained value should be rounded off to two decimal places. |
| | Other: |
| | The obtained value should be rounded off to one decimal place. |
| Summary statistics | Mean: |
| (mean and standard | The raw data should be rounded off to one decimal place. |
| deviation) | Standard deviation: |
| | The raw data should be rounded off to two decimal places. |
| P value | The obtained value should be rounded down to three decimal places. |
| | If the value is less than 0.001 after rounding down to three decimal places, it |
| | should be displayed as "p<0.001." |

#### 1.3 Level of significance

Two-sided 5%

#### 1.4 Handling of test data

Test data will be handled according to the criteria shown below. If there are multiple data for the same criterion, the one with the test date being closest to the date of protocol-specified assessment should be used. If there is no difference in the number of days from the date of protocol-specified assessment, the later value should be used. For the final assessment, \*however, the most recently measured value (including the one measured during the off-treatment period) after the date of the initial dose of Adcetris should be used. Values measured after 30 days after the last dose of Adcetris should not be used.

The number of days after the date of the initial dose of Adcetris is defined as 1 for the date of the initial dose of Adcetris and 0 for the day before the date of the initial dose of Adcetris.

\*After 16 cycles of treatment with Adcetris (or upon discontinuation of treatment with Adcetris)

| Time point for testing | Acceptable time window | Date of protocol-specified assessment |
|---|---|---|
| At the initial dose of | -21 to 1 days | Date of the initial dose of Adcetris |
| Adcetris | | |
| After 1 cycle | 2 to 31 days | Date of the initial dose of Adcetris + 21 |
| After 2 cycles | 32 to 52 days | Date of the initial dose of Adcetris + 42 |
| After 3 cycles | 53 to 73 days | Date of the initial dose of Adcetris + 63 |
| After 4 cycles | 74 to 94 days | Date of the initial dose of Adcetris + 84 |
| After 5 cycles | 95 to 115 days | Date of the initial dose of Adcetris + 105 |
| After 6 cycles | 116 to 136 days | Date of the initial dose of Adcetris + 126 |
| After 7 cycles | 137 to 157 days | Date of the initial dose of Adcetris + 147 |

| Time point for testing | Acceptable time window | Date of protocol-specified assessment |
|---|---|---|
| After 8 cycles | 158 to 178 days | Date of the initial dose of Adcetris + 168 |
| After 9 cycles | 179 to 199 days | Date of the initial dose of Adcetris + 189 |
| After 10 cycles | 200 to 220 days | Date of the initial dose of Adcetris + 210 |
| After 11 cycles | 221 to 241 days | Date of the initial dose of Adcetris + 231 |
| After 12 cycles | 242 to 262 days | Date of the initial dose of Adcetris + 252 |
| After 13 cycles | 263 to 283 days | Date of the initial dose of Adcetris + 273 |
| After 14 cycles | 284 to 304 days | Date of the initial dose of Adcetris + 294 |
| After 15 cycles | 305 to 325 days | Date of the initial dose of Adcetris + 315 |
| After 16 cycles | 326 to 346 days | Date of the initial dose of Adcetris + 336 |

#### 2.0 Patient Disposition (Patient Disposition Diagram)

#### (1) Analysis set to be used

Patients registered to this specified drug-use survey

#### (2) Data to be analyzed

Data to be analyzed includes the numbers of patients registered, institutions with patients registered, patients whose case report forms are available/not available, fixed/non-fixed patients, patients included in/excluded from the safety analysis set, and patients included in/excluded from the efficacy analysis set.

For the number of institutions with patients registered, the same institutions with different departments should not be counted more than once.

For patients whose case report forms are not available, the number of patients by reason for unavailability and the total number of patients will be calculated.

For patients excluded from the safety/efficacy analysis set, the number of patients by reason for exclusion and the total number of patients will be calculated.

It will be determined as follows whether patients meeting the following criteria should be included or excluded:

| Criterion | Registration | Safety<br>evaluation | Efficacy evaluation |
|---|---|---|---|
| Duplicate registration (of the same patient) | × | × | × |
| [found afterwards] | | | |
| Non-primary disease | 0 | 0 | × |
| Adcetris has never been administered [found | × | × | × |
| afterwards] | | | |
| No definite safety evaluation results are | 0 | × | × |
| available | | | |
| No definite efficacy evaluation results are | 0 | 0 | × |
| available | | | |
| No case report form is available | 0 | × | × |

o: Included, ×: Excluded

#### (3) Figure/table number

Figure 2.0 and Table 2.0

# 3.0 Patient Demographics and Baseline Characteristics

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the number and frequency of patients will be calculated:

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | Summary statistics |
| | <18 years, 18 to 39 years, 40 to 64 years, 65 to 74 years, or ≥75 years |
| | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| Diagnosis | Hodgkin's or anaplastic large-cell lymphoma or other |
| Status | Relapsed/refractory, or new-onset |
| CD30 | Positive, negative, or not measured |
| Sita(a) a financian | Lymph node, spleen, liver, lung, bone, central nerve, bone marrow, |
| Site(s) of involvement | skin, and/or other |
| ALK (for patients | |
| with anaplastic | Positive, negative, or unknown |
| large-cell lymphoma) | |
| Clinical stage | I, II, III, IV, or unknown |
| B symptoms | Absent or present |
| ECOG Performance | 0.1.2.2 or 4 |
| Status | 0, 1, 2, 3, or 4 |
| Therapeutic category | Outpatient or inpatient |
| Hypersensitivity | Absent, present, or unknown |
| disposition | Absent, present, or unknown |
| Specific | |
| hypersensitivity | Medications, food allergy, and/or other |
| disposition(s) | |
| HCV antibody | Negative, positive, or unknown |
| HBs antigen | Negative, positive, or unknown |
| HBs antibody | Negative, positive, or unknown |
| HBV DNA | Negative, positive, or unknown |
| Past history of | Absent or present |
| pulmonary disorders | |
| Concurrent pulmonary | Absent or present |
| disorders | |

| Data item | Category |
|---|---|
| Past history of | Alegant on progent |
| malignant tumours | Absent or present |
| Concurrent malignant | Absent or present |
| tumours | Absent of present |
| Past history (other | |
| than pulmonary | Absent, present, or unknown |
| disorders and | Absent, present, or unknown |
| malignant tumours) | |
| Concurrent illness | |
| (other than pulmonary | Absent or present |
| disorders and | Absent of present |
| malignant tumours) | |
| Specific concurrent | |
| illness(es) (other than | Diabetes mellitus, hypertension, dyslipidaemia, hyperuricaemia, |
| pulmonary disorders | hepatic disease(s), renal disease(s), infections, peripheral nerve |
| and malignant | disorders, and/or other |
| tumours) | disorders, and/or other |
| Concurrent renal | Absent or present |
| disorders | Absent or present |
| Grade of hepatic | |
| disorder | |
| (CTCAE grade based | None, Grade 1, Grade 2, or ≥Grade 3 |
| on AST and ALT | |
| levels) | |
| Concurrent renal | Absent or present |
| disorders | About of present |
| Grade of renal | |
| disorder | None, Grade 1, Grade 2, or ≥Grade 3 |
| (CTCAE grade based | Ivolic, Grade 1, Grade 2, or Editate 3 |
| on serum creatinine) | |
| Weight | Summary statistics |
| | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, ≥70 kg, or not |
| | measured |
| | Summary statistics |
| BMI | $<18.5 \text{ kg/m}^2$ , $<18.5 \text{ to } 25 \text{ kg/m}^2$ , $<25 \text{ to } 30 \text{ kg/m}^2$ , $\ge 30 \text{ kg/m}^2$ , or |
| | unknown |
| Smoking history | Never, current, past, or unknown |
| Prior drug therapy | Absent or present |

| Data item | Category |
|---|---|
| Prior drug therapy | ABVD, CHOP, and/or other |
| regimen(s) | (If more than one drug therapies in the same category is used in the |
| | same patient, it will be counted as one patient.) |
| Number of prior drug | Summary statistics |
| therapy regimens | Summary statistics |
| Days from the month | |
| of the completion of | |
| the final regimen of | |
| prior drug therapy to | |
| the date of 1 cycle of | Summary statistics |
| treatment with | |
| Adcetris | |
| (Prior drug therapy: | |
| Yes) | |
| Prior radiotherapy | Absent or present |
| Days from the month | |
| of the completion of | |
| the most recent prior | |
| radiotherapy to the | |
| date of 1 cycle of | Summary statistics |
| treatment with | |
| Adcetris | |
| (Prior radiotherapy: | |
| yes) | |
| Prior hematopoietic | |
| stem cell | Absent, present (autologous), or present (homologous) |
| transplantation | |
| Other prior therapies | Absent or present |
| Pregnancy during the | |
| observation period | Absent or present |
| (for females only) | |

# (3) Figure/table number

Tables 3.0-1 to 3.0-3

#### 4.0 Treatment Given

# 4.1 Treatment given

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the number and frequency of patients will be calculated:

| Data item | Category |
|---|---|
| Initial dose of<br>Adcetris | 1.8 mg/kg or other |
| Mean dose of Adcetris | <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg |
| Dose of Adcetris per 3 weeks | <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg |
| Duration of treatment with Adcetris | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, or 16 cycles |
| Reason(s) for | |
| discontinuation of | Treatment goal achieved, adverse event(s), lost to follow-up, transfer to |
| Adcetris | another hospital, pregnancy, inadequate response, and/or other |
| Post-baseline | |
| hematopoietic stem | Absent or present |
| cell transplantation | |
| Type of post-baseline | |
| hematopoietic stem | Autologous or homologous |
| cell transplantation | |
| Drug(s) other than | |
| Adcetris used for the | Absent or present |
| treatment of the | |
| primary disease | |
| Drug(s) used for the | |
| prevention of | Absent or present |
| infection | |
| Specific drug(s) used | Antibiotics/synthetic antibacterial agents, antifungals, antivirals, |
| for the prevention of | trimethoprim-sulfamethoxazole combinations, and/or other |
| infection | prophylactics against infections |

#### (3) Figure/table number

Tables 4.1-1 to 4.1-3

# 4.2 Premedication to prevent infusion reaction

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each cycle, patients will be stratified into the following categories, and the number and frequency of patients will be calculated:

| Data item | Category |
|---|---|
| Premedication to prevent infusion reaction | Absent or present |
| Specific premedication(s) used to prevent infusion reaction | Acetaminophen, antihistamines, and/or corticosteroids |

#### (3) Figure/table number

Tables 4.2-1 to 4.2-3

#### 5.0 Safety Analysis

#### 5.1 Occurrences of adverse events/infections and adverse drug reactions/infections

#### 5.1.1 Occurrence of adverse events/infections

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

Data listed below will be analyzed.

For data entered in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form, MedDRA PT Code for peripheral sensory neuropathy, peripheral motor neuropathy, or peripheral neuropathy should be assigned, regardless of the LLT code entered in "Symptoms" field (see Section 1.1, the same applies hereinafter).

Neutrophil count decreased (PT Code 10029366) will be replaced by Neutropenia (PT Code 10029354), Lymphocyte count decreased (PT Code 10025256) by Lymphopenia (PT Code 10025327), White blood cell count decreased (PT Code 10047942) by Leukopenia (PT Code 10024384), and Platelet count decreased (PT Code 10035528) by Thrombocytopenia (PT Code 10043554) (the same applies hereinafter).

| Data item | Data to be analyzed |
|---|---|
| Number of patients with adverse events, etc. | Number of patients experiencing adverse events, etc. |
| Number of adverse events, etc. | Number of adverse events, etc., observed If the same patient has multiple occurrences of the same adverse event, etc. (PT), the total number of occurrences will be calculated. |
| Percentage of patients with adverse events, etc. | Is calculated using the following formula: number of patients with adverse events, etc./number of patients included in the safety analysis set $\times$ 100. |
| Type of adverse events, etc. | Adverse events, etc., will first be classified by SOC, within each of which adverse events, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. For SOC, the number and percentage of patients with adverse events, etc., will be presented in the internationally agreed order. For PT, the number and percentage of adverse events, etc., will be presented in ascending order of PT codes. If the same patient has multiple occurrences of the same adverse event, etc. (PT), the event will be counted once per patient. |

#### (3) Figure/table number

Tables 5.1-1 to 5.1.1-3
# 5.1.2 Occurrence of adverse drug reactions/infections

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

Data listed below will be analyzed.

| Data item | Data to be analyzed |
|---|---|
| Number of patients with adverse drug reactions, etc. | Number of patients experiencing adverse drug reactions, etc. |
| Number of adverse drug reactions, etc. | Number of adverse drug reactions, etc., observed. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the total number of occurrences will be calculated. |
| Percentage of patients with adverse drug reactions, etc. | Is calculated using the following formula: number of patients with adverse drug reactions, etc./number of patients included in the safety analysis set $\times$ 100. |
| Type of adverse drug reactions, etc. | Adverse drug reactions, etc., will first be classified by SOC, within each of which adverse drug reactions, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. For SOC, the number and percentage of patients with adverse drug reactions, etc., will be presented in the internationally agreed order. For PT, the number and percentage of adverse drug reactions, etc., will be presented in ascending order of PT codes. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the reaction will be counted once per patient. |

# (3) Figure/table number

Tables 5.1-2 to 5.1.2-3

- 5.2 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrences of adverse events/infections and adverse drug reactions/infections by outcome
  - 5.2.1 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrence of adverse events/infections by outcome
    - (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse events, etc., will be analyzed:

| Data item | Category |
|---|---|
| Seriousness | Serious or non-serious |
| CTCAE Grade (the worst one) | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| Time of onset | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, or ≥337 days |
| | 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly using a 21-day time window thereafter), 316 to 336 days, or ≥337 days |
| | 1 to 7 days, 8 to 14 days, 15 to 21 days, (segmented similarly using a 7-day time window thereafter), 330 to 336 days, or ≥337 days |
| Time to the worst grade | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, or ≥337 days |
| | 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly using a 21-day time window thereafter), 316 to 336 days, or ≥337 days |
| | 1 to 7 days, 8 to 14 days, 15 to 21 days, (segmented similarly using a 7-day time window thereafter), 330 to 336 days, or ≥337 days |
| Outcome | Recovered/resolved, recovering/resolving, not recovered/not resolved, recovered/resolved with sequelae, died/fatal, or unknown |

The type of adverse events, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse events, etc., by SOC/PT |
| Number of adverse events, etc. | Number of adverse events, etc., observed by SOC/PT |
| | Adverse events, etc., will first be classified by SOC, within each |
| | of which adverse events, etc., will be further classified by PT. |
| | Laboratory test data will first be classified by SOC, and will then |
| | be grouped into each HLGT and will be further classified by PT. |
| | For SOC, data will be presented in the internationally agreed |
| Type of adverse events etc | order. For PT, data will be presented in ascending order of PT |
| Type of adverse events, etc. | codes. |
| | If the same patient has multiple occurrences of the same adverse |
| | event, etc. (PT), the total number of occurrences will be calculated |
| | per category (for example, if the same patient has one episode of |
| | serious diarrhea and one episode of non-serious diarrhea, these |
| | events will be counted once for each category). |

# (3) Figure/table number

Tables 5.2.1-1 to 5.2.1-3

# 5.2.2 Occurrence of adverse events/infections by CTCAE Grade (the worst one)

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse events, etc., will be analyzed:

| Data item | Category |
|------------------------|--------------------------------|
| CTCAE Grade (the worst | ≤Grade 2, ≥Grade 3, or unknown |
| one) | Solide 2, Solide 3, of unknown |

The type of adverse events, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse events, etc., by SOC/PT |
| Number of adverse events, | Number of adverse events, etc., observed by SOC/PT |
| etc. | |
| Type of adverse events, etc. | Adverse events, etc., will first be classified by SOC, within each |
| | of which adverse events, etc., will be further classified by PT. |
| | Laboratory test data will first be classified by SOC, and will then |
| | be grouped into each HLGT and will be further classified by PT. |
| | For SOC, data will be presented in the internationally agreed |

| order. For PT, data will be presented in ascending order of PT |
|------------------------------------------------------------------|
| codes. |
| If the same patient has multiple occurrences of the same adverse |
| event, etc. (PT), the event with the worst CTCAE grade will be |
| counted once. |

# (3) Figure/table number

Tables 5.2.2-1 to 5.2.2-3

# 5.2.3 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrence of adverse drug reactions/infections by outcome

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse drug reactions, etc., will be analyzed:

| Data item | Category |
|---|---|
| Seriousness | Serious or non-serious |
| CTCAE Grade (the worst | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| Time of onset | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, or ≥337 days |
| | 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly using a 21-day time window thereafter), 316 to 336 days, or ≥337 days |
| | 1 to 7 days, 8 to 14 days, 15 to 21 days, (segmented similarly using a 7-day time window thereafter), 330 to 336 days, or ≥337 days |
| Time to the worst grade | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, or ≥337 days |
| | 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly using a 21-day time window thereafter), 316 to 336 days, or ≥337 days |
| | 1 to 7 days, 8 to 14 days, 15 to 21 days, (segmented similarly using a 7-day time window thereafter), 330 to 336 days, or ≥337 days |
| Outcome | Recovered/resolved, recovering/resolving, not recovered/not resolved, recovered/resolved with sequelae, died/fatal, or unknown |

The type of adverse drug reactions, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse drug reactions, etc., by SOC/PT |
| Number of adverse drug reactions, etc. | Number of adverse drug reactions, etc., observed by SOC/PT |
| Type of adverse drug reactions, etc. | Adverse drug reactions, etc., will first be classified by SOC, within each of which adverse drug reactions, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be |

further classified by PT. For SOC, data will be presented in the internationally agreed order. For PT, data will be presented in ascending order of PT codes.

If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the total number of occurrences will be calculated per category (for example, if the same patient has one episode of serious diarrhea and one episode of non-serious diarrhea, these adverse drug reactions will be counted once for each category).

# (3) Figure/table number

Tables 5.2.3-1 to 5.2.3-3

#### 5.2.4 Occurrence of adverse drug reactions/infections by CTCAE Grade (the worst one)

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse drug reactions, etc., will be analyzed:

| Data item | Category |
|------------------------|-----------------------------------|
| CTCAE Grade (the worst | ≤Grade 2, ≥Grade 3, or unknown |
| one) | Solution 2, ≥Glade 3, of uliknown |

The type of adverse drug reactions, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse drug reactions, etc., by SOC/PT |
| Number of adverse drug reactions, etc. | Number of adverse drug reactions, etc., observed by SOC/PT |
| Type of adverse drug reactions, etc. | Adverse drug reactions, etc., will first be classified by SOC, within each of which adverse drug reactions, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. For SOC, data will be presented in the internationally agreed order. For PT, data will be presented in ascending order of PT codes. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the reaction with the worst CTCAE grade will be counted once. |

# (3) Figure/table number

Tables 5.2.4-1 to 5.2.4-3

# 5.3 Percentage of patients with adverse drug reactions/infections by patient demographics and baseline characteristics and treatment given

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the percentage of patients with adverse drug reactions, etc. (with point estimate and 95% confidence interval) will be determined.

For categories associated and not associated with ranking, Fisher's exact and Mann-Whitney U tests, respectively, will be used.

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| ALK (for patients with | |
| anaplastic large-cell | Positive, negative, or unknown |
| lymphoma) | |
| Clinical stage | I, II, III, IV, or unknown |
| B symptoms | Absent or present |
| ECOG Performance Status | 0, 1, 2, 3, or 4 |
| Past history of pulmonary disorders | Absent or present |
| Concurrent pulmonary disorders | Absent or present |
| Past history of malignant tumours | Absent or present |
| Concurrent malignant tumours | Absent or present |
| Concurrent hepatic disorders | Absent or present |
| Grade of hepatic disorder | |
| (CTCAE grade based on | None, Grade 1, Grade 2, or ≥Grade 3 |
| AST and ALT levels) | |
| Concurrent renal disorders | Absent or present |
| Grade of renal disorder | |
| (CTCAE grade based on | None, Grade 1, Grade 2, or ≥Grade 3 |
| serum creatinine) | |
| Weight | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, ≥70 kg, or not measured |
| BMI | $<18.5 \text{ kg/m}^2$ , $<18.5 \text{ to } 25 \text{ kg/m}^2$ , $<25 \text{ to } 30 \text{ kg/m}^2$ , $\ge 30 \text{ kg/m}^2$ , or unknown |
| Smoking history | Never, current, past, or unknown |
| Prior drug therapy | Absent or present |
| Prior radiotherapy | Absent or present |
| Prior hematopoietic stem cell transplantation | Absent, present (autologous), or present (homologous) |
| Initial dose of Adcetris | 1.8 mg/kg or other |
| Mean dose of Adcetris | <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg |

| Data item | Category |
|-----------------------------|--------------------------------------|
| Dose of Adcetris per 3 | <1.9 mg/kg, 1.9 mg/kg, or >1.9 mg/kg |
| weeks | <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg |
| Drug(s) other than Adcetris | |
| used for the treatment of | Absent or present |
| the primary disease | |

# (3) Figure/table number

Tables 5.3-1 to 5.3-3

# 5.4 Occurrence of adverse drug reactions/infections by age group

(1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

(2) Data to be analyzed

The type of adverse drug reactions, etc., will be analyzed by age group (<18 years, 18 to 64 years, 65 to 74 years, or  $\ge$ 75 years).

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Tables 5.4-1 to 5.4-3

5.5 Occurrence of adverse drug reactions/infections by presence or absence of concurrent hepatic disorder

(1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

(2) Data to be analyzed

The type of adverse drug reactions, etc., will be analyzed by presence or absence of concurrent hepatic disorder.

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Tables 5.5-1 to 5.5-3

- 5.6 Occurrence of adverse drug reactions/infections by presence or absence of concurrent renal disorder
  - (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

(2) Data to be analyzed

The type of adverse drug reactions, etc., will be analyzed by presence or absence of concurrent renal disorder.

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Tables 5.6-1 to 5.6-3

# 5.7 List of the occurrence of serious adverse events/infections

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

Data listed below will be analyzed.

| Data listed below will be alia Data item | Data to be analyzed |
|---|---|
| Number of patients with serious adverse events, | Number of patients experiencing serious adverse events, etc. |
| etc. | r value or panione original and some and value, over |
| | Number of serious adverse events, etc., observed |
| Number of serious | If the same patient has multiple occurrences of the same serious |
| adverse events, etc. | adverse event, etc. (PT), the total number of occurrences will be calculated. |
| Percentage of patients | Is calculated using the following formula: number of patients with |
| with serious adverse | serious adverse events, etc./number of patients included in the |
| events, etc. | safety analysis set × 100. |
| | Serious adverse events, etc., will first be classified by SOC, within |
| | each of which serious adverse events, etc., will be further classified |
| | by PT. Laboratory test data will first be classified by SOC, and will |
| | then be grouped into each HLGT and will be further classified by PT. |
| | For SOC, the number and percentage of patients with serious |
| Type of serious adverse | adverse events, etc., will be presented in the internationally agreed |
| events | order. |
| | For PT, the number and percentage of serious adverse events, etc., |
| | will be presented in ascending order of PT codes. |
| | If the same patient has multiple occurrences of the same serious |
| | adverse event, etc. (PT), the event will be counted once per patient. |
| | For serious adverse events, etc., considered not related to Adcetris, |
| | the number of these events will be presented in [ ]. |

# (3) Figure/table number

Tables 5.7-1 to 5.7-3

# 5.8 Change in test data over time

#### 5.8.1 Laboratory tests

(1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

Summary statistics of red blood cell count, hemoglobin level, white blood cell count, neutrophil count, lymphocyte count, platelet count, total bilirubin, AST, ALT, LDH, BUN, and serum creatinine will be calculated at each test time point [at baseline, after 1 cycle, ... and after 16 cycles].

# (3) Figure/table number

Tables 5.8.1-1 to 5.8.1-3

# 5.9 Analysis of items of particular interest

# 5.9.1 Occurrence of peripheral nerve disorder

(1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For CTCAE Grade (the worst one), patients will be stratified into the following categories, and the incidence of peripheral nerve disorders will be calculated:

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | |
| one) for peripheral nerve | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| disorders | |

Symptoms of peripheral nerve disorders will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Symptoms of peripheral nerve disorders | Peripheral nerve disorders will first be classified into peripheral sensory, peripheral motor, and peripheral neuropathies listed in Section 1.1, and symptoms associated with these peripheral nerve disorders will be analyzed by PT. If the same patient has multiple occurrences of the same symptom (PT), the symptom with the worst CTCAE grade will be counted once. |

# (3) Figure/table number

Tables 5.9.1-1 to 5.9.1-3

# 5.9.2 Occurrence of peripheral nerve disorders by patient demographics and baseline characteristics and treatment given

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For each data item, patients will be stratified into the categories below, and the incidence of peripheral nerve disorders will be calculated by CTCAE Grade (the worst one). If the same patient has multiple occurrences of the same peripheral nerve disorder (PT), the peripheral nerve disorder with the worst CTCAE grade will be counted once.

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| ECOG Performance Status | 0, 1, 2, 3, or 4 |
| Grade of concurrent peripheral nerve disorders | None, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |
| Weight | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, ≥70 kg, or not measured |
| Prior ABVD or CHOP | Absent or present |
| Prior radiotherapy | Absent or present |
| Prior hematopoietic stem cell transplantation | Absent, present (autologous), or present (homologous) |
| Initial dose of Adcetris | 1.8 mg/kg or other |
| Mean dose of Adcetris | <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg |
| Dose of Adcetris per 3 weeks | <1.8 mg/kg, 1.8 mg/kg, or >1.8 mg/kg |
| Concurrent diabetes mellitus | Absent or present |

# (3) Figure/table number

Tables 5.9.2-1 to 5.9.2-3

# 5.9.3 Treatment with Adcetris at the onset of peripheral nerve disorders

# (1) Analysis sets to be used

Patients included in the safety analysis set and safety analysis set (Hodgkin's lymphoma) or safety analysis set (anaplastic large-cell lymphoma) who experience peripheral nerve disorders considered related to Adcetris

# (2) Data to be analyzed

For each CTCAE Grade (the worst one) of peripheral nerve disorders, patients will be stratified into the categories below, and the number of peripheral nerve disorders will be calculated. If the same patient has multiple occurrences of the same peripheral nerve disorder (PT), the total number of occurrences will be calculated per category (for example, if the same patient has one episode of peripheral nerve disorder requiring dose reduction and one episode of peripheral nerve disorder leading to treatment discontinuation, these episodes of peripheral nerve disorder will be counted once for each category).

| 8 37 | |
|---|---|
| Data item | Category |
| Action taken to Adcetris | No action taken or action taken in response to the event |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), or |
| Adcetris | treatment discontinuation |

#### (3) Figure/table number

Tables 5.9.3-1 to 5.9.3-3

# 5.9.4 Occurrence of infections by presence or absence of drugs used for the prevention of infection

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

Patients will be stratified into the categories below and the number of patients with infection considered related to Adcetris will be calculated by presence or absence of drugs used for the prevention of infection using Mann-Whitney U test. If the same patient has multiple occurrences of the same infection, the occurrence with the worst CTCAE grade will be counted once.

Similarly, the number of patients with the onset of bacterial infection will be calculated by the use or non-use of antibiotics/synthetic antibacterial agents or trimethoprim-sulfamethoxazole combinations, the number of patients with the onset of fungal infection will be calculated by the use or non-use of antifungals, and the number of patients with the onset of viral infection will be calculated by the use or non-use of antivirals.

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | None, Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infections | |

#### (3) Figure/table number

Tables 5.9.4-1 to 5.9.4-3

# 5.9.5 Occurrence of neutropenia by patient demographics and baseline characteristics

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For each data item, patients will be stratified into the categories below, and the incidence of neutropenia considered related to Adcetris will be calculated by CTCAE Grade (the worst one). If the same patient has multiple occurrences of neutropenia, the event with the worst CTCAE grade will be counted once.

| Data item | Category |
|---|---|
| Prior hematopoietic stem | Absent, present (autologous), or present (homologous) |
| cell transplantation | |
| Degree of decreased | No decrease, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |
| neutrophil count at baseline | No decrease, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |

# (3) Figure/table number

Tables 5.9.5-1 to 5.9.5-3

#### 5.9.6 Treatment with Adcetris at the onset of neutropenia

#### (1) Analysis sets to be used

Patients included in the safety analysis set and safety analysis set (Hodgkin's lymphoma) or safety analysis set (anaplastic large-cell lymphoma) who experience neutropenia considered related to Adcetris

# (2) Data to be analyzed

For each CTCAE Grade (the worst one) of neutropenia, patients will be stratified into the categories below, and the number of events of neutropenia will be calculated. If the same patient has multiple occurrences of neutropenia, the total number of occurrences will be calculated per category (for example, if the same patient has one episode of peripheral nerve disorder requiring dose reduction and one episode of peripheral nerve disorder leading to treatment discontinuation, these episodes of peripheral nerve disorder will be counted once for each category).

| Data item | Category |
|---|---|
| Action taken to Adcetris | No action taken or action taken in response to the event |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), or |
| Adcetris | treatment discontinuation |

# (3) Figure/table number

Tables 5.9.6-1 to 5.9.6-3

#### 5.9.7 Occurrence of infusion reaction

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For CTCAE Grade (the worst one), patients will be stratified into the following categories, and the incidence of infusion reaction considered related to Adcetris will be calculated:

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infusion reaction | |

Infusion reaction will be analyzed as follows:

| Data iter | n | Data to be analyzed |
|---|---|---|
| | | Infusion reaction and its symptoms will be analyzed by PT. |
| Symptoms of | infusion | If the same patient has multiple occurrences of the same symptom |
| reaction | | (PT), the symptom with the worst CTCAE grade will be counted |
| | | once. |

#### (3) Figure/table number

Tables 5.9.7-1 to 5.9.7-3

# 5.9.8 Occurrence of infusion reaction by the use or non-use of premedication to prevent infusion reaction

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

Patients will be stratified into the following categories and the number of events of infusion reaction considered related to Adcetris will be calculated by the use or non-use of premedication to prevent infusion reaction (for example, if a patient receives no premedication and experiences "Grade 2" infusion reaction during Cycle 1 and receives premedication and experiences no infusion reaction during Cycle 2, these events of infusion reaction will be counted once for each category).

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | None, Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infusion reaction | |

# (3) Figure/table number

Tables 5.9.8-1 to 5.9.8-3

#### 5.9.9 Occurrence of pulmonary disorders

# (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

For CTCAE Grade (the worst one), patients will be stratified into the following categories, and the incidence of events of pulmonary disorder considered related to Adcetris will be calculated:

| Data item | | em | Category |
|---|---|---|---|
| CTCAE | Grade | (the worst | |
| one) | for | pulmonary | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| disorders | 5 | | |

Diagnoses or symptoms of pulmonary disorder will be analyzed as follows:

| <u> </u> | j j |
|---|---|
| Data item | Data to be analyzed |
| | Pulmonary disorders and their diagnoses or symptoms will be |
| Diagnosis or symptom of | analyzed by PT. |
| | If the same patient has multiple occurrences of the same symptom |
| pulmonary disorder | (PT), the symptom with the worst CTCAE grade will be counted |
| | once. |

# (3) Figure/table number

Tables 5.9.9-1 to 5.9.9-3

# 5.10 Occurrence of infections by presence or absence of hematopoietic stem cell transplantation

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

# (2) Data to be analyzed

Patients will be stratified into the categories below and the number of patients with infection considered related to Adcetris will be calculated by presence or absence of prior hematopoietic stem cell transplantation (Absent, present [autologous], or present [homologous]) using Mann-Whitney U test. If the same patient has multiple occurrences of the same infection, the occurrence with the worst CTCAE grade will be counted once.

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | None, Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infections | |

# (3) Figure/table number

Tables 5.10-1 to 5.10-3

# 5.11 List of actions taken with Adcetris in patients experiencing peripheral nerve disorders

(1) Analysis sets to be used

Patients included in the safety analysis set and safety analysis set (Hodgkin's lymphoma) or safety analysis set (anaplastic large-cell lymphoma) who experience peripheral nerve disorders considered related to Adcetris

#### (2) Data to be analyzed

For each patient, actions taken or not taken with Adcetris, specific action(s) taken, date of dosing and dose for each cycle, date of onset of peripheral nerve disorders, outcome, and date of outcome will be presented. If the same patient has multiple occurrences of peripheral nerve disorder, all the occurrences will be counted.

# (3) Figure/table number

Tables 5.11-1 to 5.11-3

# 5.12 List of actions taken with Adcetris in patients experiencing neutropenia

### (1) Analysis sets to be used

Patients included in the safety analysis set and safety analysis set (Hodgkin's lymphoma) or safety analysis set (anaplastic large-cell lymphoma) who experience neutropenia considered related to Adcetris

## (2) Data to be analyzed

For each patient, actions taken or not taken with Adcetris, specific action(s) taken, date of dosing and dose for each cycle, date of onset of neutropenia, outcome, and date of outcome will be presented. If the same patient has multiple occurrences of neutropenia, all the occurrences will be counted.

#### (3) Figure/table number

Tables 5.12-1 to 5.12-3

# 6.0 Efficacy Analysis

# 6.1 Best response

(1) Analysis set to be used

Efficacy analysis set

(2) Data to be analyzed

The best responses after 16 cycles of treatment with Adcetris (or upon discontinuation of treatment with Adcetris) will be analyzed in patients Hodgkin's lymphoma and patients with anaplastic large-cell lymphoma.

(3) Figure/table number

Table 6.1

#### 6.2 Overall survival

(1) Analysis set to be used

Efficacy analysis set

(2) Data to be analyzed

The survivals from the date of the initial dose of Adcetris in patients Hodgkin's lymphoma and patients with anaplastic large-cell lymphoma will be calculated, using the final observation date as the date of survival confirmation and the date of outcome of an adverse event with "Died/fetal" recorded in the Outcome field as the date of death.

Kaplan-Meier curves of the survival will also be constructed (i.e., a table of the numbers of adverse events, etc., and adverse drug reactions, etc., printed out by SAS will be attached).

(3) Figure/table number

Table 6.2 and Figure 6.2

# Appendix: Definition of Pulmonary Disorders (MedDRA Preferred Terms)

The above definition is consistent with the one used in clinical studies of Adcetris.

# Statistical Analysis Plan

# ADCETRIS IV Infusion – Special Drug Use Surveillance (All-case Surveillance) "Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell Lymphoma"

| PPD | |
|-----|---------------------------------------|
| | Takeda Pharmaceutical Company Limited |
| PPD | |
| | tistical Analysis Agent |
| PPD | |

# Table of Contents

| 1.0 | Definition of Terms and Handling of Test/Measurement Data | 1 |
|---|---|---|
| 1.1 | Definition | 1 |
| 1.2 | Display digits | 7 |
| 1.3 | Level of significance. | 7 |
| 1.4 | Handling of test data | 7 |
| 2.0 | Patient Disposition (Patient Disposition Diagram) | 9 |
| 3.0 | Patient Demographics and Baseline Characteristics | 10 |
| 4.0 | Treatment Given | 13 |
| 4.1 | Treatment given | 13 |
| 4.2 | Premedication to prevent infusion reaction | 14 |
| 5.0 | Safety Analysis | 15 |
| 5.1 | Occurrences of adverse events/infections and adverse drug reactions/infections | 15 |
| 5.1 | 1.1 Occurrence of adverse events/infections | 15 |
| 5.1 | 1.2 Occurrence of adverse drug reactions/infections | 16 |
| 5.2 | Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrent | nces of |
| | adverse events/infections and adverse drug reactions/infections by outcome | 16 |
| 5.2 | 2.1 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occur | ırrence |
| of | adverse events/infections by outcome | 16 |
| 5.2 | Occurrence of adverse events/infections by CTCAE Grade (the worst one) | 17 |
| 5.2 | 2.3 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occur | ırrence |
| of | adverse drug reactions/infections by outcome | 19 |
| 5.2 | Occurrence of adverse drug reactions/infections by CTCAE Grade (the worst one) | 20 |
| 5.3 | Percentage of patients with adverse drug reactions/infections by patient demographics and ba | aseline |
| | characteristics and treatment given | 20 |
| 5.4 | Occurrence of adverse drug reactions/infections by age group | 23 |
| 5.5 | Occurrence of adverse drug reactions/infections by presence or absence of concurrent hepatic di | isorder |
| | | 23 |
| 5.6 | Occurrence of adverse drug reactions/infections by presence or absence of concurrent renal disord | er 23 |
| 5.7 | List of the occurrence of serious adverse events/infections | 24 |
| 5.8 | Change in test data over time | 25 |
| 5.8 | 3.1 Laboratory tests | 25 |
| 5.9 | Analysis of items of particular interest | 25 |
| 5.9 | Occurrence of peripheral nerve disorder | 25 |
| 5.9 | Occurrence of peripheral nerve disorders by patient demographics and baseline characteristi | cs and |
| trea | atment given | 26 |
| 5.9 | 7.3 Treatment with Adcetris at the onset of peripheral nerve disorders | 27 |
| 5.9 | | |
| 5.9 | Occurrence of neutropenia by patient demographics and baseline characteristics | 28 |

| 5.9.0 | 6 | Treatment with Adcetris at the onset of neutropenia. | 28 |
|---|---|---|---|
| 5.9. | 7 | Occurrence of infusion reaction. | 29 |
| 5.9.8 | 8 | Occurrence of infusion reaction by the use or non-use of premedication to prevent infusion reaction | ection |
| | | 29 | |
| 5.9.9 | 9 | Occurrence of pulmonary disorders | 30 |
| 6.0 | Effic | cacy Analysis | 31 |
| 6.1 | Best | response | 31 |
| 6.2 | 2 Overall survival | | |
| Appendic | ces | | 2 |

# 1.0 Definition of Terms and Handling of Test/Measurement Data

# 1.1 Definition

| Term | Definition |
|---|---|
| This/the product | Refers to Adcetris for intravenous drip infusion in this Statistical Analysis |
| | Plan. |
| SOC | MedDRA/J System Organ Class |
| HLGT | MedDRA/J High Level Group Term |
| PT | MedDRA/J Preferred Term |
| LLT | MedDRA/J Lowest Level Term |
| Patients registered | Patients whose registration has been approved |
| Patients whose case report | Patients whose case report forms have been collected |
| forms are available | |
| Patients whose case report | Patients registered but whose case report form have not been collected |
| forms are not available | |
| Fixed patients | Patients whose case report forms are available, with the date of case report |
| | form completion entered in the PMS system |
| Non-fixed patients | Patients whose case report forms are available, with the date of case report |
| | form completion not entered in the PMS system |
| Safety analysis set | Fixed patients included in the safety analysis set |
| Patients excluded from the | Fixed patients excluded from the safety analysis set |
| safety analysis set | |
| Efficacy analysis set | Patients included in the safety analysis set who are also included in the |
| | efficacy analysis set |
| Patients excluded from the | Patients included in the safety analysis set who are excluded from the |
| efficacy analysis set | efficacy analysis set |
| Patients completing treatment | Patients completing 16 cycles of treatment with Adcetris |
| Patients discontinuing treatment | Patients not completing 16 cycles of treatment with Adcetris |
| Adverse events, etc. | Refers to "adverse events and infections." |
| | In this Statistical Analysis Plan, the term "adverse events and infections" |
| | is used in titles and the term "adverse events, etc." is used in text and |
| | tables. |
| Adverse drug reactions, etc. | Refers to "adverse drug reactions and infections." |
| | Adverse events, etc., not considered "not related" to Adcetris by the |
| | investigator. |
| | In this Statistical Analysis Plan, the term "adverse drug reactions and |
| | infections" is used in titles and the term "adverse drug reactions, etc." is |
| | used in text and tables. |
| Serious adverse events, etc. | Refers to "serious adverse events and infections." |

| Term | Definition |
|---|---|
| | Adverse events considered "serious" by the investigator. |
| | Events listed in the MedDRA Coding List in the Takeda Medically |
| | Significant AE List should be regarded as serious even if they are |
| | considered "non-serious" by the investigator. |
| | In this Statistical Analysis Plan, the term "serious adverse events and |
| | infections" is used in titles and the term "serious adverse events, etc." is |
| | used in text and tables. |
| Number of patients with | Number of patients experiencing adverse events, etc., or adverse drug |
| adverse events/adverse drug | reactions, etc. |
| reactions | |
| Number of adverse | Number of adverse events, etc., or adverse drug reactions, etc., observed |
| events/adverse drug reactions | |
| Percentage of patients with | [For safety analysis using patients included in the safety analysis set] |
| adverse events/adverse drug | Is calculated using the following formula: (number of patients with |
| reactions | adverse events/adverse drug reactions) / (number of patients included in |
| | the safety analysis set) $\times$ 100. |
| | [For safety analysis using patients excluded from the safety analysis set] |
| | Is calculated using the following formula: (number of patients with |
| | adverse events/adverse drug reactions) / (number of patients excluded |
| | from the safety analysis set) × 100. |
| Percentage of adverse | [For safety analysis using patients included in the safety analysis set] |
| events/adverse drug reactions | Is calculated using the following formula: (number of adverse |
| observed | events/adverse drug reactions observed) / (number of patients included in |
| observed | the safety analysis set) × 100. |
| | [For safety analysis using patients excluded from the safety analysis set] |
| | Is calculated using the following formula: (number of adverse |
| | • |
| | events/adverse drug reactions observed) / (number of patients excluded from the sofety analysis set) × 100 |
| Time of onset | from the safety analysis set) × 100. |
| Time of onset | Is calculated using the following formula: date of onset of adverse events, |
| | etc. (or adverse drug reactions, etc.) – date of the initial dose of Adcetris + |
| | If the day and month of onset of adverse events, etc. (or adverse drug |
| | reactions, etc.) are unknown, the date of onset should be "January 1." |
| | However, if the year of the initial dose of Adcetris is the year of onset of |
| | adverse events, etc. (or adverse drug reactions, etc.), the date of onset |
| | should be the day and month of the initial dose of Adcetris. |
| | If the day of onset of adverse events, etc. (or adverse drug reactions, etc.) |
| | is unknown, the date of onset should be the first day of the month. |
| | However, if the year and month of the initial dose of Adcetris is the year |

| Term | Definition |
|---|---|
| | and month of onset of adverse events, etc. (or adverse drug reactions, etc.), |
| | the date of the initial dose of Adcetris should be the date of onset. |
| Patients with concurrent hepatic | Patients having a concurrent illness that falls under the category of |
| disorder | Standardized MedDRA Query (SMQ) Code 20000005 (SMQ Hepatic |
| | disorders [Scope: Narrow]) |
| Patients with concurrent renal | Patients having a concurrent illness that falls under the category of Takeda |
| disorder | MedDRA Query (TMQ) (Renal disorders) |
| Patients with a past history of | Patients with a past history that falls under the category of Appendix |
| pulmonary disorder | "Definition of Pulmonary Disorders" |
| | (If "No concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | pulmonary disorders" in the case report form, the pulmonary disorder |
| | should be regarded as a past history.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of Appendix |
| pulmonary disorder | "Definition of Pulmonary Disorders" |
| | (If "A concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | pulmonary disorders" in the case report form, the pulmonary disorder |
| | should be regarded as a concurrent illness.) |
| Patients with a past history of | Patients with a past history that falls under the category of MedDRA SMQ |
| malignant tumour | Code 20000194 (SMQ Malignant tumours [Scope: Narrow]) |
| | (If "No concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | malignant tumours" in the case report form, the pulmonary disorder should |
| | be regarded as a past history.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| malignant tumour | SMQ Code 20000194 (SMQ Malignant tumours [Scope: Narrow]) |
| | (If "A concurrent illness existed at the initiation of treatment with |
| | Adcetris" is selected in the field of "Past history/concurrent illness of |
| | malignant tumours" in the case report form, the pulmonary disorder should |
| | be as a concurrent illness.) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| diabetes mellitus | SMQ Code 20000041 (SMQ Hyperglycaemia/new onset diabetes mellitus |
| | [Scope: Narrow]) |
| Patients with hypertension | Patients with a concurrent illness that falls under the category of MedDRA |
| | SMQ Code 20000147 (SMQ Hypertension [Scope: Narrow]) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| dyslipidaemia | SMQ Code 20000026 (SMQ Dyslipidaemia [Scope: Narrow]) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |

| Term | Definition |
|---|---|
| hyperuricaemia | PT Code 10020903 (Hyperuricaemia) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of MedDRA |
| infection | SOC Code 10021881 (Infections and infestations) |
| Patients with concurrent | Patients with a concurrent illness that falls under the category of SMQ |
| peripheral neuropathy | Code 20000034 (SMQ Peripheral neuropathy [Scope: Narrow]) |
| Patients with other concurrent | Patients with any concurrent illness other than those listed above |
| illnesses | |
| Antibiotics/synthetic | Prophylactics against infections that fall under the category of those with |
| antibacterial agents | the first three digits of YJ Code being 611 to 616 or 619 (If more than one |
| | antibiotics/synthetic antibacterial agents are used in the same patient, it |
| | will be counted as one patient.) |
| Antifungals | Prophylactics against infections that fall under the category of those with |
| | the first three digits of YJ Code being 617 (If more than one antifungals |
| | are used in the same patient, it will be counted as one patient.) |
| Antivirals | Prophylactics against infections that fall under the category of those with |
| | the first three digits of YJ Code being 625 (If more than one antivirals are |
| | used in the same patient, it will be counted as one patient.) |
| Trimethoprim-sulfamethoxazole | Prophylactics against infections that fall under the category of those with |
| combinations | YJ Code being 629010007 to 9 |
| Other prophylactics against | Any drug entered in the field of "Drugs used for the prevention of |
| infections | infection" other than prophylactics against infections listed above (If more |
| | than one other prophylactics against infections are used in the same |
| | patient, it will be counted as one patient.) |
| Peripheral sensory neuropathy | Adverse events with "Sensory neuropathy" entered in the "Category of |
| (as an adverse event) | peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral |
| | nerve disorders] in the case report form. MedDRA PT Code 10034620 |
| | should be assigned regardless of data entered in "Symptoms" in the field. |
| Peripheral motor neuropathy | Adverse events with "Motor neuropathy" entered in the "Category of |
| (as an adverse event) | peripheral nerve disorders" in the field of "Adverse events: [1] Peripheral |
| | nerve disorders] in the case report form. MedDRA PT Code 10034580 |
| | should be assigned regardless of data entered in "Symptoms" in the field. |
| Peripheral neuropathy | Adverse events with "Other" entered in the "Category of peripheral nerve |
| (as an adverse event) | disorders" in the field of "Adverse events: [1] Peripheral nerve disorders] |
| | in the case report form. MedDRA PT Code 10029331 should be assigned, |
| | regardless of data entered in "Symptoms" in the field. |
| Pulmonary disorders | Adverse events that fall under the category of Appendix "Definition of |
| (as adverse events) | Pulmonary Disorders" |
| Infusion reaction | Adverse events entered in the field of "Adverse events: [4] Infusion |
| | reaction," regardless of data entered in "Symptoms" in the field. |

| Term | Definition |
|---|---|
| Patients with the onset of | Patients with adverse drug reactions that fall under the category of |
| infection | MedDRA SOC Code 10021881 (Infections and infestations) |
| Patients with the onset of | Patients with adverse drug reactions that fall under the category of |
| bacterial infection | MedDRA HGLT Code 10004018 (Bacterial infection), 10008555 |
| | (Chlamydial infection), 10028474 (Mycoplasma infection) or 10039135 |
| | (Rickettsia infection) |
| Patients with the onset of fungal | Patients with adverse drug reactions that fall under the category of |
| infection | MedDRA HGLT Code 10017528 (Fungal infection) |
| Patients with the onset of viral | Patients with adverse drug reactions that fall under the category of |
| infection | MedDRA HGLT Code 10047438 (Viral infection) |
| Age | If the month and day of the initial dose of Adcetris is < the month and day |
| | of birth, the patient's age will be calculated using the following formula: |
| | Year of the initial dose of Adcetris – year of birth – 1. |
| | If the month and day of the initial dose of Adcetris is $\geq$ the month and day |
| | of birth, the patient's age will be calculated using the following formula: |
| | Year of the initial dose of Adcetris – year of birth. |
| | If the month and day of birth are unknown, they should be "January 1," |
| | and if the day of birth is unknown, it should the first day of the month. |
| BMI | BMI should be calculated using the following formula: Weight (kg) / |
| | $(0.0001 \times \text{height (cm}) \times \text{height (cm)}$ . The obtained value should be |
| | rounded off to one decimal place. |
| Disease duration | The disease duration should be calculated using the following formula: |
| | ["Date of the initial dose of Adcetris" – "date of diagnosis of Hodgkin's or |
| | anaplastic large-cell lymphoma" +1] / 365.25. |
| | The day of diagnosis should be the first day of the month provided. If the |
| | month of diagnosis is unknown, the date of diagnosis should be "January |
| | 1st" of the year provided. |
| Mean dose of Adcetris | Is calculated as the total value of each dose of Adcetris given at each |
| | treatment cycle divided by the number of cycles. |
| Dose of Adcetris per 3 weeks | Is calculated using the following formula: Total "dose of Adcetris" / |
| | (["date of the last dose of Adcetris" – "date of the initial dose of Adcetris" |
| | + 21)/21]. |
| | If only 1 cycle of treatment is given, the "date of the last dose of Adcetris" |
| | and the "date of the initial dose of Adcetris" should be regarded as the |
| D | same. |
| Degree of decreased neutrophil | Neutrophil count at baseline ≥2,000 /mm <sup>3</sup> |
| count at baseline: No decrease | No describing a service of 2000 to 1,500 / 3 |
| Degree of decreased neutrophil | Neutrophil count at baseline <2,000 to 1,500 /mm <sup>3</sup> |
| count at baseline: Grade 1 | |

| Term | Definition |
|---|---|
| Degree of decreased neutrophil | Neutrophil count at baseline <1,500 to 1,000 /mm <sup>3</sup> |
| count at baseline: Grade 2 | |
| Degree of decreased neutrophil | Neutrophil count at baseline <1,000 to 500 /mm <sup>3</sup> |
| count at baseline: Grade 3 | |
| Degree of decreased neutrophil | Neutrophil count at baseline <500 /mm <sup>3</sup> |
| count at baseline: Grade 4 | |
| Date of the final observation | "Date of the final observation" in the case report form |
| | If not provided, the most recent date entered in the case report form should |
| | be used. |
| Summary statistics | Includes mean, standard deviation, minimum, 25th percentile, median, |
| | 75th percentile, and maximum. |

# 1.2 Display digits

| Term | Definition |
|---|---|
| Percentage (%) | Percentage of patients with or percentage of adverse events, etc., or adverse drug |
| | reactions, etc.: |
| | The obtained value should be rounded off to two decimal places. |
| | Other: |
| | The obtained value should be rounded off to one decimal place. |
| Summary statistics | Mean: |
| (mean and standard | The raw data should be rounded off to one decimal place. |
| deviation) | Standard deviation: |
| | The raw data should be rounded off to two decimal places. |
| P value | The obtained value should be rounded down to three decimal places. |
| | If the value is less than 0.001 after rounding down to three decimal places, it |
| | should be displayed as "p<0.001." |

# 1.3 Level of significance

Two-sided 5%

# 1.4 Handling of test data

Test data will be handled according to the criteria shown below. If there are multiple data for the same criterion, the one with the test date being closest to the date of protocol-specified assessment should be used. If there is no difference in the number of days from the date of protocol-specified assessment, the later value should be used. For the final assessment, \*however, the most recently measured value (including the one measured during the off-treatment period) after the date of the initial dose of Adcetris should be used. Values measured after 30 days after the last dose of Adcetris should not be used.

The number of days after the date of the initial dose of Adcetris is defined as 1 for the date of the initial dose of Adcetris and 0 for the day before the date of the initial dose of Adcetris.

\*After 16 cycles of treatment with Adcetris (or upon discontinuation of treatment with Adcetris)

| Time point for testing | Acceptable time window | Date of protocol-specified assessment |
|---|---|---|
| At the initial dose of | -21 to 1 days | Date of the initial dose of Adcetris |
| Adcetris | | |
| After 1 cycle | 2 to 31 days | Date of the initial dose of Adcetris + 21 |
| After 2 cycles | 32 to 52 days | Date of the initial dose of Adcetris + 42 |
| After 3 cycles | 53 to 73 days | Date of the initial dose of Adcetris + 63 |
| After 4 cycles | 74 to 94 days | Date of the initial dose of Adcetris + 84 |
| After 5 cycles | 95 to 115 days | Date of the initial dose of Adcetris + 105 |
| After 6 cycles | 116 to 136 days | Date of the initial dose of Adcetris + 126 |
| After 7 cycles | 137 to 157 days | Date of the initial dose of Adcetris + 147 |

| Time point for testing | Acceptable time window | Date of protocol-specified assessment |
|---|---|---|
| After 8 cycles | 158 to 178 days | Date of the initial dose of Adcetris + 168 |
| After 9 cycles | 179 to 199 days | Date of the initial dose of Adcetris + 189 |
| After 10 cycles | 200 to 220 days | Date of the initial dose of Adcetris + 210 |
| After 11 cycles | 221 to 241 days | Date of the initial dose of Adcetris + 231 |
| After 12 cycles | 242 to 262 days | Date of the initial dose of Adcetris + 252 |
| After 13 cycles | 263 to 283 days | Date of the initial dose of Adcetris + 273 |
| After 14 cycles | 284 to 304 days | Date of the initial dose of Adcetris + 294 |
| After 15 cycles | 305 to 325 days | Date of the initial dose of Adcetris + 315 |
| After 16 cycles | 326 to 346 days | Date of the initial dose of Adcetris + 336 |

# 2.0 Patient Disposition (Patient Disposition Diagram)

# (1) Analysis set to be used

Patients registered to this specified drug-use survey

#### (2) Data to be analyzed

Data to be analyzed includes the numbers of patients registered, institutions with patients registered, patients whose case report forms are available/not available, fixed/non-fixed patients, patients included in/excluded from the safety analysis set, and patients included in/excluded from the efficacy analysis set.

For the number of institutions with patients registered, the same institutions with different departments should not be counted more than once.

For patients whose case report forms are not available, the number of patients by reason for unavailability and the total number of patients will be calculated.

For patients excluded from the safety/efficacy analysis set, the number of patients by reason for exclusion and the total number of patients will be calculated.

It will be determined as follows whether patients meeting the following criteria should be included or excluded:

| Criterion | Registration | Safety<br>evaluation | Efficacy evaluation |
|---|---|---|---|
| Duplicate registration (of the same patient) | 0 | × | × |
| [found afterwards] | | | |
| Non-primary disease | 0 | 0 | × |
| Adcetris has never been administered [found | 0 | × | × |
| afterwards] | | | |
| No definite safety evaluation results are | 0 | × | × |
| available | | | |
| No definite efficacy evaluation results are | 0 | 0 | × |
| available | | | |
| No case report form is available | 0 | × | × |

o: Included, ×: Excluded

# (3) Figure/table number

Figure 2.0-1 and Table 2.0-1

# 3.0 Patient Demographics and Baseline Characteristics

(1) Analysis set to be used
Safety analysis set

# (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the number and frequency of patients will be calculated:

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | Summary statistics |
| | <18 years, 18 to 39 years, 40 to 64 years, 65 to 74 years, or ≥75 years |
| | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| Diagnosis | Hodgkin's or anaplastic large-cell lymphoma or other |
| Status | Relapsed/refractory, or new-onset |
| CD30 | Positive, negative, or not measured |
| Site(s) of involvement | Lymph node, spleen, liver, lung, bone, central nerve, bone marrow, skin, and/or other |
| ALK (for patients with anaplastic large-cell lymphoma) | Positive, negative, or unknown |
| Clinical stage | I, II, III, IV, or unknown |
| B symptoms | Absent or present |
| ECOG Performance<br>Status | 0, 1, 2, 3, or 4 |
| Therapeutic category | Outpatient or inpatient |
| Hypersensitivity disposition | Absent, present, or unknown |
| Specific hypersensitivity disposition(s) | Medications, food allergy, and/or other |
| HCV antibody | Negative, positive, or unknown |
| HBs antigen | Negative, positive, or unknown |
| HBs antibody | Negative, positive, or unknown |
| HBV DNA | Negative, positive, or unknown |
| Past history of pulmonary disorders | Absent or present |
| Concurrent pulmonary disorders | Absent or present |
| Past history of | Absent or present |

| Data item | Category |
|---|---|
| malignant tumours | |
| Concurrent malignant | Absent or present |
| tumours | |
| Concurrent illness | |
| (other than pulmonary | Absent or present |
| disorders and | Atosent of present |
| malignant tumours) | |
| Specific concurrent illness(es) (other than pulmonary disorders and malignant tumours) | Diabetes mellitus, hypertension, dyslipidaemia, hyperuricaemia, hepatic disease(s), renal disease(s), infections, peripheral nerve disorders, and/or other |
| Past history (other than pulmonary disorders and malignant tumours) | Absent, present, or unknown |
| Weight | Summary statistics |
| | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, ≥70 kg, or not |
| | measured |
| BMI | Summary statistics |
| Divii | <18.5, <18.5 to 25, <25 to 30, ≥30, or unknown |
| Smoking history | Never, current, past, or unknown |
| Prior drug therapy | Absent or present |
| Prior drug therapy | ABVD, CHOP, and/or other |
| regimen(s) | (If more than one drug therapies in the same category is used in the |
| | same patient, it will be counted as one patient.) |
| Number of prior drug | Summary statistics |
| therapy regimens | |
| Prior radiotherapy | Absent or present |
| Prior hematopoietic | |
| stem cell | Absent, present (autologous), or present (homologous) |
| transplantation Other prior therepies | A broad on amorph |
| Other prior therapies | Absent or present |
| Pregnancy during the | Abcont or present |
| observation period | Absent or present |
| (for females only) | |

# (3) Figure/table number

# 4.0 Treatment Given

# 4.1 Treatment given

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the number and frequency of patients will be calculated:

| Data item | Category |
|---|---|
| Initial dose of<br>Adcetris | 1.8 mg/kg or other |
| Mean dose of Adcetris | <1.8 mg/kg, 1.8 mg/kg, or ≥1.8 mg/kg |
| Dose of Adcetris per 3 weeks | <1.8 mg/kg, 1.8 mg/kg, or ≥1.8 mg/kg |
| Duration of treatment with Adcetris | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, or 16 cycles |
| Reason(s) for discontinuation of Adcetris | Treatment goal achieved, adverse event(s), lost to follow-up, transfer to another hospital, pregnancy, inadequate response, and/or other |
| Post-baseline<br>hematopoietic stem<br>cell transplantation | Absent or present |
| Type of post-baseline<br>hematopoietic stem<br>cell transplantation | Autologous or homologous |
| Drug(s) other than Adcetris used for the treatment of the primary disease | Absent or present |
| Drug(s) used for the prevention of infection | Absent or present |
| Specific drug(s) used for the prevention of infection | Antibiotics/synthetic antibacterial agents, antifungals, antivirals, trimethoprim-sulfamethoxazole combinations, and/or other prophylactics against infections |

# (3) Figure/table number

Table 4.1-1
#### 4.2 Premedication to prevent infusion reaction

(1) Analysis set to be used

Safety analysis set

#### (2) Data to be analyzed

For each cycle, patients will be stratified into the following categories, and the number and frequency of patients will be calculated:

| Data item | Category |
|---|---|
| Premedication to prevent infusion reaction | Absent or present |
| Specific premedication(s) used to prevent infusion reaction | Acetaminophen, antihistamines, and/or corticosteroids |

#### (3) Figure/table number

Table 4.2-1

#### 5.0 Safety Analysis

#### 5.1 Occurrences of adverse events/infections and adverse drug reactions/infections

#### 5.1.1 Occurrence of adverse events/infections

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

Data listed below will be analyzed.

For data entered in the field of "Adverse events: [1] Peripheral nerve disorders] in the case report form, MedDRA PT Code for peripheral sensory neuropathy, peripheral motor neuropathy, or peripheral neuropathy should be assigned, regardless of the LLT code entered in "Symptoms" field (see Section 1.1 "Definition;" the same applies hereinafter).

Neutropenia (PT Code 10029354) will be assigned to Neutrophil count decreased (LLT Code 10029366), Lymphopenia (PT Code 10025327) to Lymphocyte count decreased (LLT Code 10025256), Leukopenia (PT Code 10024384) to White blood cell count decreased (LLT Code 10047942), and Thrombocytopenia (PT Code 10043554) to Platelet count decreased (LLT Code 10035528) (the same applies hereinafter).

| Data item | Data to be analyzed |
|---|---|
| Number of patients with adverse events, etc. | Number of patients experiencing adverse events, etc. |
| Number of adverse events, etc. | Number of adverse events, etc., observed If the same patient has multiple occurrences of the same adverse event, etc. (PT), the total number of occurrences will be calculated. |
| Percentage of patients with adverse events, etc. | Is calculated using the following formula: number of patients with adverse events, etc./number of patients included in the safety analysis set $\times$ 100. |
| Type of adverse events, etc. | Adverse events, etc., will first be classified by SOC, within each of which adverse events, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. For SOC, the number and percentage of patients with adverse events, etc., will be presented in the internationally agreed order. For PT, the number and percentage of adverse events, etc., will be presented in ascending order of PT codes. If the same patient has multiple occurrences of the same adverse event, etc. (PT), the event will be counted once per patient. |

#### (3) Figure/table number

Table 5.1-1

#### 5.1.2 Occurrence of adverse drug reactions/infections

(1) Analysis set to be used
Safety analysis set

(2) Data to be analyzed

Data listed below will be analyzed.

| Data item | Data to be analyzed |
|---|---|
| Number of patients with adverse drug reactions, etc. | Number of patients experiencing adverse drug reactions, etc. |
| Number of adverse drug reactions, etc. | Number of adverse drug reactions, etc., observed. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the total number of occurrences will be calculated. |
| Percentage of patients with adverse drug reactions, etc. | Is calculated using the following formula: number of patients with adverse drug reactions, etc./number of patients included in the safety analysis set $\times$ 100. |
| Type of adverse drug reactions, etc. | Adverse drug reactions, etc., will first be classified by SOC, within each of which adverse drug reactions, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. For SOC, the number and percentage of patients with adverse drug reactions, etc., will be presented in the internationally agreed order. For PT, the number and percentage of adverse drug reactions, etc., will be presented in ascending order of PT codes. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the reaction will be counted once per patient. |

(3) Figure/table number

Table 5.1-2

- 5.2 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrences of adverse events/infections and adverse drug reactions/infections by outcome
  - 5.2.1 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrence of adverse events/infections by outcome
    - (1) Analysis set to be used
      Safety analysis set
    - (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse events, etc., will be analyzed:

| Data item | Category |
|-----------|----------|
|-----------|----------|

| Seriousness | Serious or non-serious |
|---|---|
| CTCAE Grade (the worst one) | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| Time of onset | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, or ≥337 days |
| Time to the worst grade | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, or ≥337 days |
| Outcome | Recovered/resolved, recovering/resolving, not recovered/not resolved, recovered/resolved with sequelae, died/fatal, or unknown |

The type of adverse events, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse events, etc., by SOC/PT |
| Number of adverse events, etc. | Number of adverse events, etc., observed by SOC/PT |
| Type of adverse events, etc. | Adverse events, etc., will first be classified by SOC, within each of which adverse events, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. For SOC, data will be presented in the internationally agreed order. For PT, data will be presented in ascending order of PT codes. If the same patient has multiple occurrences of the same adverse event, etc. (PT), the total number of occurrences will be calculated per category (for example, if the same patient has one episode of serious diarrhea and one episode of non-serious diarrhea, these events will be counted once for each category). |

#### (3) Figure/table number

Table 5.2-1

#### 5.2.2 Occurrence of adverse events/infections by CTCAE Grade (the worst one)

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse events, etc., will be analyzed:

| Data item | Category |
|------------------------|--------------------------------|
| CTCAE Grade (the worst | ≤Grade 2, ≥Grade 3, or unknown |
| one) | |

The type of adverse events, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse events, etc., by SOC/PT |
| Number of adverse events, etc. | Number of adverse events, etc., observed by SOC/PT |
| | Adverse events, etc., will first be classified by SOC, within each of which adverse events, etc., will be further classified by PT. |
| | Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. |
| Type of adverse events, etc. | For SOC, data will be presented in the internationally agreed |
| | order. For PT, data will be presented in ascending order of PT codes. |
| | If the same patient has multiple occurrences of the same adverse |
| | event, etc. (PT), the event with the worst CTCAE grade will be |
| | counted once. |

#### (3) Figure/table number

Table 5.2-2

- 5.2.3 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrence of adverse drug reactions/infections by outcome
  - (1) Analysis set to be used
    Safety analysis set
  - (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse drug reactions, etc., will be analyzed:

| Data item | Category |
|---|---|
| Seriousness | Serious or non-serious |
| CTCAE Grade (the worst one) | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| Time of onset | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, or ≥337 days |
| Time to the worst grade | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, or ≥337 days |
| Outcome | Recovered/resolved, recovering/resolving, not recovered/not resolved, recovered/resolved with sequelae, died/fatal, or unknown |

The type of adverse drug reactions, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse drug reactions, etc., by SOC/PT |
| Number of adverse drug reactions, etc. | Number of adverse drug reactions, etc., observed by SOC/PT |
| Type of adverse drug reactions, etc. | Adverse drug reactions, etc., will first be classified by SOC, within each of which adverse drug reactions, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. For SOC, data will be presented in the internationally agreed order. For PT, data will be presented in ascending order of PT codes. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the total number of occurrences will be calculated per category (for example, if the same patient has one episode of serious diarrhea and one episode of non-serious diarrhea, these adverse drug reactions will be counted once for each category). |

(3) Figure/table number

Table 5.2-3

#### 5.2.4 Occurrence of adverse drug reactions/infections by CTCAE Grade (the worst one)

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse drug reactions, etc., will be analyzed:

| Data item | Category |
|------------------------|--------------------------------|
| CTCAE Grade (the worst | ≤Grade 2, ≥Grade 3, or unknown |
| one) | |

The type of adverse drug reactions, etc., will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse drug reactions, etc., by SOC/PT |
| Number of adverse drug reactions, etc. | Number of adverse drug reactions, etc., observed by SOC/PT |
| Type of adverse drug reactions, etc. | Adverse drug reactions, etc., will first be classified by SOC, within each of which adverse drug reactions, etc., will be further classified by PT. Laboratory test data will first be classified by SOC, and will then be grouped into each HLGT and will be further classified by PT. For SOC, data will be presented in the internationally agreed order. For PT, data will be presented in ascending order of PT codes. If the same patient has multiple occurrences of the same adverse drug reaction, etc. (PT), the reaction with the worst CTCAE grade will be counted once. |

#### (3) Figure/table number

Table 5.2-4

# 5.3 Percentage of patients with adverse drug reactions/infections by patient demographics and baseline characteristics and treatment given

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the percentage of patients with adverse drug reactions, etc. (with point estimate and 95% confidence interval) will be determined.

For categories associated and not associated with ranking, Fisher's exact and Mann-Whitney U tests, respectively, will be used.

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| Diagnosis | Hodgkin's or anaplastic large-cell lymphoma or other |
| ALK (for patients with | |
| anaplastic large-cell | Positive, negative, or unknown |
| lymphoma) | |
| Clinical stage | I, II, III, IV, or unknown |
| B symptoms | Absent or present |
| ECOG Performance Status | 0, 1, 2, 3, or 4 |
| Hypersensitivity disposition | Absent, present, or unknown |
| Past history of pulmonary | Absent or present |
| disorders | 1.000m 01 p.200m |
| Concurrent pulmonary | Absent or present |
| disorders | 1 |
| Past history of malignant | Absent or present |
| tumours | |
| Concurrent malignant | Absent or present |
| tumours | |
| Concurrent hepatic | Absent or present |
| disorders | |
| Concurrent renal disorders | Absent or present |
| Weight | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, ≥70 kg, or not |
| | measured |
| BMI | $<18.5, <18.5 \text{ to } 25, <25 \text{ to } 30, \ge 30, \text{ or unknown}$ |
| Smoking history | Never, current, past, or unknown |
| Prior drug therapy | Absent or present |
| Prior radiotherapy | Absent or present |
| Prior hematopoietic stem | Absent, present (autologous), or present (homologous) |
| cell transplantation | resems, present (autorogous), or present (nomorogous) |
| Initial dose of Adcetris | 1.8 mg/kg or other |
| Mean dose of Adcetris | <1.8 mg/kg, 1.8 mg/kg, or ≥1.8 mg/kg |
| Dose of Adcetris per 3 | <1.8 mg/kg, 1.8 mg/kg, or ≥1.8 mg/kg |
| weeks | 0 0, ··· 0 0, ·· 2-100 |
| Drug(s) other than Adcetris | |
| used for the treatment of | Absent or present |
| the primary disease | |

#### (3) Figure/table number

#### 5.4 Occurrence of adverse drug reactions/infections by age group

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

The type of adverse drug reactions, etc., will be analyzed by age group (<18 years, 18 to 64 years, 65 to 74 years, or  $\ge$ 75 years).

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Table 5.4-1

5.5 Occurrence of adverse drug reactions/infections by presence or absence of concurrent hepatic

disorder

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

The type of adverse drug reactions, etc., will be analyzed by presence or absence of concurrent hepatic disorder.

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Table 5.5-1

- 5.6 Occurrence of adverse drug reactions/infections by presence or absence of concurrent renal disorder
  - (1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

The type of adverse drug reactions, etc., will be analyzed by presence or absence of concurrent renal disorder.

The type of adverse drug reactions, etc., will be analyzed in the same manner as described in Section 5.1.

(3) Figure/table number

Table 5.6-1

#### 5.7 List of the occurrence of serious adverse events/infections

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

Data listed below will be analyzed.

| Data listed below will be alia Data item | Data to be analyzed |
|---|---|
| Number of patients with | |
| serious adverse events, | Number of patients experiencing serious adverse events, etc. |
| etc. | |
| | Number of serious adverse events, etc., observed |
| Number of serious | If the same patient has multiple occurrences of the same serious |
| adverse events, etc. | adverse event, etc. (PT), the total number of occurrences will be |
| | calculated. |
| Percentage of patients | Is calculated using the following formula: number of patients with |
| with serious adverse | serious adverse events, etc./number of patients included in the |
| events, etc. | safety analysis set × 100. |
| | Serious adverse events, etc., will first be classified by SOC, within |
| | each of which serious adverse events, etc., will be further classified |
| | by PT. Laboratory test data will first be classified by SOC, and will |
| | then be grouped into each HLGT and will be further classified by |
| | PT. |
| | For SOC, the number and percentage of patients with serious |
| Type of serious adverse | adverse events, etc., will be presented in the internationally agreed |
| events | order. |
| | For PT, the number and percentage of serious adverse events, etc., |
| | will be presented in ascending order of PT codes. |
| | If the same patient has multiple occurrences of the same serious |
| | adverse event, etc. (PT), the event will be counted once per patient. |
| | For serious adverse events, etc., considered not related to Adcetris, |
| | the number of these events will be presented in [ ]. |

#### (3) Figure/table number

Table 5.7-1

#### 5.8 Change in test data over time

#### 5.8.1 Laboratory tests

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

Summary statistics of red blood cell count, hemoglobin level, white blood cell count, neutrophil count, lymphocyte count, platelet count, total bilirubin, AST, ALT, LDH, BUN, and serum creatinine will be calculated at each test time point [at baseline, after 1 cycle, ... and after 16 cycles].

(3) Figure/table number

Table 5.8-1

#### 5.9 Analysis of items of particular interest

#### 5.9.1 Occurrence of peripheral nerve disorder

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

For CTCAE Grade (the worst one), patients will be stratified into the following categories, and the incidence of peripheral nerve disorders will be calculated:

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | |
| one) for peripheral nerve | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| disorders | |

Symptoms of peripheral nerve disorders will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Symptoms of peripheral nerve disorders | Peripheral nerve disorders will first be classified into peripheral sensory, peripheral motor, and peripheral neuropathies listed in Section 1.1, and symptoms associated with these peripheral nerve disorders will be analyzed by PT. If the same patient has multiple occurrences of the same symptom (PT), the symptom with the worst CTCAE grade will be counted once. |

#### (3) Figure/table number

- 5.9.2 Occurrence of peripheral nerve disorders by patient demographics and baseline characteristics and treatment given
  - (1) Analysis set to be used Safety analysis set
  - (2) Data to be analyzed

For each data item, patients will be stratified into the categories below, and the incidence of peripheral nerve disorders will be calculated by CTCAE Grade (the worst one). If the same patient has multiple occurrences of the same peripheral nerve disorder (PT), the peripheral nerve disorder with the worst CTCAE grade will be counted once.

| Data item | Category |
|---|---|
| Sex | Male or female |
| Age | <18 years, 18 to 64 years, 65 to 74 years, or ≥75 years |
| Disease duration | <1 year, <1 to 3 years, <3 to 5 years, ≥5 years, or unknown |
| ECOG Performance Status | 0, 1, 2, 3, or 4 |
| Grade of concurrent peripheral nerve disorders | None, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |
| Weight | <40 kg, <40 to 50 kg, <50 to 60 kg, <60 to 70 kg, ≥70 kg, or not measured |
| Prior ABVD or CHOP | Absent or present |
| Prior radiotherapy | Absent or present |
| Prior hematopoietic stem cell transplantation | Absent, present (autologous), or present (homologous) |
| Initial dose of Adcetris | 1.8 mg/kg or other |
| Mean dose of Adcetris | <1.8 mg/kg, 1.8 mg/kg, or ≥1.8 mg/kg |
| Dose of Adcetris per 3 weeks | <1.8 mg/kg, 1.8 mg/kg, or ≥1.8 mg/kg |
| Concurrent diabetes mellitus | Absent or present |

#### (3) Figure/table number

#### 5.9.3 Treatment with Adcetris at the onset of peripheral nerve disorders

#### (1) Analysis set to be used

Patients included in the safety analysis set who experience peripheral nerve disorders considered related to Adcetris

#### (2) Data to be analyzed

For each CTCAE Grade (the worst one) of peripheral nerve disorders, patients will be stratified into the categories below, and the number of peripheral nerve disorders will be calculated. If the same patient has multiple occurrences of the same peripheral nerve disorder (PT), the total number of occurrences will be calculated per category (for example, if the same patient has one episode of peripheral nerve disorder requiring dose reduction and one episode of peripheral nerve disorder leading to treatment discontinuation, these episodes of peripheral nerve disorder will be counted once for each category).

| Data item Category | |
|---|---|
| Action taken to Adcetris | No action taken or action taken in response to the event |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), or |
| Adcetris | treatment discontinuation |

#### (3) Figure/table number

Table 5.9-3

#### 5.9.4 Occurrence of infections by presence or absence of drugs used for the prevention of infection

#### (1) Analysis set to be used

Safety analysis set

#### (2) Data to be analyzed

Patients will be stratified into the categories below and the number of patients with infection will be calculated by presence or absence of drugs used for the prevention of infection using Mann-Whitney U test. If the same patient has multiple occurrences of the same infection, the occurrence with the worst CTCAE grade will be counted once.

Similarly, the number of patients with the onset of bacterial infection will be calculated by the use or non-use of antibiotics/synthetic antibacterial agents or trimethoprim-sulfamethoxazole combinations, the number of patients with the onset of fungal infection will be calculated by the use or non-use of antifungals, and the number of patients with the onset of viral infection will be calculated by the use or non-use of antivirals.

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | None, Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infections | |

#### (3) Figure/table number

#### 5.9.5 Occurrence of neutropenia by patient demographics and baseline characteristics

(1) Analysis set to be used

Safety analysis set

#### (2) Data to be analyzed

For each data item, patients will be stratified into the categories below, and the incidence of neutropenia will be calculated by CTCAE Grade (the worst one). If the same patient has multiple occurrences of neutropenia, the event with the worst CTCAE grade will be counted once.

| Data item | Category |
|---|---|
| Prior hematopoietic stem cell transplantation | Absent, present (autologous), or present (homologous) |
| Degree of decreased neutrophil count at baseline | No decrease, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |

#### (3) Figure/table number

Table 5.9-5

#### 5.9.6 Treatment with Adcetris at the onset of neutropenia

#### (1) Analysis set to be used

Patients included in the safety analysis set who experience neutropenia considered related to Adcetris

#### (2) Data to be analyzed

For each CTCAE Grade (the worst one) of neutropenia, patients will be stratified into the categories below, and the number of events of neutropenia will be calculated. If the same patient has multiple occurrences of neutropenia, the total number of occurrences will be calculated per category (for example, if the same patient has one episode of peripheral nerve disorder requiring dose reduction and one episode of peripheral nerve disorder leading to treatment discontinuation, these episodes of peripheral nerve disorder will be counted once for each category).

| Data item | Category |
|---|---|
| Action taken to Adcetris | No action taken or action taken in response to the event |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), or |
| Adcetris | treatment discontinuation |

#### (3) Figure/table number

#### 5.9.7 Occurrence of infusion reaction

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

For CTCAE Grade (the worst one), patients will be stratified into the following categories, and the incidence of infusion reaction will be calculated:

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infusion reaction | |

Infusion reaction will be analyzed as follows:

| Data | a item | 1 | Data to be analyzed |
|---|---|---|---|
| | | | Infusion reaction and its symptoms will be analyzed by PT. |
| Symptoms | of | infusion | If the same patient has multiple occurrences of the same symptom |
| reaction | | | (PT), the symptom with the worst CTCAE grade will be counted |
| | | | once. |

#### (3) Figure/table number

Table 5.9-7

# 5.9.8 Occurrence of infusion reaction by the use or non-use of premedication to prevent infusion reaction

(1) Analysis set to be used

Safety analysis set

(2) Data to be analyzed

Patients will be stratified into the following categories and the number of events of infusion reaction considered related to Adcetris will be calculated by the use or non-use of premedication to prevent infusion reaction (for example, if a patient receives no premedication and experiences "Grade 2" infusion reaction during Cycle 1 and receives premedication and experiences no infusion reaction during Cycle 2, these events of infusion reaction will be counted once for each category).

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | None, Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of infusion reaction | |

#### (3) Figure/table number

#### 5.9.9 Occurrence of pulmonary disorders

(1) Analysis set to be used

Safety analysis set

#### (2) Data to be analyzed

For CTCAE Grade (the worst one), patients will be stratified into the following categories, and the incidence of events of pulmonary disorder will be calculated:

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | |
| one) for pulmonary | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| disorders | |

Diagnoses or symptoms of pulmonary disorder will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Diagnosis or symptom of pulmonary disorder | Pulmonary disorders and their diagnoses or symptoms will be analyzed by PT. If the same patient has multiple occurrences of the same symptom (PT), the symptom with the worst CTCAE grade will be counted |
| | once. |

#### (3) Figure/table number

#### 6.0 Efficacy Analysis

#### 6.1 Best response

(1) Analysis set to be used

Efficacy analysis set

(2) Data to be analyzed

The best responses after 16 cycles of treatment with Adcetris (or upon discontinuation of treatment with Adcetris) will be analyzed in patients Hodgkin's lymphoma and patients with anaplastic large-cell lymphoma.

(3) Figure/table number

Table 6.1-1

#### 6.2 Overall survival

(1) Analysis set to be used

Efficacy analysis set

(2) Data to be analyzed

The survivals from the date of the initial dose of Adcetris in patients Hodgkin's lymphoma and patients with anaplastic large-cell lymphoma will be calculated, using the final observation date as the date of survival confirmation and the date of outcome of an adverse event with "Died/fetal" recorded in the Outcome field as the date of death.

Kaplan-Meier curves of the survival will also be constructed (i.e., a table of the numbers of adverse events, etc., and adverse drug reactions, etc., printed out by SAS will be attached).

(3) Figure/table number

Table 6.2-1 and Figure 6.2-1

#### Appendix: Definition of Pulmonary Disorders (MedDRA Preferred Terms)

The above definition is consistent with the one used in clinical studies of Adcetris.

# Supplemental Statistical Analysis Plan ADCETRIS IV Infusion — Special Drug Use Surveillance (All-case Surveillance) "Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell Lymphoma"



Initial version: Prepared on September 15, 2017

#### Table of Contents

| 1.0 | | Definition of Analysis sets and Terms and Handling of Test/Measurement Data | 1 |
|---|---|---|---|
| 1. | 1 | Analysis sets | 1 |
| | 1.1. | 1 Safety analysis set | 1 |
| 1. | 2 | Definition | 1 |
| 1. | 3 | Display digits | 3 |
| 1. | 4 | Handling of test data | 3 |
| 1. | 5 | Handling of missing data | 6 |
| 1. | 6 | Others | 6 |
| 2.0 | | Safety Analysis | 7 |
| 2. | 1 | Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrences | эf |
| | | adverse drug reactions/infections by outcome | 7 |
| 2. | 2 | Analysis of items of particular interest | 9 |
| | 2.2. | 1 Treatment-related infections reported within 7 days after the date of the worst grade of Grade 3 or | 4 |
| | neu | tropenia or the date of onset of Grade 3 or 4 decreased neutrophil count considered related to Adcetris | 9 |
| | 2.2. | 2 Treatment-related infections reported within 7 days after the date of the worst grade of Grade 3 or | 4 |
| | lym | phopenia or the date of onset of Grade 3 or 4 decreased lymphocyte count considered related to Adcetris | 9 |

#### 1.0 Definition of Analysis sets and Terms and Handling of Test/Measurement Data

#### 1.1 Analysis sets

#### 1.1.1 Safety analysis set

In this survey, the safety analysis set is defined as patients treated with Adcetris IV Infusion with no major protocol violation and evaluable for safety. In this Statistical Analysis Plan, the safety analysis set refers to patients included in safety evaluation.

#### 1.2 Definition

| Term | Definition |
|---|---|
| This/the product | Refers to Adcetris for intravenous drip infusion in this Statistical Analysis |
| | Plan. |
| SOC | MedDRA/J System Organ Class |
| PT | MedDRA/J Preferred Term |
| Safety analysis set | Fixed patients included in the safety analysis set |
| Safety analysis set | Patients included in the safety analysis set whose diagnosis is Hodgkin's |
| (Hodgkin's lymphoma) | lymphoma |
| Safety analysis set | Patients included in the safety analysis set whose diagnosis is anaplastic |
| (anaplastic large-cell | large-cell lymphoma |
| lymphoma) | |
| Adverse drug reactions, | Refers to "adverse drug reactions and infections." |
| etc. | Adverse events not considered "not related" to Adcetris by the investigator. |
| | In this Statistical Analysis Plan, the term "adverse drug reactions and |
| | infections" is used in titles and the term "adverse drug reactions, etc." is used |
| | in text and tables. |
| Number of patients with | Number of patients experiencing adverse events or adverse drug reactions, |
| adverse events/adverse | etc. |
| drug reactions | |
| Number of adverse | Number of adverse events or adverse drug reactions, etc., observed |
| events/adverse drug | |
| reactions | |
| Percentage of patients with | [For safety analysis using patients included in the safety analysis set] |
| adverse events/adverse | Is calculated using the following formula: (number of patients with |
| drug reactions | adverse events/adverse drug reactions) / (number of patients included in the |
| | safety analysis set) × 100. |
| | [For safety analysis using patients excluded from the safety analysis set] |
| | Is calculated using the following formula: (number of patients with |
| | adverse events/adverse drug reactions) / (number of patients excluded from |
| | the safety analysis set) $\times$ 100. |
| Percentage of adverse | [For safety analysis using patients included in the safety analysis set] |

| Term | Definition |
|---|---|
| events/adverse drug | Is calculated using the following formula: (number of adverse |
| reactions observed | events/adverse drug reactions observed) / (number of patients included in the |
| | safety analysis set) × 100. |
| | [For safety analysis using patients excluded from the safety analysis set] |
| | Is calculated using the following formula: (number of adverse |
| | events/adverse drug reactions observed) / (number of patients excluded from |
| | the safety analysis set) × 100. |
| Time of onset | Is calculated using the following formula: date of onset of adverse events (or |
| | adverse drug reactions, etc.) – date of the initial dose of Adcetris + 1. |
| | If the day, month, and year of onset of adverse events (or adverse drug |
| | reactions, etc.) are unknown, the time of onset should be handled as missing, |
| | and the category for the time of onset should be "unknown." |
| Time to the worst grade | Is calculated using the following formula: date of the worst CTCAE grade – |
| | date of the initial dose of Adcetris + 1. |
| | If the day, month, and year of the worst CTCAE grade are unknown, the date |
| | of the worst CTCAE grade should be handled as missing, and the category |
| | for the date of the worst CTCAE grade should be "unknown." |
| Infection | A concurrent illness or adverse event that falls under the category of |
| | MedDRA SOC Code 10021881 (Infections and infestations) |
| Grade 3 or 4 decreased | Neutrophil count <1,000/mm <sup>3</sup> |
| neutrophil count | |
| Grade 3 or 4 decreased | Lymphocyte count < 500/mm <sup>3</sup> |
| lymphocyte count | |
| Neutropenia | An adverse event equivalent to MedDRA PT Codes 10029366 (Neutrophil |
| | count decreased) and 10029354 (Neutropenia). |
| Lymphopenia | An adverse event equivalent to MedDRA PT Codes 10025256 (Lymphocyte |
| | count decreased) and 10025327 (Lymphopenia). |

#### 1.3 Display digits

| Term | Definition |
|---|---|
| Percentage (%) | Percentage of patients with or percentage of adverse events or adverse drug |
| | reactions, etc.: |
| | The obtained value should be rounded off to two decimal places. |
| | Other: |
| | The obtained value should be rounded off to one decimal place. |

#### 1.4 Handling of test data

Test data will be handled according to the criteria shown below. If there are multiple data for the same criterion, the one with the test date being closest to the date of protocol-specified assessment should be used. If there is no difference in the number of days from the date of protocol-specified assessment, the later value should be used.

The number of days after the date of the initial dose of Adcetris is defined as 1 for the date of the initial dose of Adcetris and 0 for the day before the date of the initial dose of Adcetris.

| Time point for testing | Date of protocol-specified assessment | Acceptable time window |
|---|---|---|
| At the initial dose of | Date of the initial dose of Adcetris | -15 days to the d ate of the initial dose of |
| Adcetris | | Adcetris |
| After 1 cycle | • If Cycle 2 is initiated: Date of Cycle | • If Cycle 2 is initiated: Date of Cycle 2 |
| | 2 | • If Cycle 2 is not initiated: 21 days after |
| | • If Cycle 2 is not initiated: 21 days | the date of the initial dose of Adcetris |
| | after the date of the initial dose of | |
| | Adcetris s | |
| After 2 cycles | • If Cycle 3 is initiated: Date of Cycle | • If Cycle 3 is initiated: From the day |
| | 3 | after the date of Cycle 2 to the day of |
| | • If Cycle 3 is not initiated: 21 days | Cycle 3 |
| | after the date of Cycle 2 | • If Cycle 3 is not initiated: From the day |
| | | after the date of Cycle 2 to 21 days |
| | | after the date of Cycle 2 |
| After 3 cycles | • If Cycle 4 is initiated: Date of Cycle | If Cycle 4 is initiated: From the day |
| | 4 | after the date of Cycle 3 to the day of |
| | • If Cycle 4 is not initiated: 21 days | Cycle 4 |
| | after the date of Cycle 3 | • If Cycle 4 is not initiated: From the day |
| | | after the date of Cycle 3 to 21 days |
| | | after the date of Cycle 3 |

| Time point for testing | Date of protocol-specified assessment | Acceptable time window |
|---|---|---|
| After 4 cycles | • If Cycle 5 is initiated: Date of Cycle | If Cycle 5 is initiated: From the day |
| | 5 | after the date of Cycle 4 to the day of |
| | • If Cycle 5 is not initiated: 21 days | Cycle 5 |
| | after the date of Cycle 4 | • If Cycle 5 is not initiated: From the day |
| | | after the date of Cycle 4 to 21 days |
| | | after the date of Cycle 4 |
| After 5 cycles | • If Cycle 6 is initiated: Date of Cycle | • If Cycle 6 is initiated: From the day |
| | 6 | after the date of Cycle 5 to the day of |
| | • If Cycle 6 is not initiated: 21 days | Cycle 6 |
| | after the date of Cycle 5 | • If Cycle 6 is not initiated: From the day |
| | | after the date of Cycle 5 to 21 days |
| | | after the date of Cycle 5 |
| After 6 cycles | If Cycle 7 is initiated: Date of Cycle | If Cycle 7 is initiated: From the day |
| | 7 | after the date of Cycle 6 to the day of |
| | • If Cycle 7 is not initiated: 21 days | Cycle 7 |
| | after the date of Cycle 6 | • If Cycle 7 is not initiated: From the day |
| | | after the date of Cycle 6 to 21 days |
| | | after the date of Cycle 6 |
| After 7 cycles | • If Cycle 8 is initiated: Date of Cycle | If Cycle 8 is initiated: From the day |
| | 8 | after the date of Cycle 7 to the day of |
| | • If Cycle 8 is not initiated: 21 days | Cycle 8 |
| | after the date of Cycle 7 | If Cycle 8 is not initiated: From the day |
| | | after the date of Cycle 7 to 21 days |
| | | after the date of Cycle 7 |
| After 8 cycles | • If Cycle 9 is initiated: Date of Cycle | • If Cycle 9 is initiated: From the day |
| | 9 | after the date of Cycle 8 to the day of |
| | • If Cycle 9 is not initiated: 21 days | Cycle 9 |
| | after the date of Cycle 8 | • If Cycle 9 is not initiated: From the day |
| | | after the date of Cycle 8 to 21 days |
| | | after the date of Cycle 8 |
| After 9 cycles | • If Cycle 10 is initiated: Date of | If Cycle 10 is initiated: From the day |
| | Cycle 10 | after the date of Cycle 9 to the day of |
| | • If Cycle 10 is not initiated: 21 days | Cycle 10 |
| | after the date of Cycle 9 | • If Cycle 10 is not initiated: From the |
| | | day after the date of Cycle 9 to 21 days |
| | | after the date of Cycle 9 |

| Time point for testing | Date of protocol-specified assessment | Acceptable time window |
|---|---|---|
| After 10 cycles | If Cycle 11 is initiated: Date of | If Cycle 11 is initiated: From the day |
| | Cycle 11 | after the date of Cycle 10 to the day of |
| | • If Cycle 11 is not initiated: 21 days | Cycle 11 |
| | after the date of Cycle 10 | If Cycle 11 is not initiated: From the |
| | | day after the date of Cycle 10 to 21 |
| | | days after the date of Cycle 10 |
| After 11 cycles | If Cycle 12 is initiated: Date of | If Cycle 12 is initiated: From the day |
| | Cycle 12 | after the date of Cycle 11 to the day of |
| | If Cycle 12 is not initiated: 21 days | Cycle 12 |
| | after the date of Cycle 11 | • If Cycle 12 is not initiated: From the |
| | | day after the date of Cycle 11 to 21 |
| | | days after the date of Cycle 11 |
| After 12 cycles | If Cycle 13 is initiated: Date of | If Cycle 13 is initiated: From the day |
| | Cycle 13 | after the date of Cycle 12 to the day of |
| | • If Cycle 13 is not initiated: 21 days | Cycle 13 |
| | after the date of Cycle 12 | If Cycle 13 is not initiated: From the |
| | | day after the date of Cycle 12 to 21 |
| | | days after the date of Cycle 12 |
| After 13 cycles | If Cycle 14 is initiated: Date of | If Cycle 14 is initiated: From the day |
| | Cycle 14 | after the date of Cycle 13 to the day of |
| | • If Cycle 14 is not initiated: 21 days | Cycle 14 |
| | after the date of Cycle 13 | If Cycle 14 is not initiated: From the |
| | | day after the date of Cycle 13 to 21 |
| | | days after the date of Cycle 13 |
| After 14 cycles | If Cycle 15 is initiated: Date of | If Cycle 15 is initiated: From the day |
| | Cycle 15 | after the date of Cycle 14 to the day of |
| | • If Cycle 15 is not initiated: 21 days | Cycle 15 |
| | after the date of Cycle 14 | If Cycle 15 is not initiated: From the |
| | | day after the date of Cycle 14 to 21 |
| | | days after the date of Cycle 14 |
| After 15 cycles | If Cycle 16 is initiated: Date of | If Cycle 16 is initiated: From the day |
| | Cycle 16 | after the date of Cycle 15 to the day of |
| | • If Cycle 16 is not initiated: 21 days | Cycle 16 |
| | after the date of Cycle 15 | If Cycle 16 is not initiated: From the |
| | | day after the date of Cycle 15 to 21 |
| | | days after the date of Cycle 15 |

#### 1.5 Handling of missing data

- As a general rule, missing data will not be imputed.
- In the analysis of the frequency qualitative variables, missing data will be handles as "unknown."

#### 1.6 Others

- In the analysis for the preparation of documents for the Final Survey Report, MedDRA version 19.1 will be used for adverse events, concurrent illness, and past history.
- If a patient has multiple data for a single laboratory test and date of testing, the mean value will be calculated for the analysis of laboratory test results.

#### 2.0 Safety Analysis

2.1 Seriousness, CTCAE Grade (the worst one), time of onset, time to the worst grade, and occurrences of adverse drug reactions/infections by outcome

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item, patients will be stratified into the following categories, and the type of adverse events will be analyzed:

| Data item | Category |
|---|---|
| Seriousness | Serious or non-serious |
| CTCAE Grade (the worst one) | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, ≥337 days, or unknown |
| Time of onset | 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly using a 21-day time window thereafter), 316 to 336 days, ≥337 days, or unknown |
| Time to the worst grade | 1 to 7 days, 8 to 14 days, 15 to 21 days, 22 to 84 days, 85 to 168 days, 169 to 252 days, 253 to 336 days, ≥337 days, or unknown 1 to 21 days, 22 to 42 days, 43 to 63 days, (segmented similarly using a 21-day time window thereafter), 316 to 336 days, ≥337 days, or unknown |
| Outcome | Recovered/resolved, recovering/resolving, not recovered/not resolved, recovered/resolved with sequelae, died/fatal, unknown, or not provided |

The type of adverse events will be analyzed as follows:

| Data item | Data to be analyzed |
|---|---|
| Number of patients | Number of patients with adverse events by SOC/PT |
| | Number of adverse events observed by SOC/PT |
| Number of adverse events, | If the same patient has multiple occurrences of the same adverse |
| etc. | event (PT), all these occurrences will be counted (i.e., the overlap |
| | should be reflected). |
| | The number of adverse events will be calculated by SOC and PT. |
| | SOCs will be presented in the internationally agreed order, and |
| Seriousness, time of onset, | PTs will be presented in ascending order of HLGT and PT codes |
| and outcome | if their SOCs are "Investigations," and in ascending order of PT |
| | code otherwise. |
| | If the same patient has multiple occurrences of the same adverse |

| | event (PT), the total number of occurrences will be calculated per |
|---|---|
| | category (for example, if the same patient has one episode of |
| | serious diarrhea and one episode of non-serious diarrhea, these |
| | events will be counted once for each category). If the same patient |
| | has multiple occurrences of the same adverse event classified into |
| | the same category, all these occurrences will be counted (i.e., the |
| | overlap should be reflected). |
| CTCAE Grade (the worst one) and time to the worst grade | The number of adverse events will be calculated by SOC and PT. |
| | The CTCAE grade is higher in the order of Grade 5, 4, 3, 2, 1, and |
| | unknown. The event with the highest CTCAE grade (the worst |
| | one) and the shortest time to the worst grade will be counted once. |

- 2.2 Analysis of items of particular interest
- 2.2.1 Treatment-related infections reported within 7 days after the date of the worst grade of Grade 3 or 4 neutropenia or the date of onset of Grade 3 or 4 decreased neutrophil count considered related to Adcetris
  - (1) Analysis sets to be used

Patients included in the safety analysis set with confirmed Grade 3 or 4 neutropenia or decreased neutrophil count considered related to Adcetris

(2) Data to be analyzed

The number and percentage of patients experiencing treatment-related infections reported within 7 days after the date of the worst grade of Grade 3 or 4 neutropenia or the date of onset of Grade 3 or 4 decreased neutrophil count considered related to Adcetris will be calculated by infection and PT (for the definition of infection, see Section 1.2). PTs will be presented in ascending order of PT codes.

- 2.2.2 Treatment-related infections reported within 7 days after the date of the worst grade of Grade 3 or 4 lymphopenia or the date of onset of Grade 3 or 4 decreased lymphocyte count considered related to Adcetris
  - (1) Analysis sets to be used

Patients included in the safety analysis set with confirmed Grade 3 or 4 lymphopenia or decreased lymphocyte count considered related to Adcetris

(2) Data to be analyzed

The number and percentage of patients experiencing treatment-related infections reported within 7 days after the date of the worst grade of Grade 3 or 4 lymphopenia or the date of onset of Grade 3 or 4 decreased lymphocyte count considered related to Adcetris will be calculated by infection and PT (for the definition of infection, see Section 1.2). PTs will be presented in ascending order of PT codes.

### Supplemental Statistical Analysis Plan 2

Additional Analysis on Neutropenia

# ADCETRIS IV Infusion – Special Drug Use Surveillance (All-case Surveillance) "Relapsed or Refractory CD30+ Hodgkin's Lymphoma or Anaplastic Large Cell Lymphoma"



Initial version: Prepared on November 21, 2017

#### Table of Contents

| 1.0 | Definition of Analysis sets and Terms and Handling of Test/Measurement Data | |
|---|---|---|
| 1.1 | Analysis sets | 1 |
| 1.1 | .1 Safety analysis set | 1 |
| 1.2 | Definition | 1 |
| 1.3 | Display digits | 3 |
| 1.4 | Handling of missing data | 3 |
| 1.5 | Others | 3 |
| 2.0 | Safety Analysis | 4 |
| 2.1 | Analysis of items of particular interest | 4 |
| 2.1 | .1 Occurrence of neutropenia considered related to Adcetris by patient demographics and b | aseline |
| cha | aracteristics | 4 |
| 2.1 | .2 Treatment with Adcetris at the onset of neutropenia considered related to Adcetris | 4 |
| 2.1 | | 6 |

#### 1.0 Definition of Analysis sets and Terms and Handling of Test/Measurement Data

#### 1.1 Analysis sets

#### 1.1.1 Safety analysis set

In this survey, the safety analysis set is defined as patients treated with Adcetris IV Infusion with no major protocol violation and evaluable for safety. In this Statistical Analysis Plan, the safety analysis set refers to patients included in safety evaluation.

#### 1.2 Definition

| | Definition |
|---|---|
| Refers to Adcetris | for intravenous drip infusion in this Statistical Analysis |
| Plan. | |
| MedDRA/J System Organ Class | |
| MedDRA/J Prefer | red Term |
| Fixed patients incl | luded in the safety analysis set |
| Patients included i | in the safety analysis set whose diagnosis is Hodgkin's |
| lymphoma | |
| Patients included in the safety analysis set whose diagnosis is anaplastic | |
| large-cell lymphor | na |
| Events equivalent | to MedDRA PT Codes 10029354 (Neutropenia) and |
| 10016288 (Febrile | neutropenia) will be collected and analyzed. Neutrophil |
| count decreased (F | PT Code 10029366) will be replaced with Neutropenia |
| (PT Code 1002935 | 54). |
| The neutrophil count at baseline will be classified as shown in the table | |
| below. If the neutr | ophil count at baseline is missing, the degree of |
| decreased neutrop | hil count should be handled as missing: |
| No decrease | ≥2,000 /mm <sup>3</sup> |
| Grade 1 | ≥1,500 to <2,000 /mm <sup>3</sup> |
| Grade 2 | ≥1,000 to <1,500 /mm <sup>3</sup> |
| Grade 3 | ≥500 to <1,000 /mm <sup>3</sup> |
| Grade 4 | <500 /mm <sup>3</sup> |
| Drugs with the firs | st three digits of YJ Code being either one of 611 to 616, |
| | re entered in the field of "Drugs used for the prevention |
| | ore than one antibiotics/synthetic antibacterial agents |
| , | ne patient, it will be counted as one patient.) |
| | st three digits of YJ Code being 617 or the first seven |
| | 002 or 6290004 that are entered in the field of "Drugs |
| | ntion of infection" (If more than one antifungals are |
| | Plan. MedDRA/J Syster MedDRA/J Prefer Fixed patients incl Patients included in lymphoma Patients included in large-cell lymphoma Events equivalent 10016288 (Febrille count decreased (If (PT Code 100293)) The neutrophil count decreased neutrop No decrease Grade 1 Grade 2 Grade 3 Grade 4 Drugs with the first 619, or 624 that are of infection" (If mare used in the same Drugs with the first digits being 62900) |

| Term | Definition |
|---|---|
| | used in the same patient, it will be counted as one patient.) |
| Antivirals | Drugs with the first three digits of YJ Code being 625 that are entered in |
| | the field of "Drugs used for the prevention of infection" (If more than one |
| | antivirals are used in the same patient, it will be counted as one patient.) |
| Trimethoprim-sulfamethoxazole | Drugs with YJ Code being 62901000 that are entered in the field of |
| combinations | "Drugs used for the prevention of infection" (If more than one |
| | trimethoprim-sulfamethoxazole combinations are used in the same patient, |
| | it will be counted as one patient.) |
| Other prophylactics against | Any drug entered in the field of "Drugs used for the prevention of |
| infections | infection" other than prophylactics against infections listed above (If more |
| | than one other prophylactics against infections are used in the same |
| | patient, it will be counted as one patient.) |

#### 1.3 Display digits

| Term | Definition |
|---|---|
| Percentage (%) | Percentage of patients with or percentage of adverse events or adverse drug |
| | reactions, etc.: |
| | The obtained value should be rounded off to two decimal places. |
| | Other: |
| | The obtained value should be rounded off to one decimal place. |

#### 1.4 Handling of missing data

- As a general rule, missing data will not be imputed.
- In the analysis of the frequency qualitative variables, missing data will be handles as "unknown." In the analysis of summary statistics of quantitative variables, missing data will be excluded.

#### 1.5 Others

• In the analysis for the preparation of documents for the Final Survey Report (final analysis), MedDRA version 19.1 will be used for adverse events, concurrent illness, and past history.

#### 2.0 Safety Analysis

#### 2.1 Analysis of items of particular interest

# 2.1.1 Occurrence of neutropenia considered related to Adcetris by patient demographics and baseline characteristics

#### (1) Analysis sets to be used

Safety analysis set, safety analysis set (Hodgkin's lymphoma), and safety analysis set (anaplastic large-cell lymphoma)

#### (2) Data to be analyzed

For each data item of patient demographics and baseline characteristics, patients will be stratified into the categories below, and the incidence of neutropenia considered related to Adcetris will be calculated by CTCAE Grade (the worst one). The CTCAE grade (the worst one) is higher in the order of Grades 5, 4, 3, 2, 1, and unknown. If the same patient has multiple occurrences of neutropenia, the event with the highest CTCAE grade will be counted once.

| Data item | Category |
|---|---|
| CTCAE Grade (the worst | Grade 1, Grade 2, Grade 3, Grade 4, Grade 5, or unknown |
| one) of neutropenia | |

#### Items and categories of patient demographics and baseline characteristics

| Data item | Category |
|---|---|
| Prior hematopoietic stem | Absent, present (autologous), present (homologous), present |
| cell transplantation | (autologous and homologous), or unknown |
| Degree of decreased | No decrease Crede 1 Crede 2 Crede 2 Crede 4 on university |
| neutrophil count at baseline | No decrease, Grade 1, Grade 2, Grade 3, Grade 4, or unknown |
| Drugs used for the | Absent or present |
| prevention of infection | |
| Specific drug(s) used for | Antibiotics/synthetic antibacterial agents, antifungals, antivirals, |
| the prevention of infection | trimethoprim-sulfamethoxazole combinations, or other |

#### (3) Figure/table number

Tables 2.1.1-1 to 2.1.1-3

#### 2.1.2 Treatment with Adcetris at the onset of neutropenia considered related to Adcetris

#### (1) Analysis sets to be used

Patients included in the safety analysis set and safety analysis set (Hodgkin's lymphoma) or safety analysis set (anaplastic large-cell lymphoma) who experience neutropenia considered related to Adcetris

#### (2) Data to be analyzed

For each CTCAE Grade (the worst one) of neutropenia considered related to Adcetris, patients will be stratified into the categories below, and the incidence of events of neutropenia will be calculated. If the same patient has multiple occurrences of neutropenia, the total number of occurrences will be calculated per category (for example, if the same patient has one episode of

peripheral nerve disorder requiring dose reduction and one episode of peripheral nerve disorder leading to treatment discontinuation, these episodes of peripheral nerve disorder will be counted once for each category). The percentage of neutropenia for each category will be calculated using the number of neutropenia for each CTCAE grade (the worst one) as the denominator.

For each data item, missing data will be handled as "not provided."

| Data item | Category |
|---|---|
| Action taken to Adcetris | No action taken or action taken in response to the event or not provided |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), |
| Adcetris | treatment discontinuation or not provided |

#### (3) Figure/table number

Tables 2.1.2-1 to 2.1.2-3

#### 2.1.3 Outcome of neutropenia considered related to Adcetris by action taken with Adcetris

#### (1) Analysis sets to be used

Patients included in safety evaluation and patients included in safety evaluation (Hodgkin's lymphoma) or patients included in safety evaluation (anaplastic large-cell lymphoma) who experience neutropenia considered related to Adcetris

#### (2) Data to be analyzed

For neutropenia considered related to Adcetris, patients will be stratified into the categories below for each outcome and the incidence of neutropenia will be calculated. If the same patient has multiple occurrences of neutropenia, the total number of occurrences will be calculated per category (for example, if the same patient has one episode of neutropenia requiring dose reduction and one episode of neutropenia leading to treatment discontinuation, these episodes of neutropenia will be counted once for each category). The percentage of neutropenia for each category will be calculated using the total number of neutropenia for each category as the denominator.

For each data item, missing data will be handled as "not provided."

| Data item | Category |
|---|---|
| Action taken to Adcetris | No action taken or action taken in response to the event or not |
| Action taken to Auceurs | provided |
| Specific action taken to | Dose reduction, treatment interruption (treatment delay), |
| Adcetris | treatment discontinuation, or not provided |

#### (3) Figure/table number

Tables 2.1.3-1 to 2.1.3-3